CLINICAL TRIAL: NCT02880956
Title: A Phase 2 Multiple Dose, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of ABBV-8E12 in Subjects With Early Alzheimer's Disease
Brief Title: A Study to Evaluate the Efficacy and Safety of ABBV-8E12 in Participants With Early Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M15-566; 2016-001634-10 (EudraCT Number)
Expanded Access: NCT03744546 (No longer available)
Record Dates: First submitted 2016-08-24; First posted 2016-08-26 (Estimated); Results first posted 2022-08-26 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Alzheimer's Disease
Keywords: Early Alzheimer's Disease (AD); Mild Cognitive Impairment (MCI); Mild Alzheimer's Disease (AD); Tau; Early dementia; Tauopathies; AD; Neurodegenerative diseases; Memory loss; Nervous system diseases
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Pick Disease of the Brain; Dementia; Tauopathies; Neurodegenerative Diseases; Memory Disorders; Nervous System Diseases | interventions — tilavonemab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Placebo (Placebo Comparator): Placebo for ABBV-8E12 every 4 weeks for 96 weeks
  Interventions: Drug: placebo for ABBV-8E12
- ABBV-8E12 300 mg (Experimental): ABBV-8E12 300 mg every 4 weeks for 96 weeks
  Interventions: Drug: ABBV-8E12
- ABBV-8E12 1000 mg (Experimental): ABBV-8E12 1000 mg every 4 weeks for 96 weeks
  Interventions: Drug: ABBV-8E12
- ABBV-8E12 2000 mg (Experimental): ABBV-8E12 2000 mg every 4 weeks for 96 weeks
  Interventions: Drug: ABBV-8E12

INTERVENTIONS:
Drug: ABBV-8E12 — ABBV-8E12 solution for IV infusion
  Other Names: Tilavonemab
  Arms: ABBV-8E12 1000 mg; ABBV-8E12 2000 mg; ABBV-8E12 300 mg
Drug: placebo for ABBV-8E12 — placebo solution for intravenous (IV) infusion
  Arms: Placebo

SUMMARY:
This study seeks to evaluate the efficacy and safety of ABBV-8E12 in participants with early Alzheimer's disease (AD).

ELIGIBILITY:
Inclusion Criteria:

* Subject who meets the National Institute on Aging and the Alzheimer's Association (NIA-AA) clinical criteria for mild cognitive impairment or probable AD, and have:

  * Clinical Dementia Rating (CDR)-Global Score of 0.5
  * Mini-Mental State Examination (MMSE) score of 22 to 30, inclusive
  * Repeatable Battery for the Assessment of Neuropsychological Status-Delayed Memory Index (RBANS - DMI) score of 85 or lower
* Subject has a positive amyloid positron emission tomography (PET) scan.
* Subject has a Modified Hachinski Ischemic Scale (MHIS) score of ≤ 4.
* The subject has an identified, reliable, study partner (e.g., family member).
* If using medications to treat symptoms related to AD, doses must be stable for at least 12 weeks prior to randomization.

Exclusion Criteria:

* Subject has any contraindications or inability to tolerate brain magnetic resonance imaging (MRI), PET scans or lumbar puncture.
* Subject has evidence of any other clinically significant neurological disorder other than early AD.
* In the opinion of the investigator, the subject has any clinically significant or uncontrolled medical or psychiatric illness, or has had an infection requiring medical intervention in the past 30 days.
* Subject has had a myocardial infarction, unstable angina, stroke, transient ischemic attack or required intervention for any of these conditions within 6 months of Screening.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 453 (Actual)
Dates: Start 2017-01-26 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (68):
- United States (38):
  - Banner University of Arizona Medical Center Phoenix /ID# 151536, Phoenix, Arizona
  - Banner Sun Health Res Inst /ID# 151895, Sun City, Arizona
  - Irvine Clinical Research /ID# 162331, Irvine, California
  - Ucsd /Id# 152467, La Jolla, California
  - Ray Dolby Brain Health Center /ID# 154965, San Francisco, California
  - Univ California, San Francisco /ID# 152053, San Francisco, California
  - Brain Matters Research /ID# 147796, Delray Beach, Florida
  - Neuropsychiatric Research Center of Southwest Florida /ID# 162332, Fort Myers, Florida
  - Mayo Clinic /ID# 151236, Jacksonville, Florida
  - Synexus Clinical Research US, Inc. /ID# 147804, Orlando, Florida
  - University of South Florida /ID# 151890, Tampa, Florida
  - Synexus Clinical Research US, Inc /ID# 151633, The Villages, Florida
  - Emory Midtown Infectious Disease Clinic /ID# 151492, Atlanta, Georgia
  - Atlanta Center for Medical Research /ID# 151550, Atlanta, Georgia
  - NeuroStudies.net, LLC /ID# 152746, Decatur, Georgia
  - Great Lakes Clinical Trials /ID# 152754, Chicago, Illinois
  - Advocate Lutheran General Hospital /ID# 152052, Park Ridge, Illinois
  - Southern IL Univ School of Med /ID# 151769, Springfield, Illinois
  - Indiana University /ID# 151861, Indianapolis, Indiana
  - University of Kansas Medical Center - Alzheimer's Disease Center /ID# 151554, Fairway, Kansas
  - University of Kentucky Chandler Medical Center /ID# 152753, Lexington, Kentucky
  - Johns Hopkins Bayview Med Cnt /ID# 151893, Baltimore, Maryland
  - Massachusetts General Hospital /ID# 151770, Boston, Massachusetts
  - Brigham and Women's Physicians /ID# 151882, Boston, Massachusetts
  - Hattiesburg Clinic /ID# 202388, Hattiesburg, Mississippi
  - Princeton Medical Institute /ID# 152934, Princeton, New Jersey
  - Scott Research Inc. /ID# 151880, Laurelton, New York
  - North Shore University Hospital /ID# 151632, New Hyde Park, New York
  - Duke Cancer Center /ID# 147828, Durham, North Carolina
  - Oregon Health and Science University /ID# 151690, Portland, Oregon
  - Keystone Clinical Studies LLC /ID# 202305, Plymouth Meeting, Pennsylvania
  - Rhode Island Hospital /ID# 151538, Providence, Rhode Island
  - Vanderbilt University Medical Center /ID# 154547, Nashville, Tennessee
  - Kerwin Research Center /ID# 147815, Dallas, Texas
  - Houston Methodist Hospital /ID# 154810, Houston, Texas
  - McGovern Medical School /ID# 204860, Houston, Texas
  - University of Utah /ID# 151858, Salt Lake City, Utah
  - Integrated Neurology Services /ID# 154863, Alexandria, Virginia
- Australia (6):
  - The Kinghorn Cancer Centre /ID# 152632, Darlinghurst, New South Wales
  - Griffith University /ID# 152635, Southport, Queensland
  - Austin Health /ID# 152637, Heidelberg, Victoria
  - The Royal Melbourne Hospital /ID# 202633, Parkville, Victoria
  - Australian Alzheimer's Res Fou /ID# 152634, Nedlands, Western Australia
  - Neurodegenerative Disorders Research /ID# 152826, West Perth, Western Australia
- Belgium (3):
  - UCL Saint-Luc /ID# 152847, Woluwe-Saint-Lambert, Brussels Capital
  - Universitair Ziekenhuis Leuven /ID# 152642, Leuven, Vlaams-Brabant
  - Groupe Sante CHC - Clinique du MontLegia /ID# 152846, Liège
- Canada (2):
  - Parkwood Institute /ID# 164204, London, Ontario
  - Toronto Memory Program /ID# 147863, Toronto, Ontario
- Rigshospitalet /ID# 153192, Copenhagen Ø, Capital Region, Denmark
- Finland (2):
  - Clinical Research Services Turku /ID# 152845, Turku, Southwest Finland
  - Ita-Suomen Yliopisto /ID# 152959, Kuopio
- Italy (7):
  - AOU di Modena /ID# 152394, Modena, Emilia-Romagna
  - Policlinico Agostino Gemelli /ID# 152396, Rome, Lazio
  - Duplicate_AOU Policlinico Umberto I /ID# 163144, Rome, Lazio
  - Azienda Ospedaliera di Perugia /ID# 152397, Perugia, Umbria
  - IRCCS Istituto Centro San Giovanni di Dio Fatebenefratelli /ID# 152395, Brescia
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico /ID# 152401, Milan
  - ASST Grande Ospedale Metropolitano Niguarda /ID# 152391, Milan
- Universitair Medisch Centrum Utrecht /ID# 163576, Utrecht, Netherlands
- CGM Research Trust /ID# 152827, Burwood, New Zealand
- Spain (5):
  - Fundacion CITA Alzheimer Fundazioa /ID# 152645, Donostia / San Sebastian, Basque Country
  - Fundacio ACE /ID# 152643, Barcelona
  - Hospital Clinic de Barcelona /ID# 152646, Barcelona
  - Hospital Clinico Universitario San Carlos /ID# 153703, Madrid
  - Hospital Universitario 12 de Octubre /ID# 152647, Madrid
- Sweden (2):
  - Karolinska University Hospital Huddinge /ID# 156705, Stockholm, Stockholm County
  - Sahlgrenska University Hospital Molndal /ID# 154465, Mölndal, Västra Götaland County

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing, please refer to the link below.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Use Agreement (DUA). For more information on the process, or to submit a request, visit the following link.
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Derived] Wang D, Florian H, Lynch SY, Robieson W, Zhuang R, Kusiak C, Ross JL, Walsh JR, Graff O. Using AI-generated digital twins to boost clinical trial efficiency in Alzheimer's disease. Alzheimers Dement (N Y). 2025 Nov 22;11(4):e70181. doi: 10.1002/trc2.70181. eCollection 2025 Oct-Dec. PMID 41281734

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | ABBV-8E12 300 mg | ABBV-8E12 1000 mg | ABBV-8E12 2000 mg
Started | 116 | 108 | 116 | 113
Completed | 99 | 93 | 105 | 95
Not Completed | 17 | 15 | 11 | 18
Not completed — Adverse Event | 3 | 6 | 5 | 4
Not completed — Withdrawal by Subject | 9 | 4 | 6 | 11
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — COVID-19 Logistical Restrictions | 1 | 2 | 0 | 0
Not completed — Other, Not Specified | 4 | 2 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | ABBV-8E12 300 mg | ABBV-8E12 1000 mg | ABBV-8E12 2000 mg | Total
Number analyzed (Participants) | 116 | 108 | 116 | 113 | 453
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 15 | 24 | 17 | 29 | 85
  >= 65 years | 101 | 84 | 99 | 84 | 368
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 45 | 60 | 59 | 234
  Male | 46 | 63 | 56 | 54 | 219
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 3 | 0 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 1
  Black or African American | 2 | 3 | 1 | 1 | 7
  White | 111 | 102 | 113 | 111 | 437
  More than one race | 1 | 0 | 1 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 6 | 4 | 3 | 17
  None | 112 | 102 | 112 | 110 | 436
Clinical Dementia Rating Scale - Sum of Boxes (CDR-SB) Score [Mean (Standard Deviation); unit: score on a scale] — The CDR-SB is a numeric scale used to quantify the severity of symptoms of dementia. A qualified health professional assesses a participant's cognitive and functional performance in 6 areas: memory, orientation, judgment and problem solving, community affairs, home and hobbies, and personal care. The CDR scale gives a score from 0 to 3 for each of the 6 areas, with a lower value being desirable. The sum of these 6 areas, the CDR-SB score, can range from 0 to 18, with a lower value being desirable.
  score on a scale | 3.0 (1.22) | 3.0 (1.12) | 3.1 (1.24) | 2.9 (1.14) | 3.0 (1.18)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Over Time in CDR-SB Score
Description: The CDR-SB is a numeric scale used to quantify the severity of symptoms of dementia. A qualified health professional assesses a participant's cognitive and functional performance in 6 areas: memory, orientation, judgment and problem solving, community affairs, home and hobbies, and personal care. The CDR scale gives a score from 0 to 3 for each of the 6 areas, with a lower value being desirable. The sum of these 6 areas, the CDR-SB score, can range from 0 to 18, with a lower value being desirable.
Time Frame: Baseline, Week 24, Week 48, Week 72, Week 96
Population: Intent-to-Treat Data Set: all randomized participants who received at least 1 dose of study drug. Participants with an assessment at given time point.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | ABBV-8E12 300 mg | ABBV-8E12 1000 mg | ABBV-8E12 2000 mg
Number analyzed (Participants) | 116 | 108 | 116 | 113
score on a scale
  Change to Week 24: number analyzed (Participants) | 110 | 108 | 116 | 113
  Change to Week 24 | 0.60 (0.125) | 0.66 (0.129) | 0.44 (0.125) | 0.63 (0.130)
  Change to Week 48: number analyzed (Participants) | 105 | 97 | 105 | 98
  Change to Week 48 | 1.06 (0.155) | 1.15 (0.161) | 1.05 (0.154) | 0.99 (0.161)
  Change to Week 72: number analyzed (Participants) | 100 | 93 | 101 | 95
  Change to Week 72 | 1.90 (0.213) | 1.88 (0.220) | 1.85 (0.212) | 1.81 (0.219)
  Change to Week 96: number analyzed (Participants) | 85 | 85 | 91 | 81
  Change to Week 96 | 2.54 (0.271) | 2.47 (0.277) | 2.48 (0.267) | 2.70 (0.279)
Statistical Analysis 1: Comparison: Placebo vs ABBV-8E12 300 mg; Week 24; Test type: Superiority; p = 0.740, repeated measures model — The statistical model: CDR change from baseline = baseline + treatment + site + visit + baseline*visit + treatment*visit; variance-covariance structure = Unstructured; Least Squares (LS) Mean of Difference = 0.06, 95% CI 2-sided [-0.291 to 0.409], Standard Error of Mean 0.178
Statistical Analysis 2: Comparison: Placebo vs ABBV-8E12 300 mg; Week 24; Test type: Superiority; Effect size/pooled SD = -0.04, Standard Deviation 1.38 — Effect size at a specific visit is calculated as LS mean difference (placebo - 8E12) divided by pooled standard deviation of change scores for a ABBV-8E12 dose and placebo at that visit
Statistical Analysis 3: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 24; Test type: Superiority; p = 0.367, repeated measures model — [p-value comment as in outcome 1, analysis 1]; LS Mean of Difference = -0.16, 95% CI 2-sided [-0.504 to 0.187], Standard Error of Mean 0.176
Statistical Analysis 4: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 24; Test type: Superiority; Effect size/pooled SD = 0.12, Standard Deviation 1.33 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 24; Test type: Superiority; p = 0.843, repeated measures model — [p-value comment as in outcome 1, analysis 1]; LS Mean of Difference = 0.04, 95% CI 2-sided [-0.318 to 0.389], Standard Error of Mean 0.180
Statistical Analysis 6: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 24; Test type: Superiority; Effect size/pooled SD = -0.03, Standard Deviation 1.37 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 7: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; p = 0.703, repeated measures model — [p-value comment as in outcome 1, analysis 1]; LS Mean of Difference = 0.08, 95% CI 2-sided [-0.351 to 0.520], Standard Error of Mean 0.222
Statistical Analysis 8: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; Effect size/pooled SD = -0.05, Standard Deviation 1.62 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 9: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; p = 0.947, repeated measures model — [p-value comment as in outcome 1, analysis 1]; LS Mean of Difference = -0.01, 95% CI 2-sided [-0.442 to 0.413], Standard Error of Mean 0.218
Statistical Analysis 10: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = -0.01, Standard Deviation 1.69 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 11: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Superiority; p = 0.732, repeated measures model — [p-value comment as in outcome 1, analysis 1]; LS Mean of Difference = -0.08, 95% CI 2-sided [-0.514 to 0.361], Standard Error of Mean 0.222
Statistical Analysis 12: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.05, Standard Deviation 1.51 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 13: Comparison: Placebo vs ABBV-8E12 300 mg; Week 72; Test type: Superiority; p = 0.939, repeated measures model — [p-value comment as in outcome 1, analysis 1]; LS Mean of Difference = -0.02, 95% CI 2-sided [-0.623 to 0.576], Standard Error of Mean 0.305
Statistical Analysis 14: Comparison: Placebo vs ABBV-8E12 300 mg; Week 72; Test type: Superiority; Effect size/pooled SD = 0.01, Standard Deviation 2.19 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 15: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 72; Test type: Superiority; p = 0.872, repeated measures model — [p-value comment as in outcome 1, analysis 1]; LS Mean of Difference = -0.05, 95% CI 2-sided [-0.637 to 0.540], Standard Error of Mean 0.299
Statistical Analysis 16: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 72; Test type: Superiority; Effect size/pooled SD = 0.02, Standard Deviation 2.27 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 17: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 72; Test type: Superiority; p = 0.773, repeated measures model — [p-value comment as in outcome 1, analysis 1]; LS Mean of Difference = -0.09, 95% CI 2-sided [-0.688 to 0.512], Standard Error of Mean 0.305
Statistical Analysis 18: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 72; Test type: Superiority; Effect size/pooled SD = 0.04, Standard Deviation 2.13 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 19: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; p = 0.848, repeated measures model — [p-value comment as in outcome 1, analysis 1]; LS Mean of Difference = -0.07, 95% CI 2-sided [-0.834 to 0.686], Standard Error of Mean 0.387
Statistical Analysis 20: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; Effect size/pooled SD = 0.03, Standard Deviation 2.64 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 21: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; p = 0.869, repeated measures model — [p-value comment as in outcome 1, analysis 1]; LS Mean of Difference = -0.06, 95% CI 2-sided [-0.810 to 0.684], Standard Error of Mean 0.380
Statistical Analysis 22: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = 0.02, Standard Deviation 2.75 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 23: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; p = 0.679, repeated measures model — [p-value comment as in outcome 1, analysis 1]; LS Mean of Difference = 0.16, 95% CI 2-sided [-0.603 to 0.925], Standard Error of Mean 0.389
Statistical Analysis 24: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = -0.06, Standard Deviation 2.72 — [estimate comment as in outcome 1, analysis 2]

2. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: A TEAE was defined as an adverse event (AE) that began on or after the first study drug dose date and no more than 20 weeks after the last dose of study drug. An adverse event (AE) was defined as any untoward medical occurrence which does not necessarily have a causal relationship with this treatment. Serious AEs (SAEs) were defined as an event that results in death, is life-threatening, results in hospitalization or prolongs hospitalization, is a congenital abnormality, results in persistent or significant disability/incapacity, or is an important medical event. Events were rated in severity as mild, moderate, or severe, and were categorized as having a reasonable possibility or no reasonable possibility of relationship to study drug.
Time Frame: From first dose of study drug up to last dose of study drug plus 20 weeks (up to Week 112)
Population: Safety Dataset: participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Placebo | ABBV-8E12 300 mg | ABBV-8E12 1000 mg | ABBV-8E12 2000 mg
Number analyzed (Participants) | 116 | 108 | 116 | 113
participants
  Any TEAE | 108 | 94 | 108 | 104
  Severe TEAE | 12 | 13 | 14 | 11
  TEAE With a Reasonable Possibility to Study Drug | 28 | 32 | 31 | 33
  SAE | 26 | 19 | 22 | 17
  TEAE Leading to Discontinuation of Study Drug | 4 | 6 | 6 | 4
  Fatal TEAE | 1 | 2 | 2 | 1
  All Deaths | 1 | 2 | 2 | 1

3. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) for ABBV-8E12 Over the Dosing Interval After the First and Fourth Doses
Time Frame: Day 1 (Dose 1): Pre-infusion, post-infusion (within 15 minutes), 1 and 2 hours post-infusion; Days 5 and 15. Day 85 (Dose 4): Pre-infusion (0 hour), post-infusion (within 15 minutes) and 1 and 2 hours post-infusion; Days 89 and 99.
Population: Intensive Pharmacokinetic Cohort: Among the first 48 participants enrolled in the study, those who received ABBV-8E12 and had an evaluable PK assessment at given time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | ABBV-8E12 300 mg | ABBV-8E12 1000 mg | ABBV-8E12 2000 mg
Number analyzed (Participants) | 12 | 17 | 9
µg/mL
  First Dosing Interval | 108 (28) | 284 (21) | 528 (27)
  Fourth Dosing Interval: number analyzed (Participants) | 11 | 17 | 8
  Fourth Dosing Interval | 168 (23) | 426 (20) | 806 (37)

4. Secondary Outcome: Time to Cmax (Tmax) for ABBV-8E12 Over the Dosing Interval After the First and Fourth Doses
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Median (Full Range); unit: hours
Arm/Group | ABBV-8E12 300 mg | ABBV-8E12 1000 mg | ABBV-8E12 2000 mg
Number analyzed (Participants) | 12 | 17 | 9
hours
  First Dosing Interval | 3 [1.8 to 4.2] | 2.5 [1.3 to 4.2] | 2.7 [1.7 to 3.6]
  Fourth Dosing Interval: number analyzed (Participants) | 11 | 17 | 8
  Fourth Dosing Interval | 2.4 [1.1 to 4.1] | 2.5 [1.7 to 4.3] | 2.3 [1.7 to 3.6]

5. Secondary Outcome: Serum Concentration at the End of a Dose Interval (Ctrough) for ABBV-8E12 Over the Dosing Interval After the First and Fourth Doses
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | ABBV-8E12 300 mg | ABBV-8E12 1000 mg | ABBV-8E12 2000 mg
Number analyzed (Participants) | 12 | 17 | 9
µg/mL
  First Dosing Interval | 28.6 (22) | 75.1 (33) | 163 (26)
  Fourth Dosing Interval: number analyzed (Participants) | 11 | 17 | 8
  Fourth Dosing Interval | 56.4 (25) | 182 (29) | 320 (36)

6. Secondary Outcome: Half-Life (T1/2) for ABBV-8E12 Over the Dosing Interval After the First and Fourth Doses
Description: Harmonic mean is presented in the data table.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: days
Arm/Group | ABBV-8E12 300 mg | ABBV-8E12 1000 mg | ABBV-8E12 2000 mg
Number analyzed (Participants) | 12 | 17 | 9
days
  First Dosing Interval | 22.0 (17.2) | 19.4 (8.87) | 33.2 (10.5)
  Fourth Dosing Interval: number analyzed (Participants) | 11 | 17 | 8
  Fourth Dosing Interval | 19.6 (6.09) | 24.0 (16.6) | 37.5 (13.5)

7. Secondary Outcome: Area Under the Concentration-Time Curve From Dosing (Time 0) to Day 28 (AUC0-28) for ABBV-8E12 Over the Dosing Interval After the First and Fourth Doses
Description: * The AUC0-28 for Dose 1 included the following timepoints: pre-infusion, post-infusion (within 15 min), 1 and 2 hours post-infusion, Day 5, Day 15 and Day 29 (trough level before Dose 2).
  * The AUC0-28 for Dose 4 included the following timepoints: Day 85 pre-infusion, post-infusion (within 15 min), 1 and 2 hours post-infusion, Day 89, Day 99 and Day 113 (trough level before Dose 5).
Time Frame: Day 1 (Dose 1): pre-infusion, up to Day 29 (trough level before Dose 2). Day 85 (Dose 4): pre-infusion, up to Day 113 (trough level before Dose 5). See Outcome Measure description above for complete time point details.
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg.day/mL
Arm/Group | ABBV-8E12 300 mg | ABBV-8E12 1000 mg | ABBV-8E12 2000 mg
Number analyzed (Participants) | 12 | 17 | 9
µg.day/mL
  First Dosing Interval | 2520 (28) | 6090 (37) | 14800 (25)
  Fourth Dosing Interval: number analyzed (Participants) | 11 | 17 | 8
  Fourth Dosing Interval | 4230 (33) | 13100 (36) | 30200 (36)

8. Secondary Outcome: Cmax/Dose for ABBV-8E12 Over the Dosing Interval After the First and Fourth Doses
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL/mg
Arm/Group | ABBV-8E12 300 mg | ABBV-8E12 1000 mg | ABBV-8E12 2000 mg
Number analyzed (Participants) | 12 | 17 | 9
µg/mL/mg
  First Dosing Interval | 0.359 (28) | 0.284 (21) | 0.264 (27)
  Fourth Dosing Interval: number analyzed (Participants) | 11 | 17 | 8
  Fourth Dosing Interval | 0.561 (23) | 0.426 (20) | 0.403 (37)

9. Secondary Outcome: AUC0-28/Dose for ABBV-8E12 Over the Dosing Interval After the First and Fourth Doses
Description: * The AUC0-28/dose for Dose 1 included the following timepoints: pre-infusion, post-infusion (within 15 min), 1 and 2 hours post-infusion, Day 5, Day 15 and Day 29 (trough level before Dose 2).
  * The AUC0-28/dose for Dose 4 included the following timepoints: Day 85 pre-infusion, post-infusion (within 15 min), 1 and 2 hours post-infusion, Day 89, Day 99 and Day 113 (trough level before Dose 5).
Time Frame: as for outcome 7
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg.day/mL/mg
Arm/Group | ABBV-8E12 300 mg | ABBV-8E12 1000 mg | ABBV-8E12 2000 mg
Number analyzed (Participants) | 12 | 17 | 9
µg.day/mL/mg
  First Dosing Interval | 8.40 (28) | 6.09 (37) | 7.41 (25)
  Fourth Dosing Interval: number analyzed (Participants) | 11 | 17 | 8
  Fourth Dosing Interval | 14.1 (33) | 13.1 (36) | 15.1 (36)

10. Secondary Outcome: Change From Baseline Over Time in Alzheimer's Disease Assessment Scale (14-Item) Cognition Portion (ADAS-Cog-14) Total Score
Description: The ADAS-Cog was designed to assess the cognitive impairments most common in AD. The ADAS-Cog-14 includes the original 11 items from the ADAS-Cog-11 [1. Spoken language ability, 2. Comprehension of spoken language, 3. Recall of test instructions, 4. Word-findings difficulty in spontaneous speech, 5. Following commands, 6. Naming objects and fingers, 7. Constructional praxis, 8. Ideational praxis, 9. Orientation, 10. Word-recall task, 11. Word-recognition task] and includes 3 additional tasks [12. Number cancellation task, 13. Delayed word recall task, 14. Executive functioning], for increased sensitivity in mild cognitive impairment (MCI) patients. The Total Score of the ADAS-Cog-14 ranges from 0 to 90, with a higher score representing greater impairment.
Time Frame: Baseline, Week 24, Week 48, Week 72, Week 96
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | ABBV-8E12 300 mg | ABBV-8E12 1000 mg | ABBV-8E12 2000 mg
Number analyzed (Participants) | 116 | 108 | 116 | 113
score on a scale
  Change at Week 24: number analyzed (Participants) | 104 | 103 | 110 | 99
  Change at Week 24 | 1.82 (0.492) | 1.42 (0.498) | 0.56 (0.480) | 1.86 (0.503)
  Change at Week 48: number analyzed (Participants) | 98 | 89 | 102 | 87
  Change at Week 48 | 4.50 (0.621) | 3.51 (0.642) | 3.42 (0.605) | 4.03 (0.647)
  Change at Week 72: number analyzed (Participants) | 91 | 88 | 92 | 85
  Change at Week 72 | 5.26 (0.718) | 4.78 (0.730) | 5.00 (0.706) | 6.37 (0.738)
  Change at Week 96: number analyzed (Participants) | 72 | 78 | 77 | 64
  Change at Week 96 | 8.43 (0.898) | 7.99 (0.891) | 7.84 (0.872) | 9.46 (0.935)
Statistical Analysis 1: Comparison: Placebo vs ABBV-8E12 300 mg; Week 24; Test type: Superiority; p = 0.562, repeated measures model — The statistical model: ADAS-Cog change from baseline = baseline + treatment + site + visit + baseline*visit + treatment*visit; variance-covariance structure = Unstructured; LS Mean of Difference = -0.40, 95% CI 2-sided [-1.764 to 0.960], Standard Error of Mean 0.693
Statistical Analysis 2: Comparison: Placebo vs ABBV-8E12 300 mg; Week 24; Test type: Superiority; Effect size/pooled SD = 0.08, Standard Deviation 4.92 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 24; Test type: Superiority; p = 0.066, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -1.26, 95% CI 2-sided [-2.602 to 0.081], Standard Error of Mean 0.682
Statistical Analysis 4: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 24; Test type: Superiority; Effect size/pooled SD = 0.25, Standard Deviation 5.08 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 24; Test type: Superiority; p = 0.962, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = 0.03, 95% CI 2-sided [-1.343 to 1.410], Standard Error of Mean 0.700
Statistical Analysis 6: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 24; Test type: Superiority; Effect size/pooled SD = -0.01, Standard Deviation 5.33 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 7: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; p = 0.265, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.99, 95% CI 2-sided [-2.734 to 0.755], Standard Error of Mean 0.887
Statistical Analysis 8: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.16, Standard Deviation 6.32 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 9: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; p = 0.212, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -1.08, 95% CI 2-sided [-2.775 to 0.618], Standard Error of Mean 0.863
Statistical Analysis 10: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.17, Standard Deviation 6.29 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 11: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Superiority; p = 0.602, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.47, 95% CI 2-sided [-2.223 to 1.290], Standard Error of Mean 0.893
Statistical Analysis 12: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.07, Standard Deviation 6.35 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 13: Comparison: Placebo vs ABBV-8E12 300 mg; Week 72; Test type: Superiority; p = 0.635, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.48, 95% CI 2-sided [-2.489 to 1.519], Standard Error of Mean 1.019
Statistical Analysis 14: Comparison: Placebo vs ABBV-8E12 300 mg; Week 72; Test type: Superiority; Effect size/pooled SD = 0.08, Standard Deviation 6.31 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 15: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 72; Test type: Superiority; p = 0.795, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.26, 95% CI 2-sided [-2.233 to 1.712], Standard Error of Mean 1.003
Statistical Analysis 16: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 72; Test type: Superiority; Effect size/pooled SD = 0.04, Standard Deviation 7.02 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 17: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 72; Test type: Superiority; p = 0.281, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = 1.11, 95% CI 2-sided [-0.910 to 3.128], Standard Error of Mean 1.027
Statistical Analysis 18: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 72; Test type: Superiority; Effect size/pooled SD = -0.16, Standard Deviation 7.02 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 19: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; p = 0.729, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.44, 95% CI 2-sided [-2.918 to 2.043], Standard Error of Mean 1.261
Statistical Analysis 20: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; Effect size/pooled SD = 0.06, Standard Deviation 7.40 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 21: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; p = 0.636, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.59, 95% CI 2-sided [-3.047 to 1.863], Standard Error of Mean 1.248
Statistical Analysis 22: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = 0.08, Standard Deviation 7.46 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 23: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; p = 0.427, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = 1.03, 95% CI 2-sided [-1.515 to 3.575], Standard Error of Mean 1.294
Statistical Analysis 24: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = -0.13, Standard Deviation 7.90 — [estimate comment as in outcome 1, analysis 2]

11. Secondary Outcome: Change From Baseline Over Time in ADAS-Cog-14 Comprehension of Spoken Language Score
Description: The ADAS-Cog was designed to assess the cognitive impairments most common in AD. The ADAS-Cog-14 includes the original 11 items from the ADAS-Cog-11 [1. Spoken language ability, 2. Comprehension of spoken language, 3. Recall of test instructions, 4. Word-findings difficulty in spontaneous speech, 5. Following commands, 6. Naming objects and fingers, 7. Constructional praxis, 8. Ideational praxis, 9. Orientation, 10. Word-recall task, 11. Word-recognition task] and includes 3 additional tasks [12. Number cancellation task, 13. Delayed word recall task, 14. Executive functioning], for increased sensitivity in MCI patients. The Comprehension of Spoken Language score of the ADAS-Cog-14 ranges from 0 to 5, with a higher score representing greater impairment.
Time Frame: Baseline, Week 24, Week 48, Week 72, Week 96
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | ABBV-8E12 300 mg | ABBV-8E12 1000 mg | ABBV-8E12 2000 mg
Number analyzed (Participants) | 116 | 108 | 116 | 113
score on a scale
  Change at Week 24: number analyzed (Participants) | 110 | 106 | 113 | 102
  Change at Week 24 | 0.01 (0.038) | 0.03 (0.038) | 0.04 (0.037) | 0.08 (0.039)
  Change at Week 48: number analyzed (Participants) | 102 | 92 | 105 | 93
  Change at Week 48 | 0.03 (0.044) | 0.09 (0.046) | 0.07 (0.044) | 0.12 (0.046)
  Change at Week 72: number analyzed (Participants) | 100 | 92 | 96 | 95
  Change at Week 72 | 0.17 (0.064) | 0.11 (0.066) | 0.14 (0.064) | 0.31 (0.066)
  Change at Week 96: number analyzed (Participants) | 81 | 81 | 87 | 76
  Change at Week 96 | 0.30 (0.083) | 0.26 (0.083) | 0.19 (0.080) | 0.29 (0.085)
Statistical Analysis 1: Comparison: Placebo vs ABBV-8E12 300 mg; Week 24; Test type: Superiority; p = 0.690, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = 0.02, 95% CI 2-sided [-0.083 to 0.126], Standard Error of Mean 0.053
Statistical Analysis 2: Comparison: Placebo vs ABBV-8E12 300 mg; Week 24; Test type: Superiority; Effect size/pooled SD = -0.05, Standard Deviation 0.39 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 24; Test type: Superiority; p = 0.595, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = 0.03, 95% CI 2-sided [-0.075 to 0.131], Standard Error of Mean 0.052
Statistical Analysis 4: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 24; Test type: Superiority; Effect size/pooled SD = -0.08, Standard Deviation 0.36 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 24; Test type: Superiority; p = 0.201, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = 0.07, 95% CI 2-sided [0.037 to 0.175], Standard Error of Mean 0.054
Statistical Analysis 6: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 24; Test type: Superiority; Effect size/pooled SD = -0.15, Standard Deviation 0.45 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 7: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; p = 0.361, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = 0.06, 95% CI 2-sided [-0.067 to 0.184], Standard Error of Mean 0.064
Statistical Analysis 8: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; Effect size/pooled SD = -0.12, Standard Deviation 0.49 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 9: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; p = 0.522, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = 0.04, 95% CI 2-sided [-0.082 to 0.162], Standard Error of Mean 0.062 — The statistical model: ADAS-Cog change from baseline = baseline + treatment + site + visit + baseline*visit + treatment*visit; variance-covariance structure = Unstructured
Statistical Analysis 10: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = -0.10, Standard Deviation 0.41 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 11: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Superiority; p = 0.147, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = 0.09, 95% CI 2-sided [-0.033 to 0.219], Standard Error of Mean 0.064
Statistical Analysis 12: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = -0.17, Standard Deviation 0.53 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 13: Comparison: Placebo vs ABBV-8E12 300 mg; Week 72; Test type: Superiority; p = 0.492, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.06, 95% CI 2-sided [-0.243 to 0.117], Standard Error of Mean 0.091
Statistical Analysis 14: Comparison: Placebo vs ABBV-8E12 300 mg; Week 72; Test type: Superiority; Effect size/pooled SD = 0.11, Standard Deviation 0.57 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 15: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 72; Test type: Superiority; p = 0.691, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.04, 95% CI 2-sided [-0.213 to 0.141], Standard Error of Mean 0.090
Statistical Analysis 16: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 72; Test type: Superiority; Effect size/pooled SD = 0.06, Standard Deviation 0.60 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 17: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 72; Test type: Superiority; p = 0.135, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = 0.14, 95% CI 2-sided [-0.043 to 0.317], Standard Error of Mean 0.091
Statistical Analysis 18: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 72; Test type: Superiority; Effect size/pooled SD = -0.19, Standard Deviation 0.74 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 19: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; p = 0.713, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.04, 95% CI 2-sided [-0.273 to 0.187], Standard Error of Mean 0.117
Statistical Analysis 20: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; Effect size/pooled SD = 0.06, Standard Error of Mean 0.74 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 21: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; p = 0.318, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.11, 95% CI 2-sided [-0.341 to 0.111], Standard Error of Mean 0.115
Statistical Analysis 22: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = 0.14, Standard Deviation 0.80 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 23: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; p = 0.927, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.01, 95% CI 2-sided [-0.244 to 0.222], Standard Error of Mean 0.119
Statistical Analysis 24: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = 0.01, Standard Deviation 0.84 — [estimate comment as in outcome 1, analysis 2]

12. Secondary Outcome: Change From Baseline Over Time in ADAS-Cog-14 Constructional Praxis Score
Description: The ADAS-Cog was designed to assess the cognitive impairments most common in AD. The ADAS-Cog-14 includes the original 11 items from the ADAS-Cog-11 [1. Spoken language ability, 2. Comprehension of spoken language, 3. Recall of test instructions, 4. Word-findings difficulty in spontaneous speech, 5. Following commands, 6. Naming objects and fingers, 7. Constructional praxis, 8. Ideational praxis, 9. Orientation, 10. Word-recall task, 11. Word-recognition task] and includes 3 additional tasks [12. Number cancellation task, 13. Delayed word recall task, 14. Executive functioning], for increased sensitivity in MCI patients. The Constructional Praxis Score of the ADAS-Cog-14 ranges from 0 to 5, with a higher score representing greater impairment.
Time Frame: Baseline, Week 24, Week 48, Week 72, Week 96
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | ABBV-8E12 300 mg | ABBV-8E12 1000 mg | ABBV-8E12 2000 mg
Number analyzed (Participants) | 116 | 108 | 116 | 113
score on a scale
  Change at Week 24: number analyzed (Participants) | 110 | 106 | 113 | 102
  Change at Week 24 | 0.11 (0.057) | 0.05 (0.058) | -0.02 (0.056) | 0.09 (0.059)
  Change at Week 48: number analyzed (Participants) | 102 | 92 | 105 | 93
  Change at Week 48 | 0.07 (0.073) | 0.23 (0.077) | 0.17 (0.072) | 0.20 (0.077)
  Change at Week 72: number analyzed (Participants) | 100 | 92 | 96 | 94
  Change at Week 72 | 0.25 (0.069) | 0.22 (0.072) | 0.16 (0.070) | 0.16 (0.071)
  Change at Week 96: number analyzed (Participants) | 80 | 81 | 86 | 75
  Change at Week 96 | 0.41 (0.089) | 0.25 (0.089) | 0.026 (0.086) | 0.33 (0.092)
Statistical Analysis 1: Comparison: Placebo vs ABBV-8E12 300 mg; Week 24; Test type: Superiority; p = 0.456, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.06, 95% CI 2-sided [-0.219 to 0.098], Standard Error of Mean 0.081
Statistical Analysis 2: Comparison: Placebo vs ABBV-8E12 300 mg; Week 24; Test type: Superiority; Effect size/pooled SD = 0.09, Standard Deviation 0.64 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 24; Test type: Superiority; p = 0.093, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.13, 95% CI 2-sided [-0.290 to 0.023], Standard Error of Mean 0.079
Statistical Analysis 4: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 24; Test type: Superiority; Effect size/pooled SD = 0.23, Standard Deviation 0.59 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 24; Test type: Superiority; p = 0.750, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.03, 95% CI 2-sided [-0.187 to 0.135], Standard Error of Mean 0.082
Statistical Analysis 6: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 24; Test type: Superiority; Effect size/pooled SD = 0.04, Standard Deviation 0.63 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 7: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; p = 0.134, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = 0.16, 95% CI 2-sided [-0.049 to 0.366], Standard Error of Mean 0.106
Statistical Analysis 8: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; Effect size/pooled SD = -0.20, Standard Deviation 0.79 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 9: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; p = 0.316, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = 0.10, 95% CI 2-sided [-0.099 to 0.305], Standard Error of Mean 0.103
Statistical Analysis 10: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = -0.14, Standard Deviation 0.72 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 11: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Superiority; p = 0.218, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = 0.13, 95% CI 2-sided [-0.078 to 0.339], Standard Error of Mean 0.106
Statistical Analysis 12: Comparison: ABBV-8E12 2000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = -0.17, Standard Deviation 0.76 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 13: Comparison: Placebo vs ABBV-8E12 300 mg; Week 72; Test type: Superiority; p = 0.799, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.03, 95% CI 2-sided [-0.219 to 0.169], Standard Error of Mean 0.099
Statistical Analysis 14: Comparison: Placebo vs ABBV-8E12 300 mg; Week 72; Test type: Superiority; Effect size/pooled SD = 0.04, Standard Deviation 0.70 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 15: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 72; Test type: Superiority; p = 0.406, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.08, 95% CI 2-sided [-0.273 to 0.111], Standard Error of Mean 0.098
Statistical Analysis 16: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 72; Test type: Superiority; Effect size/pooled SD = 0.11, Standard Deviation 0.74 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 17: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 72; Test type: Superiority; p = 0.363, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.09, 95% CI 2-sided [-0.285 to 0.105], Standard Error of Mean 0.099
Statistical Analysis 18: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 72; Test type: Superiority; Effect size/pooled SD = 0.12, Standard Deviation 0.76 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 19: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; p = 0.220, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.15, 95% CI 2-sided [-0.400 to 0.093], Standard Error of Mean 0.125
Statistical Analysis 20: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; Effect size/pooled SD = 0.18, Standard Deviation 0.85 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 21: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; p = 0.245, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.14, 95% CI 2-sided [-0.386 to 0.099], Standard Error of Mean 0.123
Statistical Analysis 22: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = 0.17, Standard Deviation 0.83 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 23: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; p = 0.569, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.07, 95% CI 2-sided [-0.323 to 0.178], Standard Error of Mean 0.127
Statistical Analysis 24: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = 0.08, Standard Deviation 0.95 — [estimate comment as in outcome 1, analysis 2]

13. Secondary Outcome: Change From Baseline Over Time in ADAS-Cog-14 Commands Score
Description: The ADAS-Cog was designed to assess the cognitive impairments most common in AD. The ADAS-Cog-14 includes the original 11 items from the ADAS-Cog-11 [1. Spoken language ability, 2. Comprehension of spoken language, 3. Recall of test instructions, 4. Word-findings difficulty in spontaneous speech, 5. Following commands, 6. Naming objects and fingers, 7. Constructional praxis, 8. Ideational praxis, 9. Orientation, 10. Word-recall task, 11. Word-recognition task] and includes 3 additional tasks [12. Number cancellation task, 13. Delayed word recall task, 14. Executive functioning], for increased sensitivity in MCI patients. The Commands Score of the ADAS-Cog-14 ranges from 0 to 5, with a higher score representing greater impairment.
Time Frame: Baseline, Week 24, Week 48, Week 72, Week 96
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | ABBV-8E12 300 mg | ABBV-8E12 1000 mg | ABBV-8E12 2000 mg
Number analyzed (Participants) | 116 | 108 | 116 | 113
score on a scale
  Change at Week 24: number analyzed (Participants) | 110 | 106 | 113 | 102
  Change at Week 24 | 0.09 (0.066) | 0.10 (0.067) | 0.09 (0.065) | 0.09 (0.068)
  Change at Week 48: number analyzed (Participants) | 102 | 92 | 105 | 93
  Change at Week 48 | 0.17 (0.072) | 0.12 (0.076) | 0.09 (0.071) | 0.22 (0.075)
  Change at Week 72: number analyzed (Participants) | 100 | 92 | 96 | 95
  Change at Week 72 | 0.09 (0.078) | 0.11 (0.081) | 0.36 (0.079) | 0.21 (0.080)
  Change at Week 96: number analyzed (Participants) | 81 | 81 | 86 | 76
  Change at Week 96 | 0.30 (0.102) | 0.36 (0.103) | 0.40 (0.100) | 0.40 (0.106)
Statistical Analysis 1: Comparison: Placebo vs ABBV-8E12 300 mg; Week 24; Test type: Superiority; p = 0.945, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = 0.01, 95% CI 2-sided [-0.177 to 0.190], Standard Error of Mean 0.093
Statistical Analysis 2: Comparison: Placebo vs ABBV-8E12 300 mg; Week 24; Test type: Superiority; Effect size/pooled SD = -0.01, Standard Deviation 0.86 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 24; Test type: Superiority; p = 0.974, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.00, 95% CI 2-sided [-0.184 to 0.178], Standard Error of Mean 0.092
Statistical Analysis 4: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 24; Test type: Superiority; Effect size/pooled SD = 0.00, Standard Deviation 0.74 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Placebo vs ABBV-8E12 2000 mg; Test type: Superiority; p = 0.963, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.00, 95% CI 2-sided [-0.190 to 0.181], Standard Error of Mean 0.094
Statistical Analysis 6: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 24; Test type: Superiority; Effect size/pooled SD = 0.01, Standard Deviation 0.76 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 7: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; p = 0.625, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.05, 95% CI 2-sided [-0.255 to 0.154], Standard Error of Mean 0.104
Statistical Analysis 8: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.07, Standard Deviation 0.74 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 9: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; p = 0.468, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.07, 95% CI 2-sided [-0.272 to 0.125], Standard Error of Mean 0.101
Statistical Analysis 10: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.10, Standard Deviation 0.71 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 11: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Superiority; p = 0.636, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = 0.05, 95% CI 2-sided [-0.155 to 0.254], Standard Error of Mean 0.104
Statistical Analysis 12: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = -0.06, Standard Deviation 0.88 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 13: Comparison: Placebo vs ABBV-8E12 300 mg; Week 72; Test type: Superiority; p = 0.887, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = 0.02, 95% CI 2-sided [-0.204 to 0.236], Standard Error of Mean 0.112
Statistical Analysis 14: Comparison: Placebo vs ABBV-8E12 300 mg; Week 72; Test type: Superiority; Effect size/pooled SD = -0.02, Standard Deviation 0.84 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 15: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 72; Test type: Superiority; p = 0.016, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = 0.27, 95% CI 2-sided [0.051 to 0.486], Standard Error of Mean 0.111
Statistical Analysis 16: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 72; Test type: Superiority; Effect size/pooled SD = -0.33, Standard Deviation 0.80 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 17: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 72; Test type: Superiority; p = 0.272, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = 0.12, 95% CI 2-sided [-0.097 to 0.342], Standard Error of Mean 0.112
Statistical Analysis 18: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 72; Test type: Superiority; Effect size/pooled SD = -0.15, Standard Deviation 0.81 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 19: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; p = 0.671, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = 0.06, 95% CI 2-sided [-0.223 to 0.347], Standard Error of Mean 0.145
Statistical Analysis 20: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; Effect size/pooled SD = -0.07, Standard Deviation 0.88 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 21: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; p = 0.493, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = 0.10, 95% CI 2-sided [-0.183 to 0.378], Standard Error of Mean 0.143
Statistical Analysis 22: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = -0.11, Standard Deviation 0.92 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 23: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; p = 0.501, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = 0.10, 95% CI 2-sided [-0.190 to 0.387], Standard Error of Mean 0.147
Statistical Analysis 24: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = -0.10, Standard Deviation 0.98 — [estimate comment as in outcome 1, analysis 2]

14. Secondary Outcome: Change From Baseline Over Time in ADAS-Cog-14 Delayed Word Recall Score
Description: The ADAS-Cog was designed to assess the cognitive impairments most common in AD. The ADAS-Cog-14 includes the original 11 items from the ADAS-Cog-11 [1. Spoken language ability, 2. Comprehension of spoken language, 3. Recall of test instructions, 4. Word-findings difficulty in spontaneous speech, 5. Following commands, 6. Naming objects and fingers, 7. Constructional praxis, 8. Ideational praxis, 9. Orientation, 10. Word-recall task, 11. Word-recognition task] and includes 3 additional tasks [12. Number cancellation task, 13. Delayed word recall task, 14. Executive functioning], for increased sensitivity in MCI patients. The Delayed Word Recall Score of the ADAS-Cog-14 ranges from 0 to 10, with a higher score representing greater impairment.
Time Frame: Baseline, Week 24, Week 48, Week 72, Week 96
Population: Intent-to-Treat Data Set: all randomized participants who received at least 1 dose of study drug. Participants with an assessment at baseline and given time point.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | ABBV-8E12 300 mg | ABBV-8E12 1000 mg | ABBV-8E12 2000 mg
Number analyzed (Participants) | 115 | 108 | 116 | 113
score on a scale
  Change at Week 24: number analyzed (Participants) | 109 | 106 | 113 | 102
  Change at Week 24 | 0.11 (0.133) | 0.17 (0.135) | -0.04 (0.131) | -0.09 (0.137)
  Change at Week 48: number analyzed (Participants) | 101 | 92 | 105 | 93
  Change at Week 48 | 0.41 (0.133) | 0.30 (0.138) | 0.32 (0.131) | 0.27 (0.138)
  Change at Week 72: number analyzed (Participants) | 99 | 92 | 96 | 95
  Change at Week 72 | 0.39 (0.132) | 0.61 (0.136) | 0.52 (0.133) | 0.67 (0.135)
  Change at Week 96: number analyzed (Participants) | 79 | 81 | 86 | 76
  Change at Week 96 | 0.86 (0.135) | 0.80 (0.135) | 0.60 (0.131) | 0.66 (0.138)
Statistical Analysis 1: Comparison: Placebo vs ABBV-8E12 300 mg; Week 24; Test type: Superiority; p = 0.742, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = 0.06, 95% CI 2-sided [-0.307 to 0.431], Standard Error of Mean 0.188
Statistical Analysis 2: Comparison: Placebo vs ABBV-8E12 300 mg; Week 24; Test type: Superiority; Effect size/pooled SD = -0.04, Standard Deviation 1.50 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 24; Test type: Superiority; p = 0.431, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.15, 95% CI 2-sided [-0.511 to 0.218], Standard Error of Mean 0.185
Statistical Analysis 4: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 24; Test type: Superiority; Effect size/pooled SD = 0.10, Standard Deviation 1.50 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 24; Test type: Superiority; p = 0.290, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.20, 95% CI 2-sided [-0.574 to 0.172], Standard Error of Mean 0.190
Statistical Analysis 6: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 24; Test type: Superiority; effect size = 0.13, Standard Deviation 1.51 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 7: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; p = 0.541, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.12, 95% CI 2-sided [-0.492 to 0.258], Standard Error of Mean 0.191
Statistical Analysis 8: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.08, Standard Deviation 1.55 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 9: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; p = 0.617, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.09, 95% CI 2-sided [-0.459 to 0.272], Standard Error of Mean 0.186
Statistical Analysis 10: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.06, Standard Deviation 1.49 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 11: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Superiority; p = 0.457, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.14, 95% CI 2-sided [-0.517 to 0.233], Standard Error of Mean 0.191
Statistical Analysis 12: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.09, Standard Deviation 1.50 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 13: Comparison: Placebo vs ABBV-8E12 300 mg; Week 72; Test type: Superiority; p = 0.245, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = 0.22, 95% CI 2-sided [-0.151 to 0.590], Standard Error of Mean 0.188
Statistical Analysis 14: Comparison: Placebo vs ABBV-8E12 300 mg; Week 72; Test type: Superiority; Effect size/pooled SD = -0.15, Standard Deviation 1.49 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 15: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 72; Test type: Superiority; p = 0.491, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = 0.13, 95% CI 2-sided [-0.238 to 0.496], Standard Error of Mean 0.187
Statistical Analysis 16: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 72; Test type: Superiority; Effect size/pooled SD = -0.08, Standard Deviation 1.60 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 17: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 72; Test type: Superiority; p = 0.132, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = 0.28, 95% CI 2-sided [-0.085 to 0.652], Standard Error of Mean 0.188
Statistical Analysis 18: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 72; Test type: Superiority; Effect size/pooled SD = -0.18, Standard Deviation 1.58 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 19: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; p = 0.751, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.06, 95% CI 2-sided [-0.434 to 0.313], Standard Error of Mean 0.190
Statistical Analysis 20: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; Effect size/pooled SD = 0.04, Standard Deviation 1.53 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 21: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; p = 0.157, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.27, 95% CI 2-sided [-0.635 to 0.103], Standard Error of Mean 0.188
Statistical Analysis 22: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = 0.16, Standard Deviation 1.63 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 23: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; p = 0.283, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.21, 95% CI 2-sided [-0.585 to 0.172], Standard Error of Mean 0.192
Statistical Analysis 24: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 24; Test type: Superiority; Effect size/pooled SD = 0.14, Standard Deviation 1.44 — [estimate comment as in outcome 1, analysis 2]

15. Secondary Outcome: Change From Baseline Over Time in ADAS-Cog-14 Ideational Praxis Score
Description: The ADAS-Cog was designed to assess the cognitive impairments most common in AD. The ADAS-Cog-14 includes the original 11 items from the ADAS-Cog-11 [1. Spoken language ability, 2. Comprehension of spoken language, 3. Recall of test instructions, 4. Word-findings difficulty in spontaneous speech, 5. Following commands, 6. Naming objects and fingers, 7. Constructional praxis, 8. Ideational praxis, 9. Orientation, 10. Word-recall task, 11. Word-recognition task] and includes 3 additional tasks [12. Number cancellation task, 13. Delayed word recall task, 14. Executive functioning], for increased sensitivity in MCI patients. The Ideational Praxis Score of the ADAS-Cog-14 ranges from 0 to 5, with a higher score representing greater impairment.
Time Frame: Baseline, Week 24, Week 48, Week 72, Week 96
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | ABBV-8E12 300 mg | ABBV-8E12 1000 mg | ABBV-8E12 2000 mg
Number analyzed (Participants) | 116 | 108 | 116 | 113
score on a scale
  Change at Week 24: number analyzed (Participants) | 110 | 106 | 112 | 102
  Change at Week 24 | 0.05 (0.057) | 0.13 (0.058) | 0.02 (0.056) | 0.18 (0.059)
  Change at Week 48: number analyzed (Participants) | 102 | 92 | 105 | 93
  Change at Week 48 | 0.21 (0.075) | 0.12 (0.078) | 0.09 (0.073) | 0.16 (0.078)
  Change at Week 72: number analyzed (Participants) | 99 | 92 | 96 | 94
  Change at Week 72 | 0.18 (0.083) | 0.25 (0.086) | 0.21 (0.083) | 0.35 (0.085)
  Change at Week 96: number analyzed (Participants) | 80 | 81 | 86 | 75
  Change at Week 96 | 0.35 (0.111) | 0.26 (0.112) | 0.41 (0.108) | 0.42 (0.114)
Statistical Analysis 1: Comparison: Placebo vs ABBV-8E12 300 mg; Week 24; Test type: Superiority; p = 0.363, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = 0.07, 95% CI 2-sided [-0.085 to 0.231], Standard Error of Mean 0.080
Statistical Analysis 2: Comparison: Placebo vs ABBV-8E12 300 mg; Week 24; Test type: Superiority; Effect size/pooled SD = -0.11, Standard Deviation 0.66 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 24; Test type: Superiority; p = 0.688, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.03, 95% CI 2-sided [-0.188 to 0.124], Standard Error of Mean 0.079
Statistical Analysis 4: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 24; Test type: Superiority; Effect size/pooled SD = 0.05, Standard Deviation 0.64 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 24; Test type: Superiority; p = 0.137, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = 0.12, 95% CI 2-sided [-0.039 to 0.281], Standard Error of Mean 0.081
Statistical Analysis 6: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 24; Test type: Superiority; Effect size/pooled SD = -0.18, Standard Deviation 0.67 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 7: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; p = 0.408, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.09, 95% CI 2-sided [-0.300 to 0.122], Standard Error of Mean 0.107
Statistical Analysis 8: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.10, Standard Deviation 0.89 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 9: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; p = 0.249, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.12, 95% CI 2-sided [-0.325 to 0.085], Standard Error of Mean 0.104
Statistical Analysis 10: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.15, Standard Deviation 0.79 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 11: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Superiority; p = 0.616, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.05, 95% CI 2-sided [-0.265 to 0.157], Standard Error of Mean 0.107
Statistical Analysis 12: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.06, Standard Deviation 0.95 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 13: Comparison: Placebo vs ABBV-8E12 300 mg; Week 72; Test type: Superiority; p = 0.555, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = 0.07, 95% CI 2-sided [-0.163 to 0.304], Standard Error of Mean 0.119
Statistical Analysis 14: Comparison: Placebo vs ABBV-8E12 300 mg; Week 72; Test type: Superiority; Effect size/pooled SD = -0.08, Standard Deviation 0.83 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 15: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 72; Test type: Superiority; p = 0.815, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = 0.03, 95% CI 2-sided [-0.203 to 0.258], Standard Error of Mean 0.117
Statistical Analysis 16: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 72; Test type: Superiority; Effect size/pooled SD = -0.03, Standard Deviation 0.82 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 17: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 72; Test type: Superiority; p = 0.138, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = 0.18, 95% CI 2-sided [-0.057 to 0.409], Standard Error of Mean 0.119
Statistical Analysis 18: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 72; Test type: Superiority; Effect size/pooled SD = -0.20, Standard Deviation 0.89 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 19: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; p = 0.573, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.09, 95% CI 2-sided [-0.397 to 0.220], Standard Error of Mean 0.157
Statistical Analysis 20: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; Effect size/pooled SD = 0.09, Standard Deviation 1.00 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 21: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; p = 0.689, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = 0.06, 95% CI 2-sided [-0.241 to 0.365], Standard Error of Mean 0.154
Statistical Analysis 22: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = -0.06, Standard Error of Mean 1.11 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 23: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; p = 0.662, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = 0.07, 95% CI 2-sided [-0.243 to 0.382], Standard Error of Mean 0.159
Statistical Analysis 24: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = -0.06, Standard Deviation 1.14 — [estimate comment as in outcome 1, analysis 2]

16. Secondary Outcome: Change From Baseline Over Time in ADAS-Cog-14 Maze Task Score
Description: The ADAS-Cog was designed to assess the cognitive impairments most common in AD. The ADAS-Cog-14 includes the original 11 items from the ADAS-Cog-11 [1. Spoken language ability, 2. Comprehension of spoken language, 3. Recall of test instructions, 4. Word-findings difficulty in spontaneous speech, 5. Following commands, 6. Naming objects and fingers, 7. Constructional praxis, 8. Ideational praxis, 9. Orientation, 10. Word-recall task, 11. Word-recognition task] and includes 3 additional tasks [12. Number cancellation task, 13. Delayed word recall task, 14. Executive functioning], for increased sensitivity in MCI patients. The Maze Task Score of the ADAS-Cog-14 ranges from 0 to 5, with a higher score representing greater impairment.
Time Frame: Baseline, Week 24, Week 48, Week 72, Week 96
Population: as for outcome 14
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | ABBV-8E12 300 mg | ABBV-8E12 1000 mg | ABBV-8E12 2000 mg
Number analyzed (Participants) | 114 | 107 | 116 | 112
score on a scale
  Change at Week 24: number analyzed (Participants) | 107 | 104 | 111 | 101
  Change at Week 24 | 0.15 (0.130) | -0.04 (0.132) | -0.20 (0.129) | 0.17 (0.134)
  Change at Week 48: number analyzed (Participants) | 100 | 89 | 104 | 88
  Change at Week 48 | 0.37 (0.147) | 0.07 (0.154) | 0.21 (0.145) | 0.28 (0.155)
  Change at Week 72: number analyzed (Participants) | 97 | 89 | 93 | 88
  Change at Week 72 | 0.32 (0.160) | 0.14 (0.166) | 0.04 (0.162) | 0.40 (0.167)
  Change at Week 96: number analyzed (Participants) | 74 | 80 | 80 | 70
  Change at Week 96 | 0.52 (0.184) | 0.29 (0.181) | 0.60 (0.179) | 0.52 (0.190)
Statistical Analysis 1: Comparison: Placebo vs ABBV-8E12 300 mg; Week 24; Test type: Superiority; p = 0.291, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.19, 95% CI 2-sided [-0.555 to 0.167], Standard Error of Mean 0.184
Statistical Analysis 2: Comparison: Placebo vs ABBV-8E12 300 mg; Week 24; Test type: Superiority; Effect size/pooled SD = 0.13, Standard Deviation 1.48 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 24; Test type: Superiority; p = 0.051, repeated measures model — [p-value comment as in outcome 10, analysis 1]; Effect size/pooled SD = -0.36, 95% CI 2-sided [-0.713 to 0.001], Standard Error of Mean 0.182
Statistical Analysis 4: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 24; Test type: Superiority; Effect size/pooled SD = 0.23, Standard Deviation 1.52 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 24; Test type: Superiority; p = 0.921, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = 0.02, 95% CI 2-sided [-0.346 to 0.383], Standard Error of Mean 0.185
Statistical Analysis 6: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 24; Test type: Superiority; Effect size/pooled SD = -0.01, Standard Deviation 1.53 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 7: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; p = 0.163, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.30, 95% CI 2-sided [-0.711 to 0.120], Standard Error of Mean 0.211
Statistical Analysis 8: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.18, Standard Deviation 1.67 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 9: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; p = 0.424, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.16, 95% CI 2-sided [-0.567 to 0.239], Standard Error of Mean 0.205
Statistical Analysis 10: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.10, Standard Deviation 1.61 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 11: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Superiority; p = 0.664, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.09, 95% CI 2-sided [-0.510 to 0.326], Standard Error of Mean 0.213
Statistical Analysis 12: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.06, Standard Deviation 1.67 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 13: Comparison: Placebo vs ABBV-8E12 300 mg; Week 72; Test type: Superiority; p = 0.417, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.19, 95% CI 2-sided [-0.638 to 0.265], Standard Error of Mean 0.229
Statistical Analysis 14: Comparison: Placebo vs ABBV-8E12 300 mg; Week 72; Test type: Superiority; Effect size/pooled SD = 0.11, Standard Deviation 1.71 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 15: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 72; Test type: Superiority; p = 0.217, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.28, 95% CI 2-sided [-0.727 to 0.166], Standard Error of Mean 0.227
Statistical Analysis 16: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 72; Test type: Superiority; Effect size/pooled SD = 0.17, Standard Deviation 1.68 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 17: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 72; Test type: Superiority; p = 0.753, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = 0.07, 95% CI 2-sided [-0.381 to 0.526], Standard Error of Mean 0.231
Statistical Analysis 18: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 72; Test type: Superiority; Effect size/pooled SD = -0.04, Standard Deviation 1.80 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 19: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; p = 0.362, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.23, 95% CI 2-sided [-0.740 to 0.270], Standard Error of Mean 0.257
Statistical Analysis 20: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; Effect size/pooled SD = 0.14, Standard Deviation 1.62 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 21: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; p = 0.780, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = 0.07, 95% CI 2-sided [-0.432 to 0.575], Standard Error of Mean 0.256
Statistical Analysis 22: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = -0.04, Standard Deviation 1.72 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 23: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; p = 0.974, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.01, 95% CI 2-sided [-0.526 to 0.509], Standard Error of Mean 0.263
Statistical Analysis 24: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = 0.01, Standard Deviation 1.67 — [estimate comment as in outcome 1, analysis 2]

17. Secondary Outcome: Change From Baseline Over Time in ADAS-Cog-14 Number Cancellation Score
Description: The ADAS-Cog was designed to assess the cognitive impairments most common in AD. The ADAS-Cog-14 includes the original 11 items from the ADAS-Cog-11 [1. Spoken language ability, 2. Comprehension of spoken language, 3. Recall of test instructions, 4. Word-findings difficulty in spontaneous speech, 5. Following commands, 6. Naming objects and fingers, 7. Constructional praxis, 8. Ideational praxis, 9. Orientation, 10. Word-recall task, 11. Word-recognition task] and includes 3 additional tasks [12. Number cancellation task, 13. Delayed word recall task, 14. Executive functioning], for increased sensitivity in MCI patients. The Number Cancellation Score of the ADAS-Cog-14 ranges from 0 to 5, with a higher score representing greater impairment.
Time Frame: Baseline, Week 24, Week 48, Week 72, Week 96
Population: as for outcome 14
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | ABBV-8E12 300 mg | ABBV-8E12 1000 mg | ABBV-8E12 2000 mg
Number analyzed (Participants) | 113 | 108 | 115 | 112
score on a scale
  Change at Week 24: number analyzed (Participants) | 107 | 106 | 112 | 100
  Change at Week 24 | 0.33 (0.099) | 0.33 (0.100) | 0.35 (0.097) | 0.32 (0.102)
  Change at Week 48: number analyzed (Participants) | 99 | 92 | 103 | 92
  Change at Week 48 | 0.43 (0.114) | 0.42 (0.118) | 0.42 (0.112) | 0.22 (0.118)
  Change at Week 72: number analyzed (Participants) | 95 | 92 | 93 | 91
  Change at Week 72 | 0.75 (0.115) | 0.68 (0.117) | 0.44 (0.115) | 0.68 (0.118)
  Change at Week 96: number analyzed (Participants) | 76 | 80 | 83 | 70
  Change at Week 96 | 0.87 (0.138) | 0.84 (0.137) | 0.74 (0.133) | 0.77 (0.143)
Statistical Analysis 1: Comparison: Placebo vs ABBV-8E12 300 mg; Week 24; Test type: Superiority; p = 0.976, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = 0.00, 95% CI 2-sided [-0.269 to 0.278], Standard Error of Mean 0.139
Statistical Analysis 2: Comparison: Placebo vs ABBV-8E12 300 mg; Week 24; Test type: Superiority; Effect size/pooled SD = -0.00, Standard Deviation 1.10
Statistical Analysis 3: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 24; Test type: Superiority; p = 0.850, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = 0.03, 95% CI 2-sided [-0.244 to 0.296], Standard Error of Mean 0.137
Statistical Analysis 4: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 24; Test type: Superiority; Effect size/pooled SD = -0.02, Standard Deviation 1.13 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 24; Test type: Superiority; p = 0.981, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.00, 95% CI 2-sided [-0.281 to 0.275], Standard Error of Mean 0.141
Statistical Analysis 6: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 24; Test type: Superiority; Effect size/pooled SD = 0.00, Standard Deviation 1.05 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 7: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; p = 0.989, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.00, 95% CI 2-sided [-0.323 to 0.318], Standard Error of Mean 0.163
Statistical Analysis 8: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.00, Standard Deviation 1.32 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 9: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; p = 0.970, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.01, 95% CI 2-sided [-0.319 to 0.307], Standard Error of Mean 0.159
Statistical Analysis 10: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; effect size = 0.00, Standard Deviation 1.23 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 11: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Superiority; p = 0.215, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.20, 95% CI 2-sided [-0.526 to 0.119], Standard Error of Mean 0.164
Statistical Analysis 12: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.17, Standard Deviation 1.18 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 13: Comparison: Placebo vs ABBV-8E12 300 mg; Week 72; Test type: Superiority; p = 0.665, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.07, 95% CI 2-sided [-0.392 to 0.250], Standard Error of Mean 0.163
Statistical Analysis 14: Comparison: Placebo vs ABBV-8E12 300 mg; Week 72; Test type: Superiority; Effect size/pooled SD = 0.06, Standard Deviation 1.28 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 15: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 72; Test type: Superiority; p = 0.059, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.31, 95% CI 2-sided [-0.625 to 0.012], Standard Error of Mean 0.162
Statistical Analysis 16: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 72; Test type: Superiority; Effect size/pooled SD = 0.28, Standard Deviation 1.11 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 17: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 72; Test type: Superiority; p = 0.663, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.07, 95% CI 2-sided [-0.394 to 0.251], Standard Error of Mean 0.164
Statistical Analysis 18: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 72; Test type: Superiority; Effect size/pooled SD = 0.06, Standard Deviation 1.27 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 19: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; p = 0.866, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.03, 95% CI 2-sided [-0.413 to 0.348], Standard Error of Mean 0.193
Statistical Analysis 20: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; Effect size/pooled SD = 0.03, Standard Deviation 1.23 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 21: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; p = 0.471, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.14, 95% CI 2-sided [-0.514 to 0.238], Standard Error of Mean 0.191
Statistical Analysis 22: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = 0.11, Standard Deviation 1.24 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 23: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; p = 0.604, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.10, 95% CI 2-sided [-0.493 to 0.287], Standard Error of Mean 0.198
Statistical Analysis 24: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = 0.09, Standard Deviation 1.21 — [estimate comment as in outcome 1, analysis 2]

18. Secondary Outcome: Change From Baseline Over Time in ADAS-Cog-14 Naming Score
Description: The ADAS-Cog was designed to assess the cognitive impairments most common in AD. The ADAS-Cog-14 includes the original 11 items from the ADAS-Cog-11 [1. Spoken language ability, 2. Comprehension of spoken language, 3. Recall of test instructions, 4. Word-findings difficulty in spontaneous speech, 5. Following commands, 6. Naming objects and fingers, 7. Constructional praxis, 8. Ideational praxis, 9. Orientation, 10. Word-recall task, 11. Word-recognition task] and includes 3 additional tasks [12. Number cancellation task, 13. Delayed word recall task, 14. Executive functioning], for increased sensitivity in MCI patients. The Naming Score of the ADAS-Cog-14 ranges from 0 to 5 with a higher score representing greater impairment.
Time Frame: Baseline, Week 24, Week 48, Week 72, Week 96
Population: as for outcome 14
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | ABBV-8E12 300 mg | ABBV-8E12 1000 mg | ABBV-8E12 2000 mg
Number analyzed (Participants) | 114 | 108 | 116 | 113
score on a scale
  Change at Week 24: number analyzed (Participants) | 108 | 106 | 113 | 102
  Change at Week 24 | 0.02 (0.048) | 0.08 (0.049) | -0.03 (0.047) | 0.05 (0.050)
  Change at Week 48: number analyzed (Participants) | 101 | 92 | 105 | 93
  Change at Week 48 | 0.11 (0.049) | 0.09 (0.051) | 0.08 (0.048) | 0.03 (0.050)
  Change at Week 72: number analyzed (Participants) | 97 | 92 | 96 | 95
  Change at Week 72 | 0.21 (0.063) | 0.14 (0.065) | 0.08 (0.063) | 0.07 (0.064)
  Change at Week 96: number analyzed (Participants) | 79 | 80 | 86 | 75
  Change at Week 96 | 0.34 (0.085) | 0.34 (0.086) | 0.28 (0.082) | 0.20 (0.087)
Statistical Analysis 1: Comparison: Placebo vs ABBV-8E12 300 mg; Week 24; Test type: Superiority; p = 0.325, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = 0.07, 95% CI 2-sided [-0.067 to 0.202], Standard Error of Mean 0.069
Statistical Analysis 2: Comparison: Placebo vs ABBV-8E12 300 mg; Week 24; Test type: Superiority; Effect size/pooled SD = -0.12, Standard Deviation 0.57 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 24; Test type: Superiority; p = 0.510, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.04, 95% CI 2-sided [-0.177 to 0.088], Standard Error of Mean 0.067
Statistical Analysis 4: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 24; Test type: Superiority; Effect size/pooled SD = 0.10, Standard Deviation 0.44 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 24; Test type: Superiority; p = 0.601, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = 0.04, 95% CI 2-sided [-0.100 to 0.172], Standard Error of Mean 0.069
Statistical Analysis 6: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 24; Test type: Superiority; Effect size/pooled SD = -0.07, Standard Deviation 0.49 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 7: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; p = 0.783, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.02, 95% CI 2-sided [-0.157 to 0.119], Standard Error of Mean 0.070
Statistical Analysis 8: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.04, Standard Deviation 0.52 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 9: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; p = 0.646, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.03, 95% CI 2-sided [-0.165 to 0.103], Standard Error of Mean 0.068
Statistical Analysis 10: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.06, Standard Deviation 0.48 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 11: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Superiority; p = 0.209, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.09, 95% CI 2-sided [-0.226 to 0.050], Standard Error of Mean 0.070
Statistical Analysis 12: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.18, Standard Deviation 0.49 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 13: Comparison: Placebo vs ABBV-8E12 300 mg; Week 72; Test type: Superiority; p = 0.454, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.07, 95% CI 2-sided [-0.246 to 0.110], Standard Error of Mean 0.091
Statistical Analysis 14: Comparison: Placebo vs ABBV-8E12 300 mg; Week 72; Test type: Superiority; Effect size/pooled SD = 0.10, Standard Deviation 0.66 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 15: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 72; Test type: Superiority; p = 0.141, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.13, 95% CI 2-sided [-0.306 to 0.043], Standard Error of Mean 0.089
Statistical Analysis 16: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 72; Test type: Superiority; Effect size/pooled SD = 0.23, Standard Deviation 0.58 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 17: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 72; Test type: Superiority; p = 0.107, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.15, 95% CI 2-sided [-0.323 to 0.031], Standard Error of Mean 0.090
Statistical Analysis 18: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 72; Test type: Superiority; Effect size/pooled SD = 0.24, Standard Deviation 0.59
Statistical Analysis 19: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; p = 0.961, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.01, 95% CI 2-sided [-0.243 to 0.232], Standard Error of Mean 0.121
Statistical Analysis 20: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; Effect size/pooled SD = 0.01, Standard Deviation 0.79 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 21: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; p = 0.618, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.06, 95% CI 2-sided [-0.290 to 0.173], Standard Error of Mean 0.118
Statistical Analysis 22: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = 0.08, Standard Deviation 0.77 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 23: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; p = 0.227, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.15, 95% CI 2-sided [-0.385 to 0.092], Standard Error of Mean 0.121
Statistical Analysis 24: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = 0.18, Standard Deviation 0.79

19. Secondary Outcome: Change From Baseline Over Time in ADAS-Cog-14 Orientation Score
Description: The ADAS-Cog was designed to assess the cognitive impairments most common in AD. The ADAS-Cog-14 includes the original 11 items from the ADAS-Cog-11 [1. Spoken language ability, 2. Comprehension of spoken language, 3. Recall of test instructions, 4. Word-findings difficulty in spontaneous speech, 5. Following commands, 6. Naming objects and fingers, 7. Constructional praxis, 8. Ideational praxis, 9. Orientation, 10. Word-recall task, 11. Word-recognition task] and includes 3 additional tasks [12. Number cancellation task, 13. Delayed word recall task, 14. Executive functioning], for increased sensitivity in MCI patients. The Orientation Score of the ADAS-Cog-14 ranges from 0 to 8, with a higher score representing greater impairment.
Time Frame: Baseline, Week 24, Week 48, Week 72, Week 96
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | ABBV-8E12 300 mg | ABBV-8E12 1000 mg | ABBV-8E12 2000 mg
Number analyzed (Participants) | 116 | 108 | 116 | 113
score on a scale
  Change at Week 24: number analyzed (Participants) | 110 | 106 | 113 | 102
  Change at Week 24 | 0.08 (0.127) | 0.42 (0.130) | 0.08 (0.125) | 0.49 (0.132)
  Change at Week 48: number analyzed (Participants) | 102 | 92 | 105 | 93
  Change at Week 48 | 0.63 (0.147) | 0.77 (0.154) | 0.45 (0.145) | 0.61 (0.153)
  Change at Week 72: number analyzed (Participants) | 100 | 92 | 96 | 95
  Change at Week 72 | 1.01 (0.166) | 0.84 (0.172) | 1.02 (0.167) | 1.05 (0.171)
  Change at Week 96: number analyzed (Participants) | 80 | 81 | 86 | 76
  Change at Week 96 | 1.26 (0.196) | 1.46 (0.197) | 1.28 (0.191) | 2.00 (0.202)
Statistical Analysis 1: Comparison: Placebo vs ABBV-8E12 300 mg; Week 24; Test type: Superiority; p = 0.056, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = 0.34, 95% CI 2-sided [-0.009 to 0.697], Standard Error of Mean 0.180
Statistical Analysis 2: Comparison: Placebo vs ABBV-8E12 300 mg; Week 24; Test type: Superiority; Effect size/pooled SD = -0.23, Standard Deviation 1.49 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 24; Test type: Superiority; p = 0.997, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = 0.00, 95% CI 2-sided [-0.348 to 0.349], Standard Error of Mean 0.177
Statistical Analysis 4: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 24; Test type: Superiority; Effect size/pooled SD = -0.00, Standard Deviation 1.34 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 24; Test type: Superiority; p = 0.023, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = 0.41, 95% CI 2-sided [0.056 to 0.772], Standard Error of Mean 0.182
Statistical Analysis 6: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 24; Test type: Superiority; Effect size/pooled SD = -0.30, Standard Deviation 1.36 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 7: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; p = 0.502, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = 0.14, 95% CI 2-sided [-0.274 to 0.558], Standard Error of Mean 0.212
Statistical Analysis 8: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; Effect size/pooled SD = -0.09, Standard Deviation 1.58 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 9: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; p = 0.379, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.18, 95% CI 2-sided [-0.587 to 0.224], Standard Error of Mean 0.206
Statistical Analysis 10: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.11, Standard Deviation 1.61 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 11: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Superiority; p = 0.916, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.02, 95% CI 2-sided [-0.439 to 0.394], Standard Error of Mean 0.212
Statistical Analysis 12: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.01, Standard Deviation 1.57 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 13: Comparison: Placebo vs ABBV-8E12 300 mg; Week 72; Test type: Superiority; p = 0.487, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.17, 95% CI 2-sided [-0.633 to 0.302], Standard Error of Mean 0.238
Statistical Analysis 14: Comparison: Placebo vs ABBV-8E12 300 mg; Week 72; Test type: Superiority; Effect size/pooled SD = 0.10, Standard Deviation 1.70 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 15: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 72; Test type: Superiority; p = 0.963, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = 0.01, 95% CI 2-sided [-0.451 to 0.473], Standard Error of Mean 0.235
Statistical Analysis 16: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 72; Test type: Superiority; Effect size/pooled SD = -0.01, Standard Deviation 1.66 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 17: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 72; Test type: Superiority; p = 0.856, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = 0.04, 95% CI 2-sided [-0.424 to 0.510], Standard Error of Mean 0.238
Statistical Analysis 18: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 72; Test type: Superiority; Effect size/pooled SD = -0.03, Standard Deviation 1.71 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 19: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; p = 0.463, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = 0.20, 95% CI 2-sided [-0.341 to 0.748], Standard Error of Mean 0.277
Statistical Analysis 20: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; Effect size/pooled SD = -0.11, Standard Deviation 1.87 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 21: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; p = 0.943, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = 0.02, 95% CI 2-sided [-0.518 to 0.557], Standard Error of Mean 0.273
Statistical Analysis 22: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = -0.01, Standard Deviation 1.93 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 23: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; p = 0.009, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = 0.74, 95% CI 2-sided [0.191 to 1.295], Standard Error of Mean 0.281
Statistical Analysis 24: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = -0.38, Standard Deviation 1.97 — [estimate comment as in outcome 1, analysis 2]

20. Secondary Outcome: Change From Baseline Over Time in ADAS-Cog-14 Word Recall - Number of Words Not Recalled Score
Description: The ADAS-Cog was designed to assess the cognitive impairments most common in AD. The ADAS-Cog-14 includes the original 11 items from the ADAS-Cog-11 [1. Spoken language ability, 2. Comprehension of spoken language, 3. Recall of test instructions, 4. Word-findings difficulty in spontaneous speech, 5. Following commands, 6. Naming objects and fingers, 7. Constructional praxis, 8. Ideational praxis, 9. Orientation, 10. Word-recall task, 11. Word-recognition task] and includes 3 additional tasks [12. Number cancellation task, 13. Delayed word recall task, 14. Executive functioning], for increased sensitivity in MCI patients. The Word Recall - Number of Words Not Recalled Score of the ADAS-Cog-14 ranges from 0 to 10, with a higher score representing greater impairment.
Time Frame: Baseline, Week 24, Week 48, Week 72, Week 96
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | ABBV-8E12 300 mg | ABBV-8E12 1000 mg | ABBV-8E12 2000 mg
Number analyzed (Participants) | 116 | 108 | 116 | 113
score on a scale
  Change at Week 24: number analyzed (Participants) | 110 | 106 | 113 | 102
  Change at Week 24 | 0.16 (0.098) | 0.03 (0.100) | 0.16 (0.097) | 0.11 (0.101)
  Change at Week 48: number analyzed (Participants) | 102 | 92 | 105 | 93
  Change at Week 48 | 0.39 (0.101) | 0.32 (0.105) | 0.41 (0.100) | 0.38 (0.105)
  Change at Week 72: number analyzed (Participants) | 100 | 92 | 96 | 94
  Change at Week 72 | 0.58 (0.113) | 0.64 (0.117) | 0.60 (0.114) | 0.70 (0.116)
  Change at Week 96: number analyzed (Participants) | 81 | 81 | 88 | 76
  Change at Week 96 | 1.04 (0.131) | 0.97 (0.132) | 0.89 (0.127) | 0.91 (0.135)
Statistical Analysis 1: Comparison: Placebo vs ABBV-8E12 300 mg; Week 24; Test type: Superiority; p = 0.325, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.14, 95% CI 2-sided [-0.408 to 0.136], Standard Error of Mean 0.138
Statistical Analysis 2: Comparison: Placebo vs ABBV-8E12 300 mg; Week 24; Test type: Superiority; Effect size/pooled SD = 0.13, Standard Deviation 1.02 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 24; Test type: Superiority; p = 0.966, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.01, 95% CI 2-sided [-0.274 to 0.263], Standard Error of Mean 0.137
Statistical Analysis 4: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 24; Test type: Superiority; Effect size/pooled SD = 0.01, Standard Deviation 1.11 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 24; Test type: Superiority; p = 0.695, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.05, 95% CI 2-sided [-0.330 to 0.220], Standard Error of Mean 0.140
Statistical Analysis 6: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 24; Test type: Superiority; Effect size/pooled SD = 0.05, Standard Deviation 1.09 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 7: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; p = 0.662, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.06, 95% CI 2-sided [-0.348 to 0.221], Standard Error of Mean 0.145
Statistical Analysis 8: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.06, Standard Deviation 1.01 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 9: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; p = 0.849, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = 0.03, 95% CI 2-sided [-0.250 to 0.304], Standard Error of Mean 0.141
Statistical Analysis 10: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = -0.03, Standard Deviation 1.08 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 11: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Superiority; p = 0.995, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.00, 95% CI 2-sided [-0.286 to 0.284], Standard Error of Mean 0.145
Statistical Analysis 12: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.00, Standard Deviation 0.96 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 13: Comparison: Placebo vs ABBV-8E12 300 mg; Week 72; Test type: Superiority; p = 0.707, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = 0.06, 95% CI 2-sided [-0.256 to 0.378], Standard Error of Mean 0.161
Statistical Analysis 14: Comparison: Placebo vs ABBV-8E12 300 mg; Week 72; Test type: Superiority; Effect size/pooled SD = -0.05, Standard Deviation 1.13 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 15: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 72; Test type: Superiority; p = 0.901, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = 0.02, 95% CI 2-sided [-0.294 to 0.333], Standard Error of Mean 0.159
Statistical Analysis 16: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 72; Test type: Superiority; Effect size/pooled SD = -0.02, Standard Deviation 1.23 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 17: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 72; Test type: Superiority; p = 0.451, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = 0.12, 95% CI 2-sided [-0.195 to 0.439], Standard Error of Mean 0.161
Statistical Analysis 18: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 72; Test type: Superiority; Effect size/pooled SD = -0.11, Standard Deviation 1.13 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 19: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; p = 0.722, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.07, 95% CI 2-sided [-0.429 to 0.298], Standard Error of Mean 0.185
Statistical Analysis 20: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; Effect size/pooled SD = 0.06, Standard Deviation 1.13 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 21: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; p = 0.420, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.15, 95% CI 2-sided [-0.503 to 0.210], Standard Error of Mean 0.181
Statistical Analysis 22: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = 0.12, Standard Deviation 1.21 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 23: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; p = 0.498, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.13, 95% CI 2-sided [-0.495 to 0.241], Standard Error of Mean 0.187
Statistical Analysis 24: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = 0.11, Standard Deviation 1.20 — [estimate comment as in outcome 1, analysis 2]

21. Secondary Outcome: Change From Baseline Over Time in ADAS-Cog-14 Remember Word Recognition Instructions Score
Description: The ADAS-Cog was designed to assess the cognitive impairments most common in AD. The ADAS-Cog-14 includes the original 11 items from the ADAS-Cog-11 [1. Spoken language ability, 2. Comprehension of spoken language, 3. Recall of test instructions, 4. Word-findings difficulty in spontaneous speech, 5. Following commands, 6. Naming objects and fingers, 7. Constructional praxis, 8. Ideational praxis, 9. Orientation, 10. Word-recall task, 11. Word-recognition task] and includes 3 additional tasks [12. Number cancellation task, 13. Delayed word recall task, 14. Executive functioning], for increased sensitivity in MCI patients. The Remember Word Recognition Instructions Score of the ADAS-Cog-14 ranges from 0 to 5, with a higher score representing greater impairment.
Time Frame: Baseline, Week 24, Week 48, Week 72, Week 96
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | ABBV-8E12 300 mg | ABBV-8E12 1000 mg | ABBV-8E12 2000 mg
Number analyzed (Participants) | 116 | 108 | 116 | 113
score on a scale
  Change at Week 24: number analyzed (Participants) | 110 | 106 | 113 | 102
  Change at Week 24 | 0.03 (0.050) | 0.03 (0.051) | 0.15 (0.049) | -0.02 (0.052)
  Change at Week 48: number analyzed (Participants) | 102 | 92 | 105 | 93
  Change at Week 48 | 0.27 (0.071) | 0.10 (0.074) | 0.19 (0.070) | 0.06 (0.074)
  Change at Week 72: number analyzed (Participants) | 100 | 92 | 96 | 95
  Change at Week 72 | 0.24 (0.091) | 0.19 (0.094) | 0.29 (0.091) | 0.26 (0.093)
  Change at Week 96: number analyzed (Participants) | 80 | 81 | 82 | 72
  Change at Week 96 | 0.40 (0.112) | 0.45 (0.113) | 0.27 (0.111) | 0.46 (0.117)
Statistical Analysis 1: Comparison: Placebo vs ABBV-8E12 300 mg; Week 24; Test type: Superiority; p = 0.975, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = 0.00, 95% CI 2-sided [-0.138 to 0.142], Standard Error of Mean 0.071
Statistical Analysis 2: Comparison: Placebo vs ABBV-8E12 300 mg; Week 24; Test type: Superiority; Effect size/pooled SD = -0.00, Standard Deviation 0.45 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 24; Test type: Superiority; p = 0.078, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = 0.12, 95% CI 2-sided [-0.014 to 0.261], Standard Error of Mean 0.070
Statistical Analysis 4: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 24; Test type: Superiority; Effect size/pooled SD = -0.19, Standard Deviation 0.66 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 24; Test type: Superiority; p = 0.514, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.05, 95% CI 2-sided [-0.188 to 0.094], Standard Error of Mean 0.072
Statistical Analysis 6: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 24; Test type: Superiority; Effect size/pooled SD = 0.10, Standard Deviation 0.47 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 7: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; p = 0.107, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.17, 95% CI 2-sided [-0.367 to 0.036], Standard Error of Mean 0.102
Statistical Analysis 8: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.23, Standard Deviation 0.73 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 9: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; p = 0.425, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.08, 95% CI 2-sided [-0.275 to 0.116], Standard Error of Mean 0.099
Statistical Analysis 10: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.09, Standard Deviation 0.85 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 11: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Superiority; p = 0.039, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.21, 95% CI 2-sided [-0.413 to -0.011], Standard Error of Mean 0.102
Statistical Analysis 12: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.28, Standard Deviation 0.77 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 13: Comparison: Placebo vs ABBV-8E12 300 mg; Week 72; Test type: Superiority; p = 0.729, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.05, 95% CI 2-sided [-0.302 to 0.212], Standard Error of Mean 0.131
Statistical Analysis 14: Comparison: Placebo vs ABBV-8E12 300 mg; Week 72; Test type: Superiority; Effect size/pooled SD = 0.06, Standard Deviation 0.81 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 15: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 72; Test type: Superiority; p = 0.671, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = 0.05, 95% CI 2-sided [-0.198 to 0.307], Standard Error of Mean 0.128
Statistical Analysis 16: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 72; Test type: Superiority; Effect size/pooled SD = -0.06, Standard Deviation 0.94 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 17: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 72; Test type: Superiority; p = 0.876, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = 0.02, 95% CI 2-sided [-0.235 to 0.276], Standard Error of Mean 0.130
Statistical Analysis 18: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 72; Test type: Superiority; Effect size/pooled SD = -0.02, Standard Deviation 0.92 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 19: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; p = 0.763, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = 0.05, 95% CI 2-sided [-0.266 to 0.362], Standard Error of Mean 0.159
Statistical Analysis 20: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; Effect size/pooled SD = -0.04, Standard Deviation 1.11 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 21: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; p = 0.429, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.12, 95% CI 2-sided [-0.434 to 0.185], Standard Error of Mean 0.157
Statistical Analysis 22: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = 0.12, Standard Deviation 1.01 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 23: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; p = 0.701, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = 0.06, 95% CI 2-sided [-0.256 to 0.381], Standard Error of Mean 0.162
Statistical Analysis 24: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = -0.06, Standard Deviation 1.02 — [estimate comment as in outcome 1, analysis 2]

22. Secondary Outcome: Change From Baseline Over Time in ADAS-Cog-14 Spoken Language Ability Score
Description: The ADAS-Cog was designed to assess the cognitive impairments most common in AD. The ADAS-Cog-14 includes the original 11 items from the ADAS-Cog-11 [1. Spoken language ability, 2. Comprehension of spoken language, 3. Recall of test instructions, 4. Word-findings difficulty in spontaneous speech, 5. Following commands, 6. Naming objects and fingers, 7. Constructional praxis, 8. Ideational praxis, 9. Orientation, 10. Word-recall task, 11. Word-recognition task] and includes 3 additional tasks [12. Number cancellation task, 13. Delayed word recall task, 14. Executive functioning], for increased sensitivity in MCI patients. The Spoken Language Ability Score of the ADAS-Cog-14 ranges from 0 to 5, with a higher score representing greater impairment.
Time Frame: Baseline, Week 24, Week 48, Week 72, Week 96
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | ABBV-8E12 300 mg | ABBV-8E12 1000 mg | ABBV-8E12 2000 mg
Number analyzed (Participants) | 116 | 108 | 116 | 113
score on a scale
  Change at Week 24: number analyzed (Participants) | 110 | 106 | 113 | 102
  Change at Week 24 | 0.07 (0.045) | 0.08 (0.046) | 0.06 (0.045) | 0.11 (0.047)
  Change at Week 48: number analyzed (Participants) | 102 | 92 | 105 | 93
  Change at Week 48 | 0.14 (0.051) | 0.04 (0.054) | 0.03 (0.051) | 0.11 (0.053)
  Change at Week 72: number analyzed (Participants) | 100 | 92 | 96 | 95
  Change at Week 72 | 0.23 (0.066) | 0.11 (0.069) | 0.19 (0.066) | 0.24 (0.068)
  Change at Week 96: number analyzed (Participants) | 81 | 81 | 87 | 76
  Change at Week 96 | 0.29 (0.089) | 0.23 (0.090) | 0.25 (0.087) | 0.43 (0.092)
Statistical Analysis 1: Comparison: Placebo vs ABBV-8E12 300 mg; Week 24; Test type: Superiority; p = 0.867, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = 0.01, 95% CI 2-sided [-0.115 to 0.137], Standard Error of Mean 0.064
Statistical Analysis 2: Comparison: Placebo vs ABBV-8E12 300 mg; Week 24; Test type: Superiority; Effect size/pooled SD = -0.02, Standard Deviation 0.48 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 24; Test type: Superiority; p = 0.898, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.01, 95% CI 2-sided [-0.132 to 0.116], Standard Error of Mean 0.063
Statistical Analysis 4: Comparison: Placebo vs ABBV-8E12 300 mg; Week 24; Test type: Superiority; Effect size/pooled SD = 0.02, Standard Deviation 0.51 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 24; Test type: Superiority; p = 0.537, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = 0.04, 95% CI 2-sided [-0.088 to 0.168], Standard Error of Mean 0.065
Statistical Analysis 6: Comparison: Placebo vs ABBV-8E12 300 mg; Week 24; Test type: Superiority; Effect size/pooled SD = -0.07, Standard Deviation 0.54 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 7: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; p = 0.176, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.10, 95% CI 2-sided [-0.245 to 0.045], Standard Error of Mean 0.074
Statistical Analysis 8: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.15, Standard Deviation 0.65 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 9: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; p = 0.125, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.11, 95% CI 2-sided [-0.251 to 0.031], Standard Error of Mean 0.072
Statistical Analysis 10: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.21, Standard Deviation 0.53 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 11: Comparison: Placebo vs ABBV-8E12 2000 mg; week 48; Test type: Superiority; p = 0.676, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.03, 95% CI 2-sided [-0.176 to 0.114], Standard Error of Mean 0.074
Statistical Analysis 12: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.05, Standard Deviation 0.61 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 13: Comparison: Placebo vs ABBV-8E12 300 mg; Week 72; Test type: Superiority; p = 0.226, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.12, 95% CI 2-sided [-0.301 to 0.071], Standard Error of Mean 0.095
Statistical Analysis 14: Comparison: Placebo vs ABBV-8E12 300 mg; Week 72; Test type: Superiority; Effect size/pooled SD = 0.18, Standard Deviation 0.62 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 15: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 72; Test type: Superiority; p = 0.683, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.04, 95% CI 2-sided [-0.222 to 0.145], Standard Error of Mean 0.093
Statistical Analysis 16: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 72; Test type: Superiority; Effect size/pooled SD = 0.06, Standard Deviation 0.63 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 17: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 72; Test type: Superiority; p = 0.848, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = 0.02, 95% CI 2-sided [-0.168 to 0.204], Standard Error of Mean 0.094
Statistical Analysis 18: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 72; Test type: Superiority; Effect size/pooled SD = -0.03, Standard Deviation 0.67 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 19: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; p = 0.656, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.06, 95% CI 2-sided [-0.305 to 0.192], Standard Error of Mean 0.126
Statistical Analysis 20: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; Effect size/pooled SD = 0.07, Standard Deviation 0.78 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 21: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; p = 0.777, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.04, 95% CI 2-sided [-0.279 to 0.209], Standard Error of Mean 0.124
Statistical Analysis 22: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = 0.04, Standard Deviation 0.88 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 23: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; p = 0.256, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = 0.15, 95% CI 2-sided [-0.106 to 0.397], Standard Error of Mean 0.128
Statistical Analysis 24: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = -0.16, Standard Deviation 0.89 — [estimate comment as in outcome 1, analysis 2]

23. Secondary Outcome: Change From Baseline Over Time in ADAS-Cog-14 Word Find Difficulty Spontaneous Speech Score
Description: The ADAS-Cog was designed to assess the cognitive impairments most common in AD. The ADAS-Cog-14 includes the original 11 items from the ADAS-Cog-11 [1. Spoken language ability, 2. Comprehension of spoken language, 3. Recall of test instructions, 4. Word-findings difficulty in spontaneous speech, 5. Following commands, 6. Naming objects and fingers, 7. Constructional praxis, 8. Ideational praxis, 9. Orientation, 10. Word-recall task, 11. Word-recognition task] and includes 3 additional tasks [12. Number cancellation task, 13. Delayed word recall task, 14. Executive functioning], for increased sensitivity in MCI patients. The Word Find Difficulty Spontaneous Speech Score of the ADAS-Cog-14 ranges from 0 to 5, with a higher score representing greater impairment.
Time Frame: Baseline, Week 24, Week 48, Week 72, Week 96
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | ABBV-8E12 300 mg | ABBV-8E12 1000 mg | ABBV-8E12 2000 mg
Number analyzed (Participants) | 116 | 108 | 116 | 113
score on a scale
  Change at Week 24: number analyzed (Participants) | 110 | 106 | 113 | 102
  Change at Week 24 | 0.21 (0.071) | 0.14 (0.073) | 0.11 (0.070) | 0.23 (0.074)
  Change at Week 48: number analyzed (Participants) | 102 | 92 | 105 | 93
  Change at Week 48 | 0.25 (0.077) | 0.19 (0.081) | 0.21 (0.077) | 0.31 (0.081)
  Change at Week 72: number analyzed (Participants) | 100 | 92 | 96 | 95
  Change at Week 72 | 0.47 (0.093) | 0.28 (0.096) | 0.44 (0.094) | 0.42 (0.096)
  Change at Week 96: number analyzed (Participants) | 81 | 81 | 87 | 76
  Change at Week 96 | 0.58 (0.117) | 0.35 (0.119) | 0.47 (0.114) | 0.60 (0.121)
Statistical Analysis 1: Comparison: Placebo vs ABBV-8E12 300 mg; Week 24; Test type: Superiority; p = 0.479, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.07, 95% CI 2-sided [-0.269 to 0.126], Standard Error of Mean 0.101
Statistical Analysis 2: Comparison: Placebo vs ABBV-8E12 300 mg; Week 24; Test type: Superiority; Effect size/pooled SD = 0.09, Standard Deviation 0.78 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 24; Test type: Superiority; p = 0.295, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.10, 95% CI 2-sided [-0.299 to 0.091], Standard Error of Mean 0.099
Statistical Analysis 4: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 24; Test type: Superiority; Effect size/pooled SD = 0.13, Standard Deviation 0.77 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 24; Test type: Superiority; p = 0.884, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = 0.01, 95% CI 2-sided [-0.186 to 0.215], Standard Error of Mean 0.102
Statistical Analysis 6: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 24; Test type: Superiority; Effect size/pooled SD = -0.02, Standard Deviation 0.83 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 7: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; p = 0.569, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.06, 95% CI 2-sided [-0.281 to 0.155], Standard Error of Mean 0.111
Statistical Analysis 8: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.08, Standard Deviation 0.78 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 9: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; p = 0.702, repeated measures model — [p-value comment as in outcome 10, analysis 1]; Effect size/pooled SD = -0.04, 95% CI 2-sided [-0.254 to 0.171], Standard Error of Mean 0.108
Statistical Analysis 10: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.05, Standard Deviation 0.78 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 11: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Superiority; p = 0.566, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = 0.06, 95% CI 2-sided [-0.155 to 0.283], Standard Error of Mean 0.111
Statistical Analysis 12: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = -0.07, Standard Deviation 0.91 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 13: Comparison: Placebo vs ABBV-8E12 300 mg; Week 72; Test type: Superiority; p = 0.141, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.20, 95% CI 2-sided [-0.458 to 0.065], Standard Error of Mean 0.133
Statistical Analysis 14: Comparison: Placebo vs ABBV-8E12 300 mg; Week 72; Test type: Superiority; Effect size/pooled SD = 0.22, Standard Deviation 0.91 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 15: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 72; Test type: Superiority; p = 0.834, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.03, 95% CI 2-sided [-0.285 to 0.230], Standard Error of Mean 0.131
Statistical Analysis 16: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 72; Test type: Superiority; Effect size/pooled SD = 0.03, Standard Deviation 0.99 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 17: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 72; Test type: Superiority; p = 0.724, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.05, 95% CI 2-sided [-0.309 to 0.215], Standard Error of Mean 0.133
Statistical Analysis 18: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 72; Test type: Superiority; Effect size/pooled SD = 0.05, Standard Deviation 1.00 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 19: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; p = 0.163, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.23, 95% CI 2-sided [-0.559 to 0.095], Standard Error of Mean 0.166
Statistical Analysis 20: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; Effect size/pooled SD = 0.24, Standard Deviation 0.98 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 21: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; p = 0.497, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.11, 95% CI 2-sided [-0.432 to 0.210], Standard Error of Mean 0.163
Statistical Analysis 22: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; effect size = 0.10, Standard Deviation 1.09 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 23: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; p = 0.919, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = 0.02, 95% CI 2-sided [-0.314 to 0.349], Standard Error of Mean 0.168
Statistical Analysis 24: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = -0.01, Standard Deviation 1.17 — [estimate comment as in outcome 1, analysis 2]

24. Secondary Outcome: Change From Baseline Over Time in ADAS-Cog-14 Word Recognition Score
Description: The ADAS-Cog was designed to assess the cognitive impairments most common in AD. The ADAS-Cog-14 includes the original 11 items from the ADAS-Cog-11 [1. Spoken language ability, 2. Comprehension of spoken language, 3. Recall of test instructions, 4. Word-findings difficulty in spontaneous speech, 5. Following commands, 6. Naming objects and fingers, 7. Constructional praxis, 8. Ideational praxis, 9. Orientation, 10. Word-recall task, 11. Word-recognition task] and includes 3 additional tasks [12. Number cancellation task, 13. Delayed word recall task, 14. Executive functioning], for increased sensitivity in MCI patients. The Word Recognition Score of the ADAS-Cog-14 ranges from 0 to 12, with a higher score representing greater impairment.
Time Frame: Baseline, Week 24, Week 48, Week 72, Week 96
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | ABBV-8E12 300 mg | ABBV-8E12 1000 mg | ABBV-8E12 2000 mg
Number analyzed (Participants) | 116 | 108 | 116 | 113
score on a scale
  Change at Week 24: number analyzed (Participants) | 110 | 106 | 113 | 102
  Change at Week 24 | 0.53 (0.248) | 0.25 (0.253) | -0.20 (0.245) | -0.02 (0.257)
  Change at Week 48: number analyzed (Participants) | 102 | 92 | 105 | 93
  Change at Week 48 | 1.35 (0.257) | 0.92 (0.270) | 0.73 (0.254) | 0.80 (0.268)
  Change at Week 72: number analyzed (Participants) | 100 | 92 | 96 | 95
  Change at Week 72 | 0.65 (0.245) | 1.05 (0.255) | 0.78 (0.249) | 0.88 (0.252)
  Change at Week 96: number analyzed (Participants) | 80 | 81 | 82 | 72
  Change at Week 96 | 1.98 (0.287) | 1.97 (0.287) | 1.53 (0.283) | 2.09 (0.301)
Statistical Analysis 1: Comparison: Placebo vs ABBV-8E12 300 mg; Week 24; Test type: Superiority; p = 0.423, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.28, 95% CI 2-sided [-0.974 to 0.409], Standard Error of Mean 0.352
Statistical Analysis 2: Comparison: Placebo vs ABBV-8E12 300 mg; Week 24; Test type: Superiority; Effect size/pooled SD = 0.09, Standard Deviation 3.09 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 24; Test type: Superiority; p = 0.036, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.73, 95% CI 2-sided [-1.408 to -0.047], Standard Error of Mean 0.346
Statistical Analysis 4: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 24; Test type: Superiority; Effect size/pooled SD = 0.25, Standard Deviation 2.96 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 24; Test type: Superiority; p = 0.121, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.55, 95% CI 2-sided [-1.250 to 0.147], Standard Error of Mean 0.355
Statistical Analysis 6: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 24; Test type: Superiority; Effect size/pooled SD = 0.18, Standard Deviation 3.09 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 7: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; p = 0.244, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.43, 95% CI 2-sided [-1.163 to 0.296], Standard Error of Mean 0.371
Statistical Analysis 8: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.15, Standard Deviation 2.88 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 9: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; p = 0.085, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.62, 95% CI 2-sided [-1.330 to 0.086], Standard Error of Mean 0.360
Statistical Analysis 10: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.21, Standard Deviation 3.03 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 11: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Superiority; p = 0.137, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.55, 95% CI 2-sided [-1.280 to 0.177], Standard Error of Mean 0.371
Statistical Analysis 12: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.19, Standard Deviation 2.85 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 13: Comparison: Placebo vs ABBV-8E12 300 mg; Week 72; Test type: Superiority; p = 0.258, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = 0.40, 95% CI 2-sided [-0.294 to 1.091], Standard Error of Mean 0.352
Statistical Analysis 14: Comparison: Placebo vs ABBV-8E12 300 mg; Week 72; Test type: Superiority; Effect size/pooled SD = -0.14, Standard Deviation 2.88 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 15: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 72; Test type: Superiority; p = 0.711, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = 0.13, 95% CI 2-sided [-0.555 to 0.814], Standard Error of Mean 0.348
Statistical Analysis 16: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 72; Test type: Superiority; Effect size/pooled SD = -0.04, Standard Deviation 3.05 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 17: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 72; Test type: Superiority; p = 0.503, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = 0.24, 95% CI 2-sided [-0.454 to 0.924], Standard Error of Mean 0.350
Statistical Analysis 18: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 72; Test type: Superiority; Effect size/pooled SD = -0.08, Standard Deviation 2.99 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 19: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; p = 0.978, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.01, 95% CI 2-sided [-0.806 to 0.784], Standard Error of Mean 0.404
Statistical Analysis 20: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; Effect size/pooled SD = 0.00, Standard Deviation 3.12 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 21: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; p = 0.265, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = -0.45, 95% CI 2-sided [-1.239 to 0.342], Standard Error of Mean 0.402
Statistical Analysis 22: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = 0.14, Standard Deviation 3.15 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 23: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; p = 0.789, repeated measures model — [p-value comment as in outcome 10, analysis 1]; LS Mean of Difference = 0.11, 95% CI 2-sided [-0.704 to 0.925], Standard Error of Mean 0.414
Statistical Analysis 24: Comparison: Placebo vs ABBV-8E12 2000 mg; Effect size at a specific visit is calculated as LS mean difference (placebo - 8E12) divided by pooled standard deviation of change scores for a ABBV-8E12 dose and placebo at that visit; Test type: Superiority; Effect size/pooled SD = -0.04, Standard Deviation 2.82

25. Secondary Outcome: Change From Baseline Over Time in Functional Activities Questionnaire (FAQ) Score
Description: The FAQ measures level of assistance (functional disability) needed for carrying out instrumental activities in daily living (iADLs). The FAQ score ranges from 0 - 30 and consists of 10 items (each scored from 0 - 3), which measure a specific iADL in the past 4-weeks: [1) writing checks, paying bills, keeping financial records; 2) assembling tax or business records; 3) shopping alone; 4) playing a game of skill; 5) making coffee or tea; 6) preparing a balanced meal; 7) keeping track of current events; 8) attending to and understanding a television program, book, or magazine; 9) remembering appointments, family occasions, medications; and 10) traveling out of the neighborhood]. Performance in each category is rated from 0 - 3 as follows: 0 - normal; 1 - has difficulty, but does by self; 2 - requires assistance; or 3 - dependent. The FAQ was administered by a trained interviewer. Higher scores indicate a greater requirement of assistance.
Time Frame: Baseline, Week 24, Week 48, Week 72, Week 96
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | ABBV-8E12 300 mg | ABBV-8E12 1000 mg | ABBV-8E12 2000 mg
Number analyzed (Participants) | 116 | 108 | 116 | 113
score on a scale
  Change at Week 24: number analyzed (Participants) | 112 | 105 | 111 | 103
  Change at Week 24 | 1.63 (0.422) | 1.84 (0.435) | 1.19 (0.423) | 2.06 (0.439)
  Change at Week 48: number analyzed (Participants) | 105 | 96 | 106 | 98
  Change at Week 48 | 3.37 (0.480) | 3.53 (0.498) | 2.83 (0.477) | 3.58 (0.496)
  Change at Week 72: number analyzed (Participants) | 100 | 95 | 101 | 96
  Change at Week 72 | 5.62 (0.571) | 5.09 (0.588) | 4.57 (0.568) | 6.31 (0.586)
  Change at Week 96: number analyzed (Participants) | 86 | 85 | 92 | 82
  Change at Week 96 | 6.14 (0.650) | 7.11 (0.663) | 5.80 (0.638) | 7.94 (0.667)
Statistical Analysis 1: Comparison: Placebo vs ABBV-8E12 300 mg; Week 24; Test type: Superiority; p = 0.720, repeated measures model — The statistical model: FAQ change from baseline = baseline + treatment + site + visit + baseline*visit + treatment*visit; variance-covariance structure = Unstructured; LS Mean of Difference = 0.21, 95% CI 2-sided [-0.965 to 1.395], Standard Error of Mean 0.600
Statistical Analysis 2: Comparison: Placebo vs ABBV-8E12 300 mg; Week 24; Test type: Superiority; Effect size/pooled SD = -0.05, Standard Deviation 4.73 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 24; Test type: Superiority; p = 0.455, repeated measures model — [p-value comment as in outcome 25, analysis 1]; LS Mean of Difference = -0.44, 95% CI 2-sided [-1.607 to 0.722], Standard Error of Mean 0.592
Statistical Analysis 4: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 24; Test type: Superiority; Effect size/pooled SD = 0.10, Standard Deviation 4.55 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 24; Test type: Superiority; p = 0.473, repeated measures model — [p-value comment as in outcome 25, analysis 1]; LS Mean of Difference = 0.43, 95% CI 2-sided [-0.755 to 1.625], Standard Error of Mean 0.605
Statistical Analysis 6: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 24; Test type: Superiority; Effect size/pooled SD = -0.10, Standard Deviation 4.25 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 7: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; p = 0.813, repeated measures model — [p-value comment as in outcome 25, analysis 1]; LS Mean of Difference = 0.16, 95% CI 2-sided [-1.187 to 1.512], Standard Error of Mean 0.686
Statistical Analysis 8: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; Effect size/pooled SD = -0.03, Standard Deviation 5.30
Statistical Analysis 9: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; p = 0.421, repeated measures model — [p-value comment as in outcome 25, analysis 1]; LS Mean of Difference = -0.54, 95% CI 2-sided [-1.863 to 0.780], Standard Error of Mean 0.672
Statistical Analysis 10: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.10, Standard Deviation 5.51 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 11: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Superiority; p = 0.758, repeated measures model — [p-value comment as in outcome 25, analysis 1]; LS Mean of Difference = 0.21, 95% CI 2-sided [-1.139 to 1.564], Standard Error of Mean 0.687
Statistical Analysis 12: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = -0.04, Standard Deviation 5.18 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 13: Comparison: Placebo vs ABBV-8E12 300 mg; Week 72; Test type: Superiority; p = 0.511, repeated measures model — [p-value comment as in outcome 25, analysis 1]; LS Mean of Difference = -0.54, 95% CI 2-sided [-2.140 to 1.066], Standard Error of Mean 0.815
Statistical Analysis 14: Comparison: Placebo vs ABBV-8E12 300 mg; Week 72; Test type: Superiority; Effect size/pooled SD = 0.09, Standard Deviation 6.19 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 15: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 72; Test type: Superiority; p = 0.192, repeated measures model — [p-value comment as in outcome 25, analysis 1]; LS Mean of Difference = -1.05, 95% CI 2-sided [-2.623 to 0.527], Standard Error of Mean 0.801
Statistical Analysis 16: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 72; Test type: Superiority; Effect size/pooled SD = 0.17, Standard Deviation 6.16 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 17: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 72; Test type: Superiority; p = 0.398, repeated measures model — [p-value comment as in outcome 25, analysis 1]; LS Mean of Difference = 0.69, 95% CI 2-sided [-0.914 to 2.294], Standard Error of Mean 0.816
Statistical Analysis 18: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 72; Test type: Superiority; Effect size/pooled SD = -0.12, Standard Deviation 5.92 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 19: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; p = 0.296, repeated measures model — [p-value comment as in outcome 25, analysis 1]; LS Mean of Difference = 0.97, 95% CI 2-sided [-0.851 to 2.784], Standard Error of Mean 0.924
Statistical Analysis 20: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; Effect size/pooled SD = -0.14, Standard Deviation 6.74 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 21: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; p = 0.706, repeated measures model — [p-value comment as in outcome 25, analysis 1]; LS Mean of Difference = -0.34, 95% CI 2-sided [-2.126 to 1.442], Standard Error of Mean 0.907
Statistical Analysis 22: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = 0.05, Standard Deviation 6.49 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 23: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; p = 0.055, repeated measures model — [p-value comment as in outcome 25, analysis 1]; LS Mean of Difference = 1.79, 95% CI 2-sided [-0.036 to 3.617], Standard Error of Mean 0.929
Statistical Analysis 24: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = -0.28, Standard Deviation 6.45 — [estimate comment as in outcome 1, analysis 2]

26. Secondary Outcome: Change From Baseline Over Time in Alzheimer's Disease Cooperative Study Clinical Global Impression of Change for Mild Cognitive Impairment (ADCS-CGIC-MCI) General Condition Score
Description: The instrument assesses the physician's global impression of change in 4 major cognitive domains. The instrument covers 4 major domains: 1. General condition , 2. Cognition, 3. Behavior, and 4. Social and daily functioning. Scoring is based on a 7-point Likert Scale: 1, marked improvement; 2, moderate improvement; 3, minimal improvement; 4, no change; 5, minimal worsening; 6, moderate worsening; 7, marked worsening. Higher score indicates greater worsening.
Time Frame: Baseline, Week 48, Week 96
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | ABBV-8E12 300 mg | ABBV-8E12 1000 mg | ABBV-8E12 2000 mg
Number analyzed (Participants) | 116 | 108 | 116 | 113
score on a scale
  Change at Week 48: number analyzed (Participants) | 99 | 95 | 104 | 95
  Change at Week 48 | 4.91 (0.078) | 4.86 (0.080) | 4.80 (0.076) | 4.87 (0.079)
  Change at Week 96: number analyzed (Participants) | 83 | 83 | 89 | 80
  Change at Week 96 | 5.29 (0.087) | 5.28 (0.087) | 5.22 (0.083) | 5.34 (0.088)
Statistical Analysis 1: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; p = 0.651, repeated measures model — The statistical model: ADCS-CGIC-MCI change from baseline = treatment + site + visit + treatment*visit; variance-covariance structure = Unstructured; LS Mean of Difference = -0.05, 95% CI 2-sided [-0.266 to 0.166], Standard Error of Mean 0.110
Statistical Analysis 2: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.06, Standard Deviation 0.82 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; p = 0.320, repeated measures model — [p-value comment as in outcome 26, analysis 1]; LS Mean of Difference = -0.11, 95% CI 2-sided [-0.318 to 0.104], Standard Error of Mean 0.107
Statistical Analysis 4: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.13, Standard Deviation 0.81 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Superiority; p = 0.757, repeated measures model — [p-value comment as in outcome 26, analysis 1]; LS Mean of Difference = -0.03, 95% CI 2-sided [-0.250 to 0.182], Standard Error of Mean 0.110
Statistical Analysis 6: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.04, Standard Deviation 0.83 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 7: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; p = 0.984, repeated measures model — [p-value comment as in outcome 26, analysis 1]; LS Mean of Difference = -0.00, 95% CI 2-sided [-0.241 to 0.236], Standard Error of Mean 0.121
Statistical Analysis 8: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; Effect size/pooled SD = 0.00, Standard Deviation 0.85 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 9: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; p = 0.595, repeated measures model — [p-value comment as in outcome 26, analysis 1]; LS Mean of Difference = -0.06, 95% CI 2-sided [-0.296 to 0.170], Standard Error of Mean 0.118
Statistical Analysis 10: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = 0.07, Standard Deviation 0.93 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 11: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; p = 0.670, repeated measures model — [p-value comment as in outcome 26, analysis 1]; LS Mean of Difference = 0.05, 95% CI 2-sided [-0.187 to 0.291], Standard Error of Mean 0.122
Statistical Analysis 12: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = -0.06, Standard Deviation 0.91 — [estimate comment as in outcome 1, analysis 2]

27. Secondary Outcome: Change From Baseline Over Time in ADCS-CGIC-MCI Cognition Score
Description: as for outcome 26
Time Frame: Baseline, Week 48, Week 96
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | ABBV-8E12 300 mg | ABBV-8E12 1000 mg | ABBV-8E12 2000 mg
Number analyzed (Participants) | 116 | 108 | 116 | 113
score on a scale
  Change at Week 48: number analyzed (Participants) | 99 | 95 | 104 | 95
  Change at Week 48 | 4.85 (0.080) | 4.81 (0.081) | 4.83 (0.077) | 4.92 (0.081)
  Change at Week 96: number analyzed (Participants) | 83 | 83 | 89 | 80
  Change at Week 96 | 5.30 (0.092) | 5.29 (0.092) | 5.22 (0.088) | 5.34 (0.093)
Statistical Analysis 1: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; p = 0.722, repeated measures model — [p-value comment as in outcome 26, analysis 1]; LS Mean of Difference = -0.04, 95% CI 2-sided [-0.260 to 0.180], Standard Error of Mean 0.112
Statistical Analysis 2: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.05, Standard Deviation 0.86 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; p = 0.878, repeated measures model — [p-value comment as in outcome 26, analysis 1]; LS Mean of Difference = -0.02, 95% CI 2-sided [-0.232 to 0.198], Standard Error of Mean 0.109
Statistical Analysis 4: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.02, Standard Error of Mean 0.80 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Superiority; p = 0.535, repeated measures model — [p-value comment as in outcome 26, analysis 1]; LS Mean of Difference = 0.07, 95% CI 2-sided [-0.151 to 0.290], Standard Error of Mean 0.112
Statistical Analysis 6: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = -0.09, Standard Deviation 0.81 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 7: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; p = 0.916, repeated measures model — [p-value comment as in outcome 26, analysis 1]; Effect size/pooled SD = -0.01, 95% CI 2-sided [-0.266 to 0.239], Standard Error of Mean 0.129
Statistical Analysis 8: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; Effect size/pooled SD = 0.01, Standard Deviation 0.91 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 9: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; p = 0.511, repeated measures model — [p-value comment as in outcome 26, analysis 1]; LS Mean of Difference = -0.08, 95% CI 2-sided [-0.330 to 0.165], Standard Error of Mean 0.126
Statistical Analysis 10: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = 0.08, Standard Deviation 1.00 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 11: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; p = 0.771, repeated measures model — [p-value comment as in outcome 26, analysis 1]; LS Mean of Difference = 0.04, 95% CI 2-sided [-0.217 to 0.292], Standard Error of Mean 0.129
Statistical Analysis 12: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = -0.04, Standard Deviation 0.94

28. Secondary Outcome: Change From Baseline Over Time in ADCS-CGIC-MCI Behavior Score
Description: as for outcome 26
Time Frame: Baseline, Week 48, Week 96
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | ABBV-8E12 300 mg | ABBV-8E12 1000 mg | ABBV-8E12 2000 mg
Number analyzed (Participants) | 116 | 108 | 116 | 113
score on a scale
  Change at Week 48: number analyzed (Participants) | 99 | 95 | 104 | 95
  Change at Week 48 | 4.30 (0.061) | 4.31 (0.062) | 4.28 (0.059) | 4.33 (0.062)
  Change at Week 96: number analyzed (Participants) | 83 | 83 | 89 | 80
  Change at Week 96 | 4.61 (0.079) | 4.49 (0.078) | 4.57 (0.076) | 4.55 (0.080)
Statistical Analysis 1: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; p = 0.903, repeated measures model — [p-value comment as in outcome 26, analysis 1]; LS Mean of Difference = 0.01, 95% CI 2-sided [-0.159 to 0.180], Standard Error of Mean 0.086
Statistical Analysis 2: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; Effect size/pooled SD = -0.02, Standard Deviation 0.63 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; p = 0.811, repeated measures model — [p-value comment as in outcome 26, analysis 1]; LS Mean of Difference = -0.02, 95% CI 2-sided [-0.185 to 0.145], Standard Error of Mean 0.084
Statistical Analysis 4: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.03, Standard Deviation 0.61 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Superiority; p = 0.775, repeated measures model — [p-value comment as in outcome 26, analysis 1]; LS Mean of Difference = 0.02, 95% CI 2-sided [-0.145 to 0.194], Standard Error of Mean 0.086
Statistical Analysis 6: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = -0.04, Standard Deviation 0.62 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 7: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; p = 0.273, repeated measures model — [p-value comment as in outcome 26, analysis 1]; LS Mean of Difference = -0.12, 95% CI 2-sided [-0.337 to 0.096], Standard Error of Mean 0.110
Statistical Analysis 8: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; Effect size/pooled SD = 0.17, Standard Deviation 0.73 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 9: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; p = 0.740, repeated measures model — [p-value comment as in outcome 26, analysis 1]; LS Mean of Difference = -0.04, 95% CI 2-sided [-0.248 to 0.176], Standard Error of Mean 0.108
Statistical Analysis 10: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = 0.05, Standard Deviation 0.80 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 11: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; p = 0.567, repeated measures model — [p-value comment as in outcome 26, analysis 1]; LS Mean of Difference = -0.06, 95% CI 2-sided [-0.282 to 0.155], Standard Error of Mean 0.111
Statistical Analysis 12: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = 0.08, Standard Deviation 0.80 — [estimate comment as in outcome 1, analysis 2]

29. Secondary Outcome: Change From Baseline Over Time in ADCS-CGIC-MCI Functional Abilities Score
Description: The instrument assesses the physician's global impression of change in 4 major cognitive domains. The instrument covers 4 major domains: 1. General condition , 2. Cognition, 3. Behavior, and 4. Social and daily functioning (functional abilities). Scoring is based on a 7-point Likert Scale: 1, marked improvement; 2, moderate improvement; 3, minimal improvement; 4, no change; 5, minimal worsening; 6, moderate worsening; 7, marked worsening. Higher score indicates greater worsening.
Time Frame: Baseline, Week 48, Week 96
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | ABBV-8E12 300 mg | ABBV-8E12 1000 mg | ABBV-8E12 2000 mg
Number analyzed (Participants) | 116 | 108 | 116 | 113
score on a scale
  Change at Week 48: number analyzed (Participants) | 99 | 95 | 104 | 95
  Change at Week 48 | 4.59 (0.071) | 4.58 (0.072) | 4.46 (0.068) | 4.59 (0.072)
  Change at Week 96: number analyzed (Participants) | 83 | 83 | 89 | 80
  Change at Week 96 | 4.97 (0.088) | 4.95 (0.088) | 4.98 (0.085) | 5.03 (0.090)
Statistical Analysis 1: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; p = 0.931, repeated measures model — [p-value comment as in outcome 26, analysis 1]; LS Mean of Difference = -0.01, 95% CI 2-sided [-0.204 to 0.187], Standard Error of Mean 0.099
Statistical Analysis 2: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.01, Standard Deviation 0.73 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; p = 0.187, repeated measures model — [p-value comment as in outcome 26, analysis 1]; LS Mean of Difference = -0.13, 95% CI 2-sided [-0.320 to 0.063], Standard Error of Mean 0.097
Statistical Analysis 4: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.16, Standard Deviation 0.78 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Superiority; p = 0.961, repeated measures model — [p-value comment as in outcome 26, analysis 1]; LS Mean of Difference = 0.00, 95% CI 2-sided [-0.191 to 0.201], Standard Error of Mean 0.100
Statistical Analysis 6: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = -0.01, Standard Deviation 0.73 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 7: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; p = 0.894, repeated measures model — [p-value comment as in outcome 26, analysis 1]; LS Mean of Difference = -0.02, 95% CI 2-sided [-0.260 to 0.227], Standard Error of Mean 0.124
Statistical Analysis 8: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; Effect size/pooled SD = 0.02, Standard Deviation 0.87 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 9: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; p = 0.917, repeated measures model — [p-value comment as in outcome 26, analysis 1]; LS Mean of Difference = 0.01, 95% CI 2-sided [-0.226 to 0.251], Standard Error of Mean 0.121
Statistical Analysis 10: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = -0.01, Standard Deviation 0.91 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 11: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; p = 0.639, repeated measures model — [p-value comment as in outcome 26, analysis 1]; LS Mean of Difference = 0.06, 95% CI 2-sided [-0.186 to 0.303], Standard Error of Mean 0.124
Statistical Analysis 12: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = -0.06, Standard Deviation 0.91 — [estimate comment as in outcome 1, analysis 2]

30. Secondary Outcome: Change From Baseline Over Time in University of California's Performance Based Skills Assessment, Brief Version (UPSA-Brief) - Total Score
Description: The UPSA-Brief is a performance-based instrument which uses a series of tasks and roleplay scenarios to evaluate a person's functional capacity in two areas of basic living skills (i.e., financial skills and communication skills). Scores range from 0 to 100; a higher score of the UPSA-Brief is desirable.
Time Frame: Baseline, Week 48, Week 96
Population: as for outcome 14
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | ABBV-8E12 300 mg | ABBV-8E12 1000 mg | ABBV-8E12 2000 mg
Number analyzed (Participants) | 116 | 108 | 114 | 112
score on a scale
  Change to Week 48: number analyzed (Participants) | 98 | 93 | 102 | 88
  Change to Week 48 | -4.47 (1.533) | -6.04 (1.567) | -4.10 (1.500) | -8.96 (1.601)
  Change to Week 96: number analyzed (Participants) | 77 | 79 | 81 | 73
  Change to Week 96 | -13.36 (2.047) | -12.74 (2.037) | -11.55 (1.994) | -14.85 (2.104)
Statistical Analysis 1: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; p = 0.470, repeated measures model — The statistical model: UPSA-Brief change from baseline = baseline + treatment + site + visit + baseline*visit + treatment*visit; variance-covariance structure = Unstructured; LS Mean of Difference = -1.57, 95% CI 2-sided [-5.851 to 2.703], Standard Error of Mean 2.175
Statistical Analysis 2: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; Effect size/pooled SD = -0.10, Standard Deviation 15.44 — Effect size at a specific visit is calculated as LS mean difference (8E12 - placebo) divided by pooled standard deviation of change scores for a ABBV-8E12 dose and placebo at that visit
Statistical Analysis 3: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; p = 0.864, repeated measures model — [p-value comment as in outcome 30, analysis 1]; LS Mean of Difference = 0.36, 95% CI 2-sided [-3.819 to 4.548], Standard Error of Mean 2.127
Statistical Analysis 4: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.02, Standard Deviation 15.95 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 5: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Superiority; p = 0.043, repeated measures model — [p-value comment as in outcome 30, analysis 1]; LS Mean of Difference = -4.49, 95% CI 2-sided [-8.826 to -0.150], Standard Error of Mean 2.206
Statistical Analysis 6: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = -0.28, Standard Deviation 16.24 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 7: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; p = 0.831, repeated measures model — [p-value comment as in outcome 30, analysis 1]; LS Mean of Difference = 0.61, 95% CI 2-sided [-5.041 to 6.270], Standard Error of Mean 2.874
Statistical Analysis 8: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; Effect size/pooled SD = 0.03, Standard Deviation 18.06 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 9: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; p = 0.525, repeated measures model — [p-value comment as in outcome 30, analysis 1]; LS Mean of Difference = 1.81, 95% CI 2-sided [-3.784 to 7.404], Standard Error of Mean 2.843
Statistical Analysis 10: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Other; Effect size/pooled SD = 0.10, Standard Error of Mean 18.47 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 11: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; p = 0.610, repeated measures model — [p-value comment as in outcome 30, analysis 1]; LS Mean of Difference = -1.49, 95% CI 2-sided [-7.239 to 4.255], Standard Error of Mean 2.921
Statistical Analysis 12: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = -0.08, Standard Deviation 19.53 — [estimate comment as in outcome 30, analysis 2]

31. Secondary Outcome: Change From Baseline Over Time in 24-Item Alzheimer's Disease Cooperative Study/Activities of Daily Living Scale Adapted for Patients With Mild Cognitive Impairment (ADCS-MCI-ADL-24) Total Score
Description: The ADCS-MCI-ADL-24 is a 24-item, study partner-based assessment of activities of daily living designed specifically for AD patients and is completed by a trained rater. The scale assesses functional activities such as cooking, household chores, shopping, keeping appointments, social interactions and hobbies. Items are assessed according to whether they were performed in the past 4 weeks and, if so, some items are further assessed as to whether they were performed independently, with supervision, or with physical help. Scores on the ADCS-ADL-MCI range from 0 to 69, where higher score indicates greater capability to carry out activities of daily living.
Time Frame: Baseline, Week 48, Week 96
Population: as for outcome 14
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | ABBV-8E12 300 mg | ABBV-8E12 1000 mg | ABBV-8E12 2000 mg
Number analyzed (Participants) | 114 | 108 | 114 | 113
score on a scale
  Change to Week 48: number analyzed (Participants) | 103 | 98 | 105 | 98
  Change to Week 48 | -3.72 (0.723) | -4.51 (0.738) | -2.91 (0.712) | -3.65 (0.740)
  Change to Week 96: number analyzed (Participants) | 83 | 85 | 87 | 79
  Change to Week 96 | -9.21 (1.134) | -10.25 (1.135) | -9.16 (1.112) | -10.60 (1.163)
Statistical Analysis 1: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; p = 0.438, repeated measures model — The statistical model: ADCS-MCI-ADL-24 change from baseline = baseline + treatment + site + visit + baseline*visit + treatment*visit; var-covar structure = Unstructured; LS Mean of Difference = -0.79, 95% CI 2-sided [-2.798 to 1.214], Standard Error of Mean 1.020
Statistical Analysis 2: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; Effect size/pooled SD = -0.10, Standard Deviation 7.87 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; p = 0.419, repeated measures model — [p-value comment as in outcome 31, analysis 1]; LS Mean of Difference = 0.81, 95% CI 2-sided [-1.164 to 2.788], Standard Error of Mean 1.005
Statistical Analysis 4: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.10, Standard Deviation 7.91 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 5: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Superiority; p = 0.948, repeated measures model — [p-value comment as in outcome 31, analysis 1]; LS Mean of Difference = 0.07, 95% CI 2-sided [-1.959 to 2.092], Standard Error of Mean 1.030
Statistical Analysis 6: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.01, Standard Deviation 8.01 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 7: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; p = 0.516, repeated measures model — [p-value comment as in outcome 31, analysis 1]; LS Mean of Difference = -1.04, 95% CI 2-sided [-4.180 to 2.101], Standard Error of Mean 1.597
Statistical Analysis 8: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; Effect size/pooled SD = -0.10, Standard Deviation 10.87 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 9: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; p = 0.971, repeated measures model — [p-value comment as in outcome 31, analysis 1]; LS Mean of Difference = 0.06, 95% CI 2-sided [-3.055 to 3.168], Standard Error of Mean 1.582
Statistical Analysis 10: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = 0.01, Standard Deviation 11.24
Statistical Analysis 11: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; p = 0.392, repeated measures model — [p-value comment as in outcome 31, analysis 1]; LS Mean of Difference = -1.39, 95% CI 2-sided [-4.577 to 1.800], Standard Error of Mean 1.621
Statistical Analysis 12: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = -0.13, Standard Deviation 10.87 — [estimate comment as in outcome 30, analysis 2]

32. Secondary Outcome: Change From Baseline Over Time in Repeatable Battery for Assessment of Neuropsychological Status (RBANS) - Total Scale Score
Description: The RBANS is a 25-minute, standardized neurocognitive battery with North American population-based normative data. The RBANS measures five neurocognitive domains, with age-based scaling. Twelve subtests measure cognitive decline or improvement across the following domains: 1. Immediate Memory - List Learning and Story Memory, 2. Visuospatial/Constructional - Figure Copy and Line Orientation, 3. Language - Picture naming and Semantic Fluency, 4. Attention - Digit Span and Coding, and 5. Delayed Memory - List Recall, List Recognition, Story Memory, and Figure Recall. Total score can range from 40 to 160 with a higher score representing a better outcome.
Time Frame: Baseline, Week 24, Week 48, Week 72, Week 96
Population: as for outcome 14
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | ABBV-8E12 300 mg | ABBV-8E12 1000 mg | ABBV-8E12 2000 mg
Number analyzed (Participants) | 115 | 108 | 116 | 113
score on a scale
  Change to Week 24: number analyzed (Participants) | 108 | 105 | 107 | 100
  Change to Week 24 | -3.52 (0.640) | -4.83 (0.649) | -5.04 (0.637) | -5.17 (0.664)
  Change to Week 48: number analyzed (Participants) | 98 | 90 | 101 | 88
  Change to Week 48 | -1.85 (0.757) | -1.37 (0.782) | -1.86 (0.746) | -2.67 (0.792)
  Change to Week 72: number analyzed (Participants) | 94 | 87 | 90 | 86
  Change to Week 72 | -5.27 (0.861) | -5.95 (0.885) | -6.86 (0.862) | -6.38 (0.897)
  Change to Week 96: number analyzed (Participants) | 74 | 75 | 79 | 64
  Change to Week 96 | -6.79 (0.923) | -7.78 (0.928) | -6.59 (0.901) | -7.03 (0.977)
Statistical Analysis 1: Comparison: Placebo vs ABBV-8E12 300 mg; Week 24; Test type: Superiority; p = 0.148, repeated measures model — The statistical model: RBANS change from baseline = baseline + treatment + site + visit + baseline*visit + treatment*visit; variance-covariance structure = Unstructured; LS Mean of Difference = -1.31, 95% CI 2-sided [-3.080 to 0.465], Standard Error of Mean 0.902
Statistical Analysis 2: Comparison: Placebo vs ABBV-8E12 300 mg; Week 24; Test type: Superiority; Effect size/pooled SD = -0.19, Standard Deviation 6.81 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 24; Test type: Superiority; p = 0.092, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -1.52, 95% CI 2-sided [-3.278 to 0.246], Standard Error of Mean 0.896
Statistical Analysis 4: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 24; Test type: Superiority; Effect size/pooled SD = -0.21, Standard Deviation 7.14 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 5: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 24; Test type: Superiority; p = 0.073, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -1.65, 95% CI 2-sided [-3.446 to 0.152], Standard Error of Mean 0.915
Statistical Analysis 6: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 24; Test type: Superiority; Effect size/pooled SD = -0.25, Standard Deviation 6.55 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 7: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; p = 0.662, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = 0.47, 95% CI 2-sided [-1.652 to 2.599], Standard Error of Mean 1.081
Statistical Analysis 8: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.06, Standard Deviation 8.07 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 9: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; p = 0.992, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.01, 95% CI 2-sided [-2.089 to 2.068], Standard Error of Mean 1.057
Statistical Analysis 10: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = -0.00, Standard Deviation 8.38 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 11: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Superiority; p = 0.451, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.82, 95% CI 2-sided [-2.961 to 1.320], Standard Error of Mean 1.088
Statistical Analysis 12: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = -0.11, Standard Deviation 7.72 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 13: Comparison: Placebo vs ABBV-8E12 300 mg; Week 72; Test type: Superiority; p = 0.583, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.67, 95% CI 2-sided [-3.088 to 1.739], Standard Error of Mean 1.227
Statistical Analysis 14: Comparison: Placebo vs ABBV-8E12 300 mg; Week 72; Test type: Superiority; Effect size/pooled SD = -0.08, Standard Deviation 8.67 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 15: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 72; Test type: Superiority; p = 0.191, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -1.59, 95% CI 2-sided [-3.975 to 0.795], Standard Error of Mean 1.213
Statistical Analysis 16: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 72; Test type: Superiority; Effect size/pooled SD = -0.17, Standard Deviation 9.37 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 17: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 72; Test type: Superiority; p = 0.372, repeated measures model; LS Mean of Difference = -1.11, 95% CI 2-sided [-3.541 to 1.329], Standard Error of Mean 1.238
Statistical Analysis 18: Comparison: ABBV-8E12 2000 mg; Week 72; Test type: Superiority; Effect size/pooled SD = -0.12, Standard Deviation 8.96
Statistical Analysis 19: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; p = 0.447, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.99, 95% CI 2-sided [-3.553 to 1.571], Standard Error of Mean 1.303
Statistical Analysis 20: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; Effect size/pooled SD = -0.11, Standard Deviation 9.35
Statistical Analysis 21: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; p = 0.881, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = 0.19, 95% CI 2-sided [-2.334 to 2.719], Standard Error of Mean 1.285
Statistical Analysis 22: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = 0.02, Standard Deviation 8.68 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 23: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; p = 0.853, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.25, 95% CI 2-sided [-2.881 to 2.383], Standard Error of Mean 1.338
Statistical Analysis 24: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = -0.03, Standard Deviation 8.54 — [estimate comment as in outcome 30, analysis 2]

33. Secondary Outcome: Change From Baseline Over Time in RBANS - Coding Total Score
Description: The RBANS is a 25-minute, standardized neurocognitive battery with North American population-based normative data. The RBANS measures five neurocognitive domains, with age-based scaling. Twelve subtests measure cognitive decline or improvement across the following domains: 1. Immediate Memory - List Learning and Story Memory, 2. Visuospatial/Constructional - Figure Copy and Line Orientation, 3. Language - Picture naming and Semantic Fluency, 4. Attention - Digit Span and Coding, and 5. Delayed Memory - List Recall, List Recognition, Story Memory, and Figure Recall. The Coding Total Score of the RBANS ranges from 0 to 89, with a higher score representing a better outcome.
Time Frame: Baseline, Week 24, Week 48, Week 72, Week 96
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | ABBV-8E12 300 mg | ABBV-8E12 1000 mg | ABBV-8E12 2000 mg
Number analyzed (Participants) | 116 | 108 | 116 | 113
score on a scale
  Change to Week 24: number analyzed (Participants) | 109 | 105 | 110 | 100
  Change to Week 24 | -0.39 (0.600) | -1.29 (0.611) | -1.40 (0.595) | -1.40 (0.623)
  Change to Week 48: number analyzed (Participants) | 98 | 90 | 103 | 90
  Change to Week 48 | -1.98 (0.673) | -1.17 (0.694) | -2.38 (0.660) | -3.14 (0.698)
  Change to Week 72: number analyzed (Participants) | 95 | 89 | 91 | 88
  Change to Week 72 | -5.26 (0.799) | -2.80 (0.819) | -4.58 (0.799) | -4.53 (0.828)
  Change to Week 96: number analyzed (Participants) | 77 | 76 | 80 | 65
  Change to Week 96 | -6.12 (0.957) | -6.95 (0.970) | -6.70 (0.940) | -7.30 (1.016)
Statistical Analysis 1: Comparison: Placebo vs ABBV-8E12 300 mg; Week 24; Test type: Superiority; p = 0.287, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.90, 95% CI 2-sided [-2.567 to 0.762], Standard Error of Mean 0.846
Statistical Analysis 2: Comparison: Placebo vs ABBV-8E12 300 mg; Week 24; Test type: Superiority; Effect size/pooled SD = -0.13, Standard Deviation 6.76 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 24; Test type: Superiority; p = 0.227, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -1.01, 95% CI 2-sided [-2.661 to 0.633], Standard Error of Mean 0.838
Statistical Analysis 4: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 24; Test type: Superiority; Effect size/pooled SD = -0.15, Standard Deviation 6.83 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 5: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 24; Test type: Superiority; p = 0.241, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -1.01, 95% CI 2-sided [-2.698 to 0.681], Standard Error of Mean 0.859
Statistical Analysis 6: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 24; Test type: Superiority; Effect size/pooled SD = -0.16, Standard Deviation 6.22 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 7: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; p = 0.397, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = 0.81, 95% CI 2-sided [-1.073 to 2.696], Standard Error of Mean 0.958
Statistical Analysis 8: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.11, Standard Deviation 7.45 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 9: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; p = 0.671, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.40, 95% CI 2-sided [-2.239 to 1.443], Standard Error of Mean 0.936
Statistical Analysis 10: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = -0.05, Standard Deviation 7.59 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 11: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Superiority; p = 0.231, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -1.16, 95% CI 2-sided [-3.052 to 0.738], Standard Error of Mean 0.964
Statistical Analysis 12: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = -0.16, Standard Deviation 7.25 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 13: Comparison: Placebo vs ABBV-8E12 300 mg; Week 72; Test type: Superiority; p = 0.031, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = 2.47, 95% CI 2-sided [0.230 to 4.701], Standard Error of Mean 1.137
Statistical Analysis 14: Comparison: Placebo vs ABBV-8E12 300 mg; Week 72; Test type: Superiority; Effect size/pooled SD = 0.29, Standard Deviation 8.65 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 15: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 72; Test type: Superiority; p = 0.547, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = 0.68, 95% CI 2-sided [-1.532 to 2.888], Standard Error of Mean 1.124
Statistical Analysis 16: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 72; Test type: Superiority; Effect size/pooled SD = 0.07, Standard Deviation 9.10 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 17: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 72; Test type: Superiority; p = 0.524, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = 0.73, 95% CI 2-sided [-1.521 to 2.984], Standard Error of Mean 1.145
Statistical Analysis 18: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 72; Test type: Superiority; Effect size/pooled SD = 0.09, Standard Deviation 8.42 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 19: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; p = 0.540, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.83, 95% CI 2-sided [-3.499 to 1.836], Standard Error of Mean 1.356
Statistical Analysis 20: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; Effect size/pooled SD = -0.08, Standard Deviation 10.02 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 21: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; p = 0.664, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.58, 95% CI 2-sided [-3.208 to 2.046], Standard Error of Mean 1.336
Statistical Analysis 22: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = -0.06, Standard Deviation 10.16 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 23: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; p = 0.393, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -1.19, 95% CI 2-sided [-3.923 to 1.546], Standard Error of Mean 1.390
Statistical Analysis 24: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = -0.13, Standard Deviation 9.48 — [estimate comment as in outcome 30, analysis 2]

34. Secondary Outcome: Change From Baseline Over Time in RBANS - Digit Span Total Score
Description: The RBANS is a 25-minute, standardized neurocognitive battery with North American population-based normative data. The RBANS measures five neurocognitive domains, with age-based scaling. Twelve subtests measure cognitive decline or improvement across the following domains: 1. Immediate Memory - List Learning and Story Memory, 2. Visuospatial/Constructional - Figure Copy and Line Orientation, 3. Language - Picture naming and Semantic Fluency, 4. Attention - Digit Span and Coding, and 5. Delayed Memory - List Recall, List Recognition, Story Memory, and Figure Recall. The Digit Span Total Score of the RBANS ranges from 0 to 8, with a higher score representing a better outcome.
Time Frame: Baseline, Week 24, Week 48, Week 72, Week 96
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | ABBV-8E12 300 mg | ABBV-8E12 1000 mg | ABBV-8E12 2000 mg
Number analyzed (Participants) | 116 | 108 | 116 | 113
score on a scale
  Change to Week 24: number analyzed (Participants) | 111 | 106 | 112 | 102
  Change to Week 24 | -0.48 (0.185) | -0.50 (0.189) | -0.78 (0.184) | -0.64 (0.193)
  Change to Week 48: number analyzed (Participants) | 101 | 91 | 105 | 93
  Change to Week 48 | -0.75 (0.207) | -0.65 (0.217) | -0.41 (0.204) | -0.65 (0.216)
  Change to Week 72: number analyzed (Participants) | 100 | 92 | 96 | 95
  Change to Week 72 | -0.94 (0.194) | -0.89 (0.201) | -1.13 (0.196) | -0.79 (0.199)
  Change to Week 96: number analyzed (Participants) | 81 | 79 | 85 | 73
  Change to Week 96 | -1.07 (0.229) | -0.81 (0.232) | -0.83 (0.224) | -0.90 (0.239)
Statistical Analysis 1: Comparison: Placebo vs ABBV-8E12 300 mg; Week 24; Test type: Superiority; p = 0.946, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.02, 95% CI 2-sided [-0.534 to 0.498], Standard Error of Mean 0.262
Statistical Analysis 2: Comparison: Placebo vs ABBV-8E12 300 mg; Week 24; Test type: Superiority; Effect size/pooled SD = -0.01, Standard Deviation 2.13 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 24; Test type: Superiority; p = 0.242, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.30, 95% CI 2-sided [-0.813 to 0.206], Standard Error of Mean 0.259
Statistical Analysis 4: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 24; Test type: Superiority; Effect size/pooled SD = -0.14, Standard Deviation 2.12 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 5: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 24; Test type: Superiority; p = 0.541, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.16, 95% CI 2-sided [-0.685 to 0.360], Standard Error of Mean 0.266
Statistical Analysis 6: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 24; Test type: Superiority; Effect size/pooled SD = -0.07, Standard Deviation 2.30 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 7: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; p = 0.724, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = 0.11, 95% CI 2-sided [-0.481 to 0.691], Standard Error of Mean 0.298
Statistical Analysis 8: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.04, Standard Deviation 2.36 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 9: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; p = 0.236, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = 0.34, 95% CI 2-sided [-0.226 to 0.913], Standard Error of Mean 0.290
Statistical Analysis 10: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.17, Standard Deviation 2.03 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 11: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Superiority; p = 0.714, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = 0.11, 95% CI 2-sided [-0.477 to 0.695], Standard Error of Mean 0.298
Statistical Analysis 12: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.05, Standard Deviation 2.11 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 13: Comparison: Placebo vs ABBV-8E12 300 mg; Week 72; Test type: Superiority; p = 0.860, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = 0.05, 95% CI 2-sided [-0.496 to 0.593], Standard Error of Mean 0.277
Statistical Analysis 14: Comparison: Placebo vs ABBV-8E12 300 mg; Week 72; Test type: Superiority; Effect size/pooled SD = 0.02, Standard Deviation 2.08 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 15: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 72; Test type: Superiority; p = 0.476, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.20, 95% CI 2-sided [-0.733 to 0.343], Standard Error of Mean 0.274
Statistical Analysis 16: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 72; Test type: Superiority; Effect size/pooled SD = -0.10, Standard Deviation 2.00 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 17: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 72; Test type: Superiority; p = 0.586, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = 0.15, 95% CI 2-sided [-0.393 to 0.694], Standard Error of Mean 0.276
Statistical Analysis 18: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 72; Test type: Superiority; Effect size/pooled SD = 0.08, Standard Deviation 1.97 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 19: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; p = 0.412, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = 0.27, 95% CI 2-sided [-0.371 to 0.903], Standard Error of Mean 0.324
Statistical Analysis 20: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; Effect size/pooled SD = 0.12, Standard Deviation 2.20 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 21: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; p = 0.450, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = 0.24, 95% CI 2-sided [-0.386 to 0.868], Standard Error of Mean 0.319
Statistical Analysis 22: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = 0.11, Standard Deviation 2.23 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 23: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; p = 0.612, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = 0.17, 95% CI 2-sided [-0.481 to 0.816], Standard Error of Mean 0.330
Statistical Analysis 24: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = 0.08, Standard Deviation 2.10 — [estimate comment as in outcome 30, analysis 2]

35. Secondary Outcome: Change From Baseline Over Time in RBANS - Figure Copy Total Score
Description: The RBANS is a 25-minute, standardized neurocognitive battery with North American population-based normative data. The RBANS measures five neurocognitive domains, with age-based scaling. Twelve subtests measure cognitive decline or improvement across the following domains: 1. Immediate Memory - List Learning and Story Memory, 2. Visuospatial/Constructional - Figure Copy and Line Orientation, 3. Language - Picture naming and Semantic Fluency, 4. Attention - Digit Span and Coding, and 5. Delayed Memory - List Recall, List Recognition, Story Memory, and Figure Recall. The Figure Copy Total Score of the RBANS ranges from 0 to 20, with a higher score representing a better outcome.
Time Frame: Baseline, Week 24, Week 48, Week 72, Week 96
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | ABBV-8E12 300 mg | ABBV-8E12 1000 mg | ABBV-8E12 2000 mg
Number analyzed (Participants) | 116 | 108 | 116 | 113
score on a scale
  Change to Week 24: number analyzed (Participants) | 111 | 106 | 112 | 102
  Change to Week 24 | 0.29 (0.287) | 0.03 (0.293) | -0.12 (0.284) | -0.20 (0.299)
  Change to Week 48: number analyzed (Participants) | 102 | 91 | 105 | 93
  Change to Week 48 | 0.07 (0.363) | -0.60 (0.380) | -0.01 (0.359) | -0.38 (0.379)
  Change to Week 72: number analyzed (Participants) | 100 | 92 | 97 | 93
  Change to Week 72 | -0.57 (0.410) | -0.77 (0.426) | -1.04 (0.412) | -1.25 (0.425)
  Change to Week 96: number analyzed (Participants) | 81 | 79 | 84 | 74
  Change to Week 96 | -1.63 (0.470) | -1.48 (0.480) | -1.29 (0.462) | -1.95 (0.490)
Statistical Analysis 1: Comparison: Placebo vs ABBV-8E12 300 mg; Week 24; Test type: Superiority; p = 0.520, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.26, 95% CI 2-sided [-1.058 to 0.535], Standard Error of Mean 0.405
Statistical Analysis 2: Comparison: Placebo vs ABBV-8E12 300 mg; Week 24; Test type: Superiority; Effect size/pooled SD = -0.07, Standard Deviation 3.52 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 24; Test type: Superiority; p = 0.303, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.41, 95% CI 2-sided [-1.201 to 0.374], Standard Error of Mean 0.401
Statistical Analysis 4: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 24; Test type: Superiority; Effect size/pooled SD = -0.13, Standard Deviation 3.28 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 5: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 24; Test type: Superiority; p = 0.230, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.50, 95% CI 2-sided [-1.307 to 0.315], Standard Error of Mean 0.412
Statistical Analysis 6: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 24; Test type: Superiority; Effect size/pooled SD = -0.14, Standard Deviation 3.53 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 7: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; p = 0.200, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.67, 95% CI 2-sided [-1.698 to 0.356], Standard Error of Mean 0.5222
Statistical Analysis 8: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; Effect size/pooled SD = -0.16, Standard Deviation 4.07 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 9: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; p = 0.873, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.08, 95% CI 2-sided [-1.080 to 0.917], Standard Error of Mean 0.508
Statistical Analysis 10: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = -0.02, Standard Deviation 4.13 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 11: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Superiority; p = 0.388, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.45, 95% CI 2-sided [-1.482 to 0.576], Standard Error of Mean 0.524
Statistical Analysis 12: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = -0.12, Standard Deviation 3.92 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 13: Comparison: Placebo vs ABBV-8E12 300 mg; Week 72; Test type: Superiority; p = 0.734, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.20, 95% CI 2-sided [-1.355 to 0.955], Standard Error of Mean 0.587
Statistical Analysis 14: Comparison: Placebo vs ABBV-8E12 300 mg; Week 72; Test type: Superiority; Effect size/pooled SD = -0.05, Standard Deviation 3.91 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 15: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 72; Test type: Superiority; p = 0.417, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.47, 95% CI 2-sided [-1.608 to 0.668], Standard Error of Mean 0.579
Statistical Analysis 16: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 72; Test type: Superiority; Effect size/pooled SD = -0.11, Standard Deviation 4.14 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 17: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 72; Test type: Superiority; p = 0.252, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.68, 95% CI 2-sided [-1.836 to 0.482], Standard Error of Mean 0.589
Statistical Analysis 18: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 72; Test type: Superiority; Effect size/pooled SD = -0.16, Standard Deviation 4.16 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 19: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; p = 0.827, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = 0.15, 95% CI 2-sided [-1.170 to 1.462], Standard Error of Mean 0.669
Statistical Analysis 20: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; Effect size/pooled SD = 0.03, Standard Deviation 4.69 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 21: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; p = 0.615, repeated measures model — Effect size at a specific visit is calculated as LS mean difference (8E12 - placebo) divided by pooled standard deviation of change scores for a ABBV-8E12 dose and placebo at that visit; LS Mean of Difference = 0.33, 95% CI 2-sided [-0.962 to 1.624], Standard Error of Mean 0.657
Statistical Analysis 22: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = 0.07, Standard Deviation 4.61
Statistical Analysis 23: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; p = 0.637, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.32, 95% CI 2-sided [-1.653 to 1.014], Standard Error of Mean 0.678
Statistical Analysis 24: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = -0.07, Standard Deviation 4.89 — [estimate comment as in outcome 30, analysis 2]

36. Secondary Outcome: Change From Baseline Over Time in RBANS - Figure Recall Total Score
Description: The RBANS is a 25-minute, standardized neurocognitive battery with North American population-based normative data. The RBANS measures five neurocognitive domains, with age-based scaling. Twelve subtests measure cognitive decline or improvement across the following domains: 1. Immediate Memory - List Learning and Story Memory, 2. Visuospatial/Constructional - Figure Copy and Line Orientation, 3. Language - Picture naming and Semantic Fluency, 4. Attention - Digit Span and Coding, and 5. Delayed Memory - List Recall, List Recognition, Story Memory, and Figure Recall. The Figure Recall Total Score of the RBANS ranges from 0 to 18, with a higher score representing a better outcome.
Time Frame: Baseline, Week 24, Week 48, Week 72, Week 96
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | ABBV-8E12 300 mg | ABBV-8E12 1000 mg | ABBV-8E12 2000 mg
Number analyzed (Participants) | 116 | 108 | 116 | 113
score on a scale
  Change to Week 24: number analyzed (Participants) | 110 | 106 | 112 | 102
  Change to Week 24 | -0.23 (0.259) | -0.65 (0.264) | 0.06 (0.256) | -0.60 (0.268)
  Change to Week 48: number analyzed (Participants) | 101 | 91 | 105 | 92
  Change to Week 48 | -0.97 (0.276) | -0.70 (0.288) | -0.22 (0.272) | -1.18 (0.288)
  Change to Week 72: number analyzed (Participants) | 99 | 90 | 97 | 92
  Change to Week 72 | -1.21 (0.262) | -1.16 (0.272) | -0.68 (0.263) | -1.45 (0.272)
  Change to Week 96: number analyzed (Participants) | 79 | 77 | 84 | 73
  Change to Week 96 | -1.16 (0.299) | -1.43 (0.305) | -0.86 (0.293) | -1.49 (0.310)
Statistical Analysis 1: Comparison: Placebo vs ABBV-8E12 300 mg; Week 24; Test type: Superiority; p = 0.261, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.41, 95% CI 2-sided [-1.135 to 0.308], Standard Error of Mean 0.367
Statistical Analysis 2: Comparison: Placebo vs ABBV-8E12 300 mg; Week 24; Test type: Superiority; Effect size/pooled SD = -0.13, Standard Deviation 3.12 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 24; Test type: Superiority; p = 0.423, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = 0.29, 95% CI 2-sided [-0.420 to 1.001], Standard Error of Mean 0.361
Statistical Analysis 4: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 24; Test type: Superiority; Effect size/pooled SD = 0.09, Standard Deviation 3.23 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 5: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 24; Test type: Superiority; p = 0.322, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.37, 95% CI 2-sided [-1.097 to 0.361], Standard Error of Mean 0.371
Statistical Analysis 6: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 24; Test type: Superiority; Effect size/pooled SD = -0.15, Standard Deviation 2.48 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 7: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; p = 0.498, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = 0.27, 95% CI 2-sided [-0.511 to 1.049], Standard Error of Mean 0.397
Statistical Analysis 8: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.08, Standard Deviation 3.33 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 9: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; p = 0.052, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = 0.75, 95% CI 2-sided [-0.006 to 1.510], Standard Error of Mean 0.386
Statistical Analysis 10: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.23, Standard Deviation 3.26 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 11: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Superiority; p = 0.597, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.21, 95% CI 2-sided [-0.993 to 0.572], Standard Error of Mean 0.398
Statistical Analysis 12: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = -0.08, Standard Deviation 2.57 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 13: Comparison: Placebo vs ABBV-8E12 300 mg; Week 72; Test type: Superiority; p = 0.896, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = 0.05, 95% CI 2-sided [-0.689 to 0.788], Standard Error of Mean 0.376
Statistical Analysis 14: Comparison: Placebo vs ABBV-8E12 300 mg; Week 72; Test type: Superiority; Effect size/pooled SD = 0.01, Standard Deviation 3.40
Statistical Analysis 15: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 72; Test type: Superiority; p = 0.149, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = 0.53, 95% CI 2-sided [-0.192 to 1.258], Standard Error of Mean 0.369
Statistical Analysis 16: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 72; Test type: Superiority; Effect size/pooled SD = 0.18, Standard Deviation 3.00 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 17: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 72; Test type: Superiority; p = 0.522, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.24, 95% CI 2-sided [-0.980 to 0.499], Standard Error of Mean 0.376
Statistical Analysis 18: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 72; Test type: Superiority; Effect size/pooled SD = -0.09, Standard Deviation 2.82 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 19: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; p = 0.528, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.27, 95% CI 2-sided [-1.103 to 0.567], Standard Error of Mean 0.424
Statistical Analysis 20: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; Effect size/pooled SD = -0.07, Standard Deviation 3.63 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 21: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; p = 0.474, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = 0.30, 95% CI 2-sided [-0.519 to 1.116], Standard Error of Mean 0.416
Statistical Analysis 22: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = 0.09, Standard Deviation 3.20 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 23: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; p = 0.441, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.33, 95% CI 2-sided [-1.176 to 0.513], Standard Error of Mean 0.429
Statistical Analysis 24: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = -0.11, Standard Deviation 3.02 — [estimate comment as in outcome 30, analysis 2]

37. Secondary Outcome: Change From Baseline Over Time in RBANS - List Recognition Total Score
Description: The RBANS is a 25-minute, standardized neurocognitive battery with North American population-based normative data. The RBANS measures five neurocognitive domains, with age-based scaling. Twelve subtests measure cognitive decline or improvement across the following domains: 1. Immediate Memory - List Learning and Story Memory, 2. Visuospatial/Constructional - Figure Copy and Line Orientation, 3. Language - Picture naming and Semantic Fluency, 4. Attention - Digit Span and Coding, and 5. Delayed Memory - List Recall, List Recognition, Story Memory, and Figure Recall. The List Recognition Total Score of the RBANS ranges from 0 to 20, with a higher score representing a better outcome.
Time Frame: Baseline, Week 24, Week 48, Week 72, Week 96
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | ABBV-8E12 300 mg | ABBV-8E12 1000 mg | ABBV-8E12 2000 mg
Number analyzed (Participants) | 116 | 108 | 116 | 113
score on a scale
  Change to Week 24: number analyzed (Participants) | 111 | 106 | 112 | 102
  Change to Week 24 | 0.09 (0.233) | -0.64 (0.238) | -0.38 (0.232) | -0.79 (0.242)
  Change to Week 48: number analyzed (Participants) | 101 | 91 | 105 | 93
  Change to Week 48 | 0.31 (0.231) | 0.29 (0.242) | 0.41 (0.227) | -0.23 (0.239)
  Change to Week 72: number analyzed (Participants) | 100 | 92 | 97 | 94
  Change to Week 72 | 0.13 (0.253) | -0.55 (0.262) | -0.48 (0.256) | -0.43 (0.260)
  Change to Week 96: number analyzed (Participants) | 80 | 79 | 85 | 74
  Change to Week 96 | -1.11 (0.279) | -1.42 (0.281) | -0.90 (0.271) | -1.04 (0.289)
Statistical Analysis 1: Comparison: Placebo vs ABBV-8E12 300 mg; Week 24; Test type: Superiority; p = 0.027, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.73, 95% CI 2-sided [-1.383 to -0.082], Standard Error of Mean 0.331
Statistical Analysis 2: Comparison: Placebo vs ABBV-8E12 300 mg; Week 24; Test type: Superiority; Effect size/pooled SD = -0.26, Standard Deviation 2.81 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 24; Test type: Superiority; p = 0.146, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.48, 95% CI 2-sided [-1.123 to 0.167], Standard Error of Mean 0.328
Statistical Analysis 4: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 24; Test type: Superiority; Effect size/pooled SD = -0.16, Standard Deviation 2.97 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 5: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 24; Test type: Superiority; p = 0.009, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.88, 95% CI 2-sided [-1.537 to -0.220], Standard Error of Mean 0.335
Statistical Analysis 6: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 24; Test type: Superiority; Effect size/pooled SD = -0.31, Standard Deviation 2.87 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 7: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; p = 0.952, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.02, 95% CI 2-sided [-0.674 to 0.634], Standard Error of Mean 0.333
Statistical Analysis 8: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; Effect size/pooled SD = -0.01, Standard Deviation 3.01 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 9: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; p = 0.764, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = 0.10, 95% CI 2-sided [-0.540 to 0.734], Standard Error of Mean 0.324
Statistical Analysis 10: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.03, Standard Deviation 2.85
Statistical Analysis 11: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Superiority; p = 0.103, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.54, 95% CI 2-sided [-1.191 to 0.109], Standard Error of Mean 0.331
Statistical Analysis 12: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = -0.19, Standard Deviation 2.83 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 13: Comparison: Placebo vs ABBV-8E12 300 mg; Week 72; Test type: Superiority; p = 0.060, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.68, 95% CI 2-sided [-1.396 to 0.028], Standard Error of Mean 0.362
Statistical Analysis 14: Comparison: Placebo vs ABBV-8E12 300 mg; Week 72; Test type: Superiority; Effect size/pooled SD = -0.22, Standard Deviation 3.09 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 15: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 72; Test type: Superiority; p = 0.091, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.61, 95% CI 2-sided [-1.316 to 0.098], Standard Error of Mean 0.360
Statistical Analysis 16: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 72; Test type: Superiority; Effect size/pooled SD = -0.20, Standard Deviation 3.03
Statistical Analysis 17: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 72; Test type: Superiority; p = 0.120, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.56, 95% CI 2-sided [-1.274 to 0.147], Standard Error of Mean 0.361
Statistical Analysis 18: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 72; Test type: Superiority; Effect size/pooled SD = -0.19, Standard Deviation 2.92 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 19: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; p = 0.429, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.31, 95% CI 2-sided [-1.090 to 0.464], Standard Error of Mean 0.395
Statistical Analysis 20: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; Effect size/pooled SD = -0.10, Standard Deviation 3.13
Statistical Analysis 21: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; p = 0.597, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = 0.21, 95% CI 2-sided [-0.559 to 0.970], Standard Error of Mean 0.389
Statistical Analysis 22: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = 0.07, Standard Deviation 2.98 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 23: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; p = 0.860, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = 0.07, 95% CI 2-sided [-0.717 to 0.858], Standard Error of Mean 0.400
Statistical Analysis 24: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = 0.02, Standard Deviation 3.22 — [estimate comment as in outcome 30, analysis 2]

38. Secondary Outcome: Change From Baseline Over Time in RBANS - List Learning Total Score
Description: The RBANS is a 25-minute, standardized neurocognitive battery with North American population-based normative data. The RBANS measures five neurocognitive domains, with age-based scaling. Twelve subtests measure cognitive decline or improvement across the following domains: 1. Immediate Memory - List Learning and Story Memory, 2. Visuospatial/Constructional - Figure Copy and Line Orientation, 3. Language - Picture naming and Semantic Fluency, 4. Attention - Digit Span and Coding, and 5. Delayed Memory - List Recall, List Recognition, Story Memory, and Figure Recall. The List Learning Total Score of the RBANS ranges from 0 to 40, with a higher score representing a better outcome.
Time Frame: Baseline, Week 24, Week 48, Week 72, Week 96
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | ABBV-8E12 300 mg | ABBV-8E12 1000 mg | ABBV-8E12 2000 mg
Number analyzed (Participants) | 116 | 108 | 116 | 113
score on a scale
  Change to Week 24: number analyzed (Participants) | 111 | 106 | 112 | 102
  Change to Week 24 | -0.57 (0.350) | -0.67 (0.359) | -0.98 (0.348) | -1.14 (0.364)
  Change to Week 48: number analyzed (Participants) | 102 | 91 | 105 | 93
  Change to Week 48 | -1.27 (0.397) | -0.36 (0.416) | -1.89 (0.392) | -1.17 (0.413)
  Change to Week 72: number analyzed (Participants) | 100 | 92 | 97 | 95
  Change to Week 72 | -3.18 (0.413) | -3.32 (0.428) | -3.02 (0.415) | -3.11 (0.424)
  Change to Week 96: number analyzed (Participants) | 82 | 79 | 87 | 75
  Change to Week 96 | -3.57 (0.484) | -2.93 (0.496) | -3.23 (0.474) | -3.07 (0.503)
Statistical Analysis 1: Comparison: Placebo vs ABBV-8E12 300 mg; Week 24; Test type: Superiority; p = 0.854, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.09, 95% CI 2-sided [-1.069 to 0.885], Standard Error of Mean 0.497
Statistical Analysis 2: Comparison: Placebo vs ABBV-8E12 300 mg; Week 24; Test type: Superiority; Effect size/pooled SD = -0.02, Standard Deviation 4.02 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 24; Test type: Superiority; p = 0.412, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.40, 95% CI 2-sided [-1.368 to 0.562], Standard Error of Mean 0.491
Statistical Analysis 4: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 24; Test type: Superiority; Effect size/pooled SD = -0.10, Standard Deviation 4.08 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 5: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 24; Test type: Superiority; p = 0.262, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.57, 95% CI 2-sided [-1.554 to 0.424], Standard Error of Mean 0.503
Statistical Analysis 6: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 24; Test type: Superiority; Effect size/pooled SD = -0.15, Standard Deviation 3.82 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 7: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; p = 0.110, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = 0.91, 95% CI 2-sided [-0.209 to 2.036], Standard Error of Mean 0.571
Statistical Analysis 8: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.22, Standard Deviation 4.09 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 9: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; p = 0.263, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.62, 95% CI 2-sided [-1.713 to 0.469], Standard Error of Mean 0.555
Statistical Analysis 10: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = -0.15, Standard Deviation 4.21 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 11: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Superiority; p = 0.868, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = 0.10, 95% CI 2-sided [-1.026 to 1.217], Standard Error of Mean 0.570
Statistical Analysis 12: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.02, Standard Deviation 3.92 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 13: Comparison: Placebo vs ABBV-8E12 300 mg; Week 72; Test type: Superiority; p = 0.820, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.13, 95% CI 2-sided [-1.298 to 1.029], Standard Error of Mean 0.592
Statistical Analysis 14: Comparison: Placebo vs ABBV-8E12 300 mg; Week 72; Test type: Superiority; Effect size/pooled SD = -0.03, Standard Deviation 4.49 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 15: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 72; Test type: Superiority; p = 0.781, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = 0.16, 95% CI 2-sided [-0.984 to 1.308], Standard Error of Mean 0.583
Statistical Analysis 16: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 72; Test type: Superiority; Effect size/pooled SD = 0.04, Standard Deviation 4.49 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 17: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 72; Test type: Superiority; p = 0.895, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = 0.08, 95% CI 2-sided [-1.082 to 1.238], Standard Error of Mean 0.590
Statistical Analysis 18: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 72; Test type: Superiority; Effect size/pooled SD = 0.02, Standard Deviation 4.75 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 19: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; p = 0.359, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = 0.63, 95% CI 2-sided [-0.724 to 1.991], Standard Error of Mean 0.690
Statistical Analysis 20: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; Effect size/pooled SD = 0.14, Standard Deviation 4.55 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 21: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; p = 0.612, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = 0.34, 95% CI 2-sided [-0.985 to 1.670], Standard Error of Mean 0.675
Statistical Analysis 22: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = 0.07, Standard Deviation 4.72 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 23: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; p = 0.475, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = 0.50, 95% CI 2-sided [-0.872 to 1.867], Standard Error of Mean 0.696
Statistical Analysis 24: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = 0.11, Standard Deviation 4.57 — [estimate comment as in outcome 30, analysis 2]

39. Secondary Outcome: Change From Baseline Over Time in RBANS - Line Orientation Total Score
Description: The RBANS is a 25-minute, standardized neurocognitive battery with North American population-based normative data. The RBANS measures five neurocognitive domains, with age-based scaling. Twelve subtests measure cognitive decline or improvement across the following domains: 1. Immediate Memory - List Learning and Story Memory, 2. Visuospatial/Constructional - Figure Copy and Line Orientation, 3. Language - Picture naming and Semantic Fluency, 4. Attention - Digit Span and Coding, and 5. Delayed Memory - List Recall, List Recognition, Story Memory, and Figure Recall. The Line Orientation Total Score of the RBANS ranges from 0 to 20, with a higher score representing a better outcome.
Time Frame: Baseline, Week 24, Week 48, Week 72, Week 96
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | ABBV-8E12 300 mg | ABBV-8E12 1000 mg | ABBV-8E12 2000 mg
Number analyzed (Participants) | 116 | 108 | 116 | 113
score on a scale
  Change to Week 24: number analyzed (Participants) | 111 | 106 | 110 | 102
  Change to Week 24 | 0.20 (0.301) | 0.24 (0.308) | -0.05 (0.301) | 0.03 (0.313)
  Change to Week 48: number analyzed (Participants) | 101 | 91 | 104 | 92
  Change to Week 48 | -0.84 (0.348) | 0.05 (0.363) | -0.53 (0.344) | -0.47 (0.363)
  Change to Week 72: number analyzed (Participants) | 100 | 92 | 95 | 94
  Change to Week 72 | -0.64 (0.365) | -0.07 (0.378) | -0.60 (0.369) | -0.60 (0.377)
  Change to Week 96: number analyzed (Participants) | 77 | 79 | 84 | 69
  Change to Week 96 | -1.33 (0.404) | -1.01 (0.405) | -0.99 (0.392) | -1.88 (0.424)
Statistical Analysis 1: Comparison: Placebo vs ABBV-8E12 300 mg; Week 24; Test type: Superiority; p = 0.926, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = 0.04, 95% CI 2-sided [-0.799 to 0.878], Standard Error of Mean 0.427
Statistical Analysis 2: Comparison: Placebo vs ABBV-8E12 300 mg; Week 24; Test type: Superiority; Effect size/pooled SD = 0.01, Standard Deviation 3.78 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 24; Test type: Superiority; p = 0.553, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.25, 95% CI 2-sided [-1.082 to 0.580], Standard Error of Mean 0.423
Statistical Analysis 4: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 24; Test type: Superiority; Effect size/pooled SD = -0.06, Standard Deviation 3.96 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 5: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 24; Test type: Superiority; p = 0.690, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.17, 95% CI 2-sided [-1.021 to 0.677], Standard Error of Mean 0.432
Statistical Analysis 6: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 24; Test type: Superiority; Effect size/pooled SD = -0.04, Standard Deviation 4.13 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 7: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; p = 0.073, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = 0.90, 95% CI 2-sided [-0.085 to 1.879], Standard Error of Mean 0.499
Statistical Analysis 8: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.22, Standard Deviation 4.03 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 9: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; p = 0.517, repeated measures model — [p-value comment as in outcome 35, analysis 21]; LS Mean of Difference = 0.32, 95% CI 2-sided [-0.641 to 1.273], Standard Error of Mean 0.487
Statistical Analysis 10: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.07, Standard Deviation 4.21 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 11: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Superiority; p = 0.454, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = 0.38, 95% CI 2-sided [-0.609 to 1.360], Standard Error of Mean 0.501
Statistical Analysis 12: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.08, Standard Deviation 4.45
Statistical Analysis 13: Comparison: Placebo vs ABBV-8E12 300 mg; Week 72; Test type: Superiority; p = 0.276, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = 0.57, 95% CI 2-sided [-0.456 to 1.596], Standard Error of Mean 0.522
Statistical Analysis 14: Comparison: Placebo vs ABBV-8E12 300 mg; Week 72; Test type: Superiority; Effect size/pooled SD = 0.14, Standard Deviation 3.94 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 15: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 72; Test type: Superiority; p = 0.935, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = 0.04, 95% CI 2-sided [-0.973 to 1.058], Standard Error of Mean 0.516
Statistical Analysis 16: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 72; Test type: Superiority; Effect size/pooled SD = 0.01, Standard Deviation 4.35 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 17: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 72; Test type: Superiority; p = 0.942, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = 0.04, 95% CI 2-sided [-0.990 to 1.066], Standard Error of Mean 0.523
Statistical Analysis 18: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 72; Test type: Superiority; Effect size/pooled SD = 0.01, Standard Deviation 4.35 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 19: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; p = 0.578, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = 0.32, 95% CI 2-sided [-0.802 to 1.436], Standard Error of Mean 0.569
Statistical Analysis 20: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; Effect size/pooled SD = 0.09, Standard Deviation 3.57 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 21: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; p = 0.545, repeated measures model — [p-value comment as in outcome 35, analysis 21]; LS Mean of Difference = 0.560, 95% CI 2-sided [-0.762 to 1.441], Standard Error of Mean 0.34
Statistical Analysis 22: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = 0.09, Standard Deviation 3.94 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 23: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; p = 0.346, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.55, 95% CI 2-sided [-1.697 to 0.597], Standard Error of Mean 0.583
Statistical Analysis 24: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = -0.14, Standard Deviation 3.81 — [estimate comment as in outcome 30, analysis 2]

40. Secondary Outcome: Change From Baseline Over Time in RBANS - List Recall Total Score
Description: The RBANS is a 25-minute, standardized neurocognitive battery with North American population-based normative data. The RBANS measures five neurocognitive domains, with age-based scaling. Twelve subtests measure cognitive decline or improvement across the following domains: 1. Immediate Memory - List Learning and Story Memory, 2. Visuospatial/Constructional - Figure Copy and Line Orientation, 3. Language - Picture naming and Semantic Fluency, 4. Attention - Digit Span and Coding, and 5. Delayed Memory - List Recall, List Recognition, Story Memory, and Figure Recall. The List Recall Total Score of the RBANS ranges from 0 to 10, with a higher score representing a better outcome.
Time Frame: Baseline, Week 24, Week 48, Week 72, Week 96
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | ABBV-8E12 300 mg | ABBV-8E12 1000 mg | ABBV-8E12 2000 mg
Number analyzed (Participants) | 116 | 108 | 116 | 113
score on a scale
  Change to Week 24: number analyzed (Participants) | 111 | 106 | 112 | 102
  Change to Week 24 | 0.04 (0.102) | -0.15 (0.105) | -0.01 (0.102) | -0.08 (0.106)
  Change to Week 48: number analyzed (Participants) | 101 | 91 | 105 | 93
  Change to Week 48 | 0.07 (0.120) | 0.05 (0.125) | 0.10 (0.118) | -0.10 (0.124)
  Change to Week 72: number analyzed (Participants) | 100 | 92 | 97 | 95
  Change to Week 72 | 0.01 (0.081) | -0.29 (0.084) | -0.24 (0.082) | -0.27 (0.083)
  Change to Week 96: number analyzed (Participants) | 80 | 79 | 86 | 75
  Change to Week 96 | -0.14 (0.095) | -0.39 (0.096) | -0.35 (0.092) | -0.31 (0.098)
Statistical Analysis 1: Comparison: Placebo vs ABBV-8E12 300 mg; Week 24; Test type: Superiority; p = 0.202, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.19, 95% CI 2-sided [-0.473 to 0.100], Standard Error of Mean 0.146
Statistical Analysis 2: Comparison: Placebo vs ABBV-8E12 300 mg; Week 24; Test type: Superiority; Effect size/pooled SD = -0.15, Standard Deviation 1.26 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 24; Test type: Superiority; p = 0.760, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.04, 95% CI 2-sided [-0.327 to 0.239], Standard Error of Mean 0.144
Statistical Analysis 4: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 24; Test type: Superiority; Effect size/pooled SD = -0.04, Standard Deviation 1.15 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 5: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 24; Test type: Superiority; p = 0.419, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.12, 95% CI 2-sided [-0.409 to 0.170], Standard Error of Mean 0.147
Statistical Analysis 6: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 24; Test type: Superiority; Effect size/pooled SD = -0.12, Standard Deviation 1.03 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 7: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; p = 0.893, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.02, 95% CI 2-sided [-0.363 to 0.317], Standard Error of Mean 0.173
Statistical Analysis 8: Comparison: Placebo vs ABBV-8E12 300 mg; Test type: Superiority; Effect size/pooled SD = -0.02, Standard Deviation 1.26 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 9: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; p = 0.886, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = 0.02, 95% CI 2-sided [-0.306 to 0.354], Standard Error of Mean 0.168
Statistical Analysis 10: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.02, Standard Deviation 1.46 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 11: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Superiority; p = 0.306, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.18, 95% CI 2-sided [-0.515 to 0.162], Standard Error of Mean 0.172
Statistical Analysis 12: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = -0.16, Standard Deviation 1.12 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 13: Comparison: Placebo vs ABBV-8E12 300 mg; Week 72; Test type: Superiority; p = 0.008, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.31, 95% CI 2-sided [-0.535 to -0.079], Standard Error of Mean 0.116
Statistical Analysis 14: Comparison: Placebo vs ABBV-8E12 300 mg; Week 72; Test type: Superiority; Effect size/pooled SD = -0.26, Standard Deviation 1.20 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 15: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 72; Test type: Superiority; p = 0.031, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.25, 95% CI 2-sided [-0.474 to -0.023], Standard Error of Mean 0.115
Statistical Analysis 16: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 72; Test type: Superiority; Effect size/pooled SD = -0.21, Standard Deviation 1.16 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 17: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 72; Test type: Superiority; p = 0.014, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.29, 95% CI 2-sided [-0.514 to -0.059], Standard Error of Mean 0.116
Statistical Analysis 18: Comparison: Placebo vs ABBV-8E12 2000 mg; Test type: Superiority; Effect size/pooled SD = -0.25, Standard Deviation 1.15 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 19: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; p = 0.065, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.25, 95% CI 2-sided [-0.514 to 0.016], Standard Error of Mean 0.135
Statistical Analysis 20: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; Effect size/pooled SD = -0.21, Standard Deviation 1.17 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 21: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; p = 0.121, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.21, 95% CI 2-sided [-0.465 to 0.055], Standard Error of Mean 0.132
Statistical Analysis 22: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = 1.05, Standard Deviation 1.17 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 23: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; p = 0.210, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.17, 95% CI 2-sided [-0.438 to 0.097], Standard Error of Mean 0.136
Statistical Analysis 24: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = -0.17, Standard Deviation 1.00 — [estimate comment as in outcome 30, analysis 2]

41. Secondary Outcome: Change From Baseline Over Time in RBANS - Picture Naming Total Score
Description: The RBANS is a 25-minute, standardized neurocognitive battery with North American population-based normative data. The RBANS measures five neurocognitive domains, with age-based scaling. Twelve subtests measure cognitive decline or improvement across the following domains: 1. Immediate Memory - List Learning and Story Memory, 2. Visuospatial/Constructional - Figure Copy and Line Orientation, 3. Language - Picture naming and Semantic Fluency, 4. Attention - Digit Span and Coding, and 5. Delayed Memory - List Recall, List Recognition, Story Memory, and Figure Recall. The Picture Naming Total Score of the RBANS ranges from 0 to 10, with a higher score representing a better outcome.
Time Frame: Baseline, Week 24, Week 48, Week 72, Week 96
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | ABBV-8E12 300 mg | ABBV-8E12 1000 mg | ABBV-8E12 2000 mg
Number analyzed (Participants) | 116 | 108 | 116 | 113
score on a scale
  Change to Week 24: number analyzed (Participants) | 111 | 106 | 112 | 102
  Change to Week 24 | -0.68 (0.132) | -0.87 (0.136) | -0.85 (0.132) | -0.86 (0.138)
  Change to Week 48: number analyzed (Participants) | 101 | 91 | 105 | 93
  Change to Week 48 | -0.21 (0.112) | -0.10 (0.117) | -0.09 (0.110) | -0.14 (0.116)
  Change to Week 72: number analyzed (Participants) | 100 | 92 | 97 | 95
  Change to Week 72 | -0.91 (0.162) | -0.81 (0.168) | -0.63 (0.163) | -0.75 (0.167)
  Change to Week 96: number analyzed (Participants) | 81 | 79 | 87 | 75
  Change to Week 96 | -0.68 (0.152) | -0.94 (0.155) | -0.65 (0.148) | -0.77 (0.157)
Statistical Analysis 1: Comparison: Placebo vs ABBV-8E12 300 mg; Week 24; Test type: Superiority; p = 0.303, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.19, 95% CI 2-sided [-0.564 to 0.176], Standard Error of Mean 0.188
Statistical Analysis 2: Comparison: Placebo vs ABBV-8E12 300 mg; Week 24; Test type: Superiority; Effect size/pooled SD = -0.14, Standard Deviation 1.42 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 24; Test type: Superiority; p = 0.358, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.17, 95% CI 2-sided [-0.536 to 0.194], Standard Error of Mean 0.186
Statistical Analysis 4: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 24; Test type: Superiority; Effect size/pooled SD = -0.13, Standard Error of Mean 1.31 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 5: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 24; Test type: Superiority; p = 0.347, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.18, 95% CI 2-sided [-0.553 to 0.195], Standard Error of Mean 0.190
Statistical Analysis 6: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 24; Test type: Superiority; Effect size/pooled SD = -0.15, Standard Deviation 1.21 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 7: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; p = 0.494, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = 0.11, 95% CI 2-sided [-0.205 to 0.423], Standard Error of Mean 0.160
Statistical Analysis 8: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.09, Standard Deviation 1.22 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 9: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; p = 0.454, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = 0.12, 95% CI 2-sided [-0.189 to 0.423], Standard Error of Mean 0.156
Statistical Analysis 10: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.10, Standard Deviation 1.13 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 11: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Superiority; p = 0.644, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = 0.07, 95% CI 2-sided [-0.240 to 0.388], Standard Deviation 0.160
Statistical Analysis 12: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.07, Standard Deviation 1.10 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 13: Comparison: Placebo vs ABBV-8E12 300 mg; Week 72; Test type: Superiority; p = 0.685, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = 0.09, 95% CI 2-sided [-0.363 to 0.551], Standard Error of Mean 0.232
Statistical Analysis 14: Comparison: Placebo vs ABBV-8E12 300 mg; Week 72; Test type: Superiority; Effect size/pooled SD = 0.06, Standard Deviation 1.64 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 15: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 72; Test type: Superiority; p = 0.219, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = 0.28, 95% CI 2-sided [-0.168 to 0.730], Standard Error of Mean 0.228
Statistical Analysis 16: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 72; Test type: Superiority; Effect size/pooled SD = 0.18, Standard Deviation 1.55 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 17: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 72; Test type: Superiority; p = 0.507, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = 0.15, 95% CI 2-sided [-0.302 to 0.610], Standard Error of Mean 0.232
Statistical Analysis 18: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 72; Test type: Superiority; Effect size/pooled SD = 0.10, Standard Deviation 1.49 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 19: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; p = 0.233, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.26, 95% CI 2-sided [-0.683 to 0.167], Standard Error of Mean 0.216
Statistical Analysis 20: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; Effect size/pooled SD = -0.20, Standard Deviation 1.27 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 21: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; p = 0.881, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = 0.03, 95% CI 2-sided [-0.383 to 0.446], Standard Error of Mean 0.211
Statistical Analysis 22: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = 0.02, Standard Deviation 1.42 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 23: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; p = 0.671, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.09, 95% CI 2-sided [-0.520 to 0.335], Standard Error of Mean 0.217
Statistical Analysis 24: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Other; Effect size/pooled SD = -0.08, Standard Deviation 1.20 — [estimate comment as in outcome 30, analysis 2]

42. Secondary Outcome: Change From Baseline Over Time in RBANS - Semantic Fluency Total Score
Description: The RBANS is a 25-minute, standardized neurocognitive battery with North American population-based normative data. The RBANS measures five neurocognitive domains, with age-based scaling. Twelve subtests measure cognitive decline or improvement across the following domains: 1. Immediate Memory - List Learning and Story Memory, 2. Visuospatial/Constructional - Figure Copy and Line Orientation, 3. Language - Picture naming and Semantic Fluency, 4. Attention - Digit Span and Coding, and 5. Delayed Memory - List Recall, List Recognition, Story Memory, and Figure Recall. The Semantic Fluency Total Score of the RBANS ranges from 0 to 40, with a higher score representing a better outcome.
Time Frame: Baseline, Week 24, Week 48, Week 72, Week 96
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | ABBV-8E12 300 mg | ABBV-8E12 1000 mg | ABBV-8E12 2000 mg
Number analyzed (Participants) | 116 | 108 | 116 | 113
score on a scale
  Change to Week 24: number analyzed (Participants) | 111 | 106 | 111 | 102
  Change to Week 24 | -1.47 (0.289) | -1.90 (0.296) | -1.48 (0.288) | -1.65 (0.300)
  Change to Week 48: number analyzed (Participants) | 101 | 91 | 105 | 92
  Change to Week 48 | -1.03 (0.441) | -1.00 (0.462) | -0.90 (0.434) | -0.79 (0.460)
  Change to Week 72: number analyzed (Participants) | 100 | 92 | 97 | 95
  Change to Week 72 | -4.07 (0.462) | -4.50 (0.480) | -4.38 (0.465) | -4.26 (0.475)
  Change to Week 96: number analyzed (Participants) | 81 | 79 | 87 | 74
  Change to Week 96 | -2.29 (0.408) | -2.87 (0.415) | -2.83 (0.397) | -2.78 (0.425)
Statistical Analysis 1: Comparison: Placebo vs ABBV-8E12 300 mg; Week 24; Test type: Superiority; p = 0.297, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.43, 95% CI 2-sided [-1.232 to 0.377], Standard Error of Mean 0.409
Statistical Analysis 2: Comparison: Placebo vs ABBV-8E12 300 mg; Week 24; Test type: Superiority; Effect size/pooled SD = -0.12, Standard Deviation 3.70 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 24; Test type: Superiority; p = 0.979, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.01, 95% CI 2-sided [-0.808 to 0.786], Standard Error of Mean 0.405
Statistical Analysis 4: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 24; Test type: Superiority; Effect size/pooled SD = -0.00, Standard Deviation 3.63 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 5: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 24; Test type: Superiority; p = 0.663, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.18, 95% CI 2-sided [-0.996 to 0.634], Standard Error of Mean 0.415
Statistical Analysis 6: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 24; Test type: Superiority; Effect size/pooled SD = -0.05, Standard Deviation 3.71 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 7: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; p = 0.961, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = 0.03, 95% CI 2-sided [-1.220 to 1.282], Standard Error of Mean 0.636
Statistical Analysis 8: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.01, Standard Deviation 4.88 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 9: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; p = 0.833, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = 0.13, 95% CI 2-sided [-1.083 to 1.344], Standard Error of Mean 0.617
Statistical Analysis 10: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.03, Standard Deviation 5.06 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 11: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Other; p = 0.714, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = 0.23, 95% CI 2-sided [-1.017 to 1.484], Standard Error of Mean 0.636
Statistical Analysis 12: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.05, Standard Deviation 5.13 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 13: Comparison: Placebo vs ABBV-8E12 300 mg; Week 72; Test type: Superiority; p = 0.518, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.43, 95% CI 2-sided [-1.733 to 0.876], Standard Error of Mean 0.663
Statistical Analysis 14: Comparison: Placebo vs ABBV-8E12 300 mg; Week 72; Test type: Superiority; Effect size/pooled SD = -0.08, Standard Deviation 5.17 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 15: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 72; Test type: Superiority; p = 0.633, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.31, 95% CI 2-sided [-1.598 to 0.973], Standard Error of Mean 0.654
Statistical Analysis 16: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 72; Test type: Superiority; Effect size/pooled SD = -0.06, Standard Deviation 4.90 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 17: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 72; Test type: Superiority; p = 0.776, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.19, 95% CI 2-sided [-1.488 to 1.112], Standard Error of Mean 0.661
Statistical Analysis 18: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 72; Test type: Superiority; Effect size/pooled SD = -0.04, Standard Deviation 4.93 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 19: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; p = 0.316, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.58, 95% CI 2-sided [-1.723 to 0.558], Standard Error of Mean 0.580
Statistical Analysis 20: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; Effect size/pooled SD = -0.15, Standard Deviation 4.01 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 21: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; p = 0.336, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.55, 95% CI 2-sided [-1.660 to 0.569], Standard Error of Mean 0.567
Statistical Analysis 22: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = -0.14, Standard Deviation 3.90 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 23: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; p = 0.403, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.49, 95% CI 2-sided [-1.647 to 0.663], Standard Error of Mean 0.587
Statistical Analysis 24: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = -0.13, Standard Deviation 3.92 — [estimate comment as in outcome 30, analysis 2]

43. Secondary Outcome: Change From Baseline Over Time in RBANS - Story Memory Total Score
Description: The RBANS is a 25-minute, standardized neurocognitive battery with North American population-based normative data. The RBANS measures five neurocognitive domains, with age-based scaling. Twelve subtests measure cognitive decline or improvement across the following domains: 1. Immediate Memory - List Learning and Story Memory, 2. Visuospatial/Constructional - Figure Copy and Line Orientation, 3. Language - Picture naming and Semantic Fluency, 4. Attention - Digit Span and Coding, and 5. Delayed Memory - List Recall, List Recognition, Story Memory, and Figure Recall. The Story Memory Total Score of the RBANS ranges from 0 to 24, with a higher score representing a better outcome.
Time Frame: Baseline, Week 24, Week 48, Week 72, Week 96
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | ABBV-8E12 300 mg | ABBV-8E12 1000 mg | ABBV-8E12 2000 mg
Number analyzed (Participants) | 116 | 108 | 116 | 113
score on a scale
  Change to Week 24: number analyzed (Participants) | 111 | 106 | 112 | 102
  Change to Week 24 | -3.06 (0.282) | -3.13 (0.289) | -2.93 (0.280) | -2.99 (0.293)
  Change to Week 48: number analyzed (Participants) | 102 | 91 | 105 | 93
  Change to Week 48 | -1.62 (0.324) | -1.07 (0.341) | -0.70 (0.320) | -1.01 (0.338)
  Change to Week 72: number analyzed (Participants) | 100 | 92 | 97 | 94
  Change to Week 72 | -2.15 (0.381) | -2.00 (0.396) | -1.84 (0.384) | -2.10 (0.393)
  Change to Week 96: number analyzed (Participants) | 82 | 79 | 86 | 74
  Change to Week 96 | -3.31 (0.380) | -2.67 (0.388) | -2.46 (0.372) | -2.45 (0.397)
Statistical Analysis 1: Comparison: Placebo vs ABBV-8E12 300 mg; Week 24; Test type: Superiority; p = 0.861, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.07, 95% CI 2-sided [-0.856 to 0.716], Standard Error of Mean 0.400
Statistical Analysis 2: Comparison: Placebo vs ABBV-8E12 300 mg; Week 24; Test type: Superiority; Effect size/pooled SD = -0.02, Standard Deviation 3.51 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 24; Test type: Superiority; p = 0.746, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = 0.13, 95% CI 2-sided [-0.648 to 0.905], Standard Error of Mean 0.395
Statistical Analysis 4: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 24; Test type: Superiority; Effect size/pooled SD = 0.04, Standard Deviation 3.46 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 5: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 24; Test type: Superiority; p = 0.859, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = 0.07, 95% CI 2-sided [-0.724 to 0.868], Standard Error of Mean 0.405
Statistical Analysis 6: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 24; Test type: Superiority; Effect size/pooled SD = 0.02, Standard Deviation 3.64 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 7: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; p = 0.240, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = 0.55, 95% CI 2-sided [-0.369 to 1.469], Standard Error of Mean 0.467
Statistical Analysis 8: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.16, Standard Deviation 3.41 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 9: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; p = 0.044, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = 0.91, 95% CI 2-sided [0.023 to 1.087], Standard Error of Mean 0.454
Statistical Analysis 10: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.26, Standard Deviation 3.51
Statistical Analysis 11: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Superiority; p = 0.195, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = 0.61, 95% CI 2-sided [-0.312 to 1.524], Standard Error of Mean 0.467
Statistical Analysis 12: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.17, Standard Deviation 3.53
Statistical Analysis 13: Comparison: Placebo vs ABBV-8E12 300 mg; Week 72; Test type: Superiority; p = 0.778, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = 0.15, 95% CI 2-sided [-0.921 to 1.229], Standard Error of Mean 0.547
Statistical Analysis 14: Comparison: Placebo vs ABBV-8E12 300 mg; Week 72; Test type: Other; Effect size/pooled SD = 0.04, Standard Deviation 3.99
Statistical Analysis 15: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 72; Test type: Superiority; p = 0.558, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = 0.32, 95% CI 2-sided [-0.743 to 1.376], Standard Error of Mean 0.539
Statistical Analysis 16: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 72; Test type: Superiority; Effect size/pooled SD = 0.08, Standard Deviation 3.89
Statistical Analysis 17: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 72; Test type: Superiority; p = 0.928, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = 0.05, 95% CI 2-sided [-1.025 to 1.124], Standard Error of Mean 0.546
Statistical Analysis 18: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 72; Test type: Superiority; Effect size/pooled SD = 0.01, Standard Deviation 4.27
Statistical Analysis 19: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; p = 0.238, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = 0.64, 95% CI 2-sided [-0.425 to 1.704], Standard Error of Mean 0.541
Statistical Analysis 20: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; Effect size/pooled SD = 0.18, Standard Deviation 3.61 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 21: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; p = 0.107, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = 0.86, 95% CI 2-sided [-0.186 to 1.898], Standard Error of Mean 0.530
Statistical Analysis 22: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = 0.25, Standard Deviation 3.41 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 23: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; p = 0.116, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = 0.86, 95% CI 2-sided [-0.214 to 1.942], Standard Error of Mean 0.548
Statistical Analysis 24: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = 0.23, Standard Deviation 3.75 — [estimate comment as in outcome 30, analysis 2]

44. Secondary Outcome: Change From Baseline Over Time in RBANS - Story Recall Total Score
Description: The RBANS is a 25-minute, standardized neurocognitive battery with North American population-based normative data. The RBANS measures five neurocognitive domains, with age-based scaling. Twelve subtests measure cognitive decline or improvement across the following domains: 1. Immediate Memory - List Learning and Story Memory, 2. Visuospatial/Constructional - Figure Copy and Line Orientation, 3. Language - Picture naming and Semantic Fluency, 4. Attention - Digit Span and Coding, and 5. Delayed Memory - List Recall, List Recognition, Story Memory, and Figure Recall. The Story Recall Total Score of the RBANS ranges from 0 to 12, with a higher score representing a better outcome.
Time Frame: Baseline, Week 24, Week 48, Week 72, Week 96
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | ABBV-8E12 300 mg | ABBV-8E12 1000 mg | ABBV-8E12 2000 mg
Number analyzed (Participants) | 116 | 108 | 116 | 113
score on a scale
  Change to Week 24: number analyzed (Participants) | 111 | 106 | 112 | 102
  Change to Week 24 | -0.93 (0.132) | -1.01 (0.135) | -0.93 (0.131) | -0.95 (0.137)
  Change to Week 48: number analyzed (Participants) | 101 | 91 | 105 | 93
  Change to Week 48 | -0.70 (0.178) | -0.95 (0.186) | -0.60 (0.175) | -0.69 (0.137)
  Change to Week 72: number analyzed (Participants) | 100 | 92 | 97 | 94
  Change to Week 72 | -0.90 (0.179) | -1.12 (0.186) | -0.90 (0.181) | -1.38 (0.185)
  Change to Week 96: number analyzed (Participants) | 81 | 79 | 86 | 74
  Change to Week 96 | -1.28 (0.197) | -1.10 (0.201) | -0.96 (0.192) | -1.35 (0.205)
Statistical Analysis 1: Comparison: Placebo vs ABBV-8E12 300 mg; Week 24; Test type: Superiority; p = 0.683, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.08, 95% CI 2-sided [-0.442 to 0.290], Standard Error of Mean 0.186
Statistical Analysis 2: Comparison: Placebo vs ABBV-8E12 300 mg; Week 24; Test type: Superiority; Effect size/pooled SD = -0.04, Standard Deviation 1.98 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 24; Test type: Superiority; p = 0.973, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = 0.01, 95% CI 2-sided [-0.356 to 0.368], Standard Error of Mean 0.184
Statistical Analysis 4: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 24; Test type: Superiority; Effect size/pooled SD = 0.00, Standard Deviation 1.78 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 5: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 24; Test type: Superiority; p = 0.921, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.02, 95% CI 2-sided [-0.389 to 0.352], Standard Error of Mean 0.189
Statistical Analysis 6: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 24; Test type: Superiority; Effect size/pooled SD = -0.01, Standard Deviation 1.74 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 7: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; p = 0.335, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.25, 95% CI 2-sided [-0.751 to 0.257], Standard Error of Mean 0.256
Statistical Analysis 8: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; Effect size/pooled SD = -0.11, Standard Deviation 2.20 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 9: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; p = 0.670, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = 0.11, 95% CI 2-sided [-0.383 to 0.596], Standard Error of Mean 0.249
Statistical Analysis 10: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.05, Standard Deviation 2.01 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 11: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Superiority; p = 0.950, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = 0.02, 95% CI 2-sided [-0.486 to 0.519], Standard Error of Mean 0.256
Statistical Analysis 12: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.01, Standard Deviation 2.04 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 13: Comparison: Placebo vs ABBV-8E12 300 mg; Week 72; Test type: Superiority; p = 0.383, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.22, 95% CI 2-sided [-0.729 to 0.281], Standard Error of Mean 0.257
Statistical Analysis 14: Comparison: Placebo vs ABBV-8E12 300 mg; Week 24; Test type: Superiority; Effect size/pooled SD = -0.10, Standard Deviation 2.33 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 15: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 72; Test type: Superiority; p = 0.985, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.00, 95% CI 2-sided [-0.504 to 0.494], Standard Error of Mean 0.254
Statistical Analysis 16: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 72; Test type: Superiority; Effect size/pooled SD = -0.00, Standard Deviation 2.23 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 17: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 72; Test type: Superiority; p = 0.064, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.48, 95% CI 2-sided [-0.982 to 0.027], Standard Error of Mean 0.256
Statistical Analysis 18: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 72; Test type: Superiority; Effect size/pooled SD = -0.20, Standard Deviation 2.40 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 19: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; p = 0.527, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = 0.18, 95% CI 2-sided [-0.374 to 0.729], Standard Error of Mean 0.280
Statistical Analysis 20: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; Effect size/pooled SD = 0.08, Standard Deviation 2.30 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 21: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; p = 0.254, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = 0.31, 95% CI 2-sided [-0.226 to 0.854], Standard Error of Mean 0.275
Statistical Analysis 22: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = 0.14, Standard Deviation 2.32 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 23: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; p = 0.805, repeated measures model — [p-value comment as in outcome 32, analysis 1]; LS Mean of Difference = -0.07, 95% CI 2-sided [-0.628 to 0.488], Standard Error of Mean 0.284
Statistical Analysis 24: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = -0.03, Standard Deviation 2.13 — [estimate comment as in outcome 30, analysis 2]

45. Secondary Outcome: Change From Baseline Over Time in Mini-Mental State Examination (MMSE) Total Score
Description: The MMSE is a brief, 30-point questionnaire, administered by a trained rater, which provides a quantitative measure of cognitive status in adults and is widely used to screen for cognitive impairment and to estimate the severity of cognitive impairment at a given point in time in AD participants. The MMSE ranges from 0 to 30, with lower scores indicating greater impairment.
Time Frame: Baseline, Week 24, Week 48, Week 72, Week 96
Population: as for outcome 14
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | ABBV-8E12 300 mg | ABBV-8E12 1000 mg | ABBV-8E12 2000 mg
Number analyzed (Participants) | 116 | 108 | 116 | 113
score on a scale
  Change at Week 24: number analyzed (Participants) | 111 | 106 | 113 | 103
  Change at Week 24 | -0.60 (0.255) | -0.83 (0.260) | -0.48 (0.252) | -1.56 (0.263)
  Change at Week 48: number analyzed (Participants) | 102 | 92 | 105 | 92
  Change at Week 48 | -1.78 (0.294) | -1.81 (0.305) | -1.60 (0.290) | -2.17 (0.305)
  Change at Week 72: number analyzed (Participants) | 100 | 91 | 97 | 94
  Change at Week 72 | -2.83 (0.376) | -2.92 (0.388) | -2.43 (0.375) | -3.34 (0.386)
  Change at Week 96: number analyzed (Participants) | 83 | 81 | 88 | 76
  Change at Week 96 | -3.95 (0.478) | -4.06 (0.488) | -3.70 (0.469) | -4.71 (0.494)
Statistical Analysis 1: Comparison: Placebo vs ABBV-8E12 300 mg; Week 24; Test type: Superiority; p = 0.534, repeated measures model — The statistical model: MMSE change from baseline = baseline + treatment + site + visit + baseline*visit + treatment*visit; variance-covariance structure = Unstructured; LS Mean of Difference = -0.22, 95% CI 2-sided [-0.935 to 0.485], Standard Error of Mean 0.361
Statistical Analysis 2: Comparison: Placebo vs ABBV-8E12 300 mg; Week 24; Test type: Superiority; Effect size/pooled SD = -0.08, Standard Deviation 2.76 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 24; Test type: Superiority; p = 0.735, repeated measures model — [p-value comment as in outcome 45, analysis 1]; LS Mean of Difference = 0.12, 95% CI 2-sided [-0.580 to 0.821], Standard Error of Mean 0.356
Statistical Analysis 4: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 24; Test type: Superiority; Effect size/pooled SD = 0.04, Standard Deviation 2.74 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 5: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 24; Test type: Superiority; p = 0.009, repeated measures model — [p-value comment as in outcome 45, analysis 1]; LS Mean of Difference = -0.96, 95% CI 2-sided [-1.673 to -0.240], Standard Error of Mean 0.365
Statistical Analysis 6: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 24; Test type: Superiority; Effect size/pooled SD = -0.35, Standard Deviation 2.75 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 7: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; p = 0.954, repeated measures model — [p-value comment as in outcome 45, analysis 1]; LS Mean of Difference = -0.02, 95% CI 2-sided [-0.854 to 0.806], Standard Error of Mean 0.422
Statistical Analysis 8: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; Effect size/pooled SD = -0.01, Standard Deviation 2.97 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 9: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; p = 0.649, repeated measures model — [p-value comment as in outcome 45, analysis 1]; LS Mean of Difference = 0.19, 95% CI 2-sided [-0.622 to 0.997], Standard Error of Mean 0.412
Statistical Analysis 10: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.06, Standard Deviation 2.95 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 11: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Superiority; p = 0.358, repeated measures model — [p-value comment as in outcome 45, analysis 1]; LS Mean of Difference = -0.39, 95% CI 2-sided [-1.220 to 0.443], Standard Error of Mean 0.423
Statistical Analysis 12: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = -0.13, Standard Deviation 2.99 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 13: Comparison: Placebo vs ABBV-8E12 300 mg; Week 72; Test type: Superiority; p = 0.859, repeated measures model — [p-value comment as in outcome 45, analysis 1]; LS Mean of Difference = -0.10, 95% CI 2-sided [-1.155 to 0.963], Standard Error of Mean 0.539
Statistical Analysis 14: Comparison: Placebo vs ABBV-8E12 300 mg; Week 72; Test type: Superiority; Effect size/pooled SD = -0.03, Standard Deviation 3.74 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 15: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 72; Test type: Superiority; p = 0.455, repeated measures model — [p-value comment as in outcome 45, analysis 1]; LS Mean of Difference = 0.40, 95% CI 2-sided [-0.644 to 1.437], Standard Error of Mean 0.529
Statistical Analysis 16: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 72; Test type: Superiority; Effect size/pooled SD = 0.11, Standard Deviation 3.60 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 17: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 72; Test type: Superiority; p = 0.335, repeated measures model — [p-value comment as in outcome 45, analysis 1]; LS Mean of Difference = -0.52, 95% CI 2-sided [-1.578 to 0.539], Standard Error of Mean 0.538
Statistical Analysis 18: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 72; Test type: Superiority; Effect size/pooled SD = -0.15, Standard Deviation 3.57 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 19: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; p = 0.875, repeated measures model — [p-value comment as in outcome 45, analysis 1]; LS Mean of Difference = -0.11, 95% CI 2-sided [-1.447 to 1.233], Standard Error of Mean 0.681
Statistical Analysis 20: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; Effect size/pooled SD = -0.02, Standard Deviation 4.57 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 21: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; p = 0.712, repeated measures model — [p-value comment as in outcome 45, analysis 1]; LS Mean of Difference = 0.25, 95% CI 2-sided [-1.068 to 1.561], Standard Error of Mean 0.668
Statistical Analysis 22: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = 0.05, Standard Deviation 4.62 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 23: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; p = 0.269, repeated measures model — [p-value comment as in outcome 45, analysis 1]; LS Mean of Difference = -0.76, 95% CI 2-sided [-2.112 to 0.590], Standard Error of Mean 0.687
Statistical Analysis 24: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = -0.16, Standard Deviation 4.78 — [estimate comment as in outcome 30, analysis 2]

46. Secondary Outcome: Change From Baseline Over Time in Neuropsychiatry Inventory (NPI) Total Score
Description: The NPI is used to assess changes in the participant's behavior that occurred in a defined period of time (4 weeks). The NPI assesses 12 behavioral domains on the dimensions of frequency and severity. Frequency is rated on a scale where 0 = absent, 1 = occasionally, 2 = often, 3 = frequently, 4 = very frequently. Severity is rated on a scale where 0 = absent, 1 = mild, 2 = moderate, 3 = severe. For each of the domains, 3 scores are obtained: frequency, severity, and total (product of frequency and severity; ranges from 0 to 12, with a lower score desirable). A total NPI score can be calculated by summing the domain total scores. Total Score ranges from 0 to 144 with a lower score desirable.
Time Frame: Baseline, Week 24, Week 48, Week 72, Week 96
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | ABBV-8E12 300 mg | ABBV-8E12 1000 mg | ABBV-8E12 2000 mg
Number analyzed (Participants) | 116 | 108 | 116 | 113
score on a scale
  Change at Week 24: number analyzed (Participants) | 111 | 105 | 111 | 101
  Change at Week 24 | 0.93 (0.551) | 0.96 (0.567) | 0.80 (0.551) | 1.92 (0.576)
  Change at Week 36: number analyzed (Participants) | 104 | 96 | 107 | 98
  Change at Week 36 | -0.03 (0.487) | 0.84 (0.505) | 0.99 (0.481) | 1.32 (0.502)
  Change at Week 72: number analyzed (Participants) | 102 | 95 | 100 | 96
  Change at Week 72 | 1.34 (0.742) | 1.52 (0.767) | 1.80 (0.745) | 3.25 (0.765)
  Change at Week 96: number analyzed (Participants) | 86 | 86 | 91 | 82
  Change at Week 96 | 2.38 (0.784) | 2.03 (0.794) | 2.53 (0.769) | 2.94 (0.804)
Statistical Analysis 1: Comparison: Placebo vs ABBV-8E12 300 mg; Week 24; Test type: Superiority; p = 0.966, repeated measures model — The statistical model: NPI change from baseline = baseline + treatment + site + visit + baseline*visit + treatment*visit; variance-covariance structure = Unstructured; LS Mean of Difference = 0.03, 95% CI 2-sided [-1.509 to 1.577], Standard Error of Mean 0.785
Statistical Analysis 2: Comparison: Placebo vs ABBV-8E12 300 mg; Week 24; Test type: Superiority; Effect size/pooled SD = -0.01, Standard Deviation 6.32 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 24; Test type: Superiority; p = 0.874, repeated measures model — [p-value comment as in outcome 46, analysis 1]; LS Mean of Difference = -0.12, 95% CI 2-sided [-1.646 to 1.400], Standard Error of Mean 0.775
Statistical Analysis 4: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 24; Test type: Superiority; Effect size/pooled SD = 0.02, Standard Deviation 5.89 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 5: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 24; Test type: Superiority; p = 0.213, repeated measures model — [p-value comment as in outcome 46, analysis 1]; LS Mean of Difference = 0.99, 95% CI 2-sided [-0.572 to 2.551], Standard Error of Mean 0.794
Statistical Analysis 6: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 24; Test type: Superiority; Effect size/pooled SD = -0.15, Standard Deviation 6.67 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 7: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; p = 0.208, repeated measures model — [p-value comment as in outcome 46, analysis 1]; LS Mean of Difference = 0.88, 95% CI 2-sided [-0.490 to 2.242], Standard Error of Mean 0.695
Statistical Analysis 8: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; Effect size/pooled SD = -0.17, Standard Deviation 5.26 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 9: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; p = 0.131, repeated measures model — [p-value comment as in outcome 46, analysis 1]; LS Mean of Difference = 1.03, 95% CI 2-sided [-0.307 to 2.365], Standard Error of Mean 0.680
Statistical Analysis 10: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = -0.18, Standard Deviation 5.57 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 11: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Superiority; p = 0.052, repeated measures model — [p-value comment as in outcome 46, analysis 1]; LS Mean of Difference = 1.35, 95% CI 2-sided [-0.014 to 2.719], Standard Error of Mean 0.695
Statistical Analysis 12: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = -0.24, Standard Deviation 5.55 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 13: Comparison: Placebo vs ABBV-8E12 300 mg; Week 72; Test type: Superiority; p = 0.866, repeated measures model — [p-value comment as in outcome 46, analysis 1]; LS Mean of Difference = 0.18, 95% CI 2-sided [-1.908 to 2.268], Standard Error of Mean 1.062
Statistical Analysis 14: Comparison: Placebo vs ABBV-8E12 300 mg; Week 72; Test type: Superiority; Effect size/pooled SD = -0.03, Standard Deviation 6.15 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 15: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 72; Test type: Superiority; p = 0.660, repeated measures model — [p-value comment as in outcome 46, analysis 1]; LS Mean of Difference = 0.46, 95% CI 2-sided [-1.599 to 2.523], Standard Error of Mean 1.048
Statistical Analysis 16: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 72; Test type: Superiority; Effect size/pooled SD = -0.07, Standard Deviation 6.94 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 17: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 72; Test type: Superiority; p = 0.074, repeated measures model — [p-value comment as in outcome 46, analysis 1]; LS Mean of Difference = 1.91, 95% CI 2-sided [-0.184 to 3.995], Standard Error of Mean 1.062
Statistical Analysis 18: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 72; Test type: Superiority; Effect size/pooled SD = -0.22, Standard Deviation 8.65 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 19: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; p = 0.747, repeated measures model — [p-value comment as in outcome 46, analysis 1]; LS Mean of Difference = -0.36, 95% CI 2-sided [-2.545 to 1.828], Standard Error of Mean 1.111
Statistical Analysis 20: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; Effect size/pooled SD = 0.04, Standard Deviation 7.99
Statistical Analysis 21: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; p = 0.891, repeated measures model — [p-value comment as in outcome 46, analysis 1]; LS Mean of Difference = 0.15, 95% CI 2-sided [-2.004 to 2.304], Standard Error of Mean 1.095
Statistical Analysis 22: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = -0.02, Standard Deviation 8.28 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 23: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; p = 0.621, repeated measures model — [p-value comment as in outcome 46, analysis 1]; LS Mean of Difference = 0.55, 95% CI 2-sided [-1.650 to 2.759], Standard Error of Mean 1.120
Statistical Analysis 24: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = -0.07, Standard Deviation 8.19 — [estimate comment as in outcome 30, analysis 2]

47. Secondary Outcome: Change From Baseline Over Time in Alzheimer's Disease Composite Score (ADCOMS) Score
Description: ADCOMS score is a composite score which is a weighted linear combination of the selected individual scale items from ADAS-Cog-14 (see description in Outcome Measure 10) , MMSE (see description in Outcome Measure 45), and CDR-SB (see description in Outcome Measure 1) scales. The ADCOMS score ranges from 0 to 1.97, with a lower score desirable.
Time Frame: Baseline, Week 24, Week 48, Week 72, Week 96
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | ABBV-8E12 300 mg | ABBV-8E12 1000 mg | ABBV-8E12 2000 mg
Number analyzed (Participants) | 116 | 108 | 116 | 113
score on a scale
  Change at Week 24: number analyzed (Participants) | 100 | 98 | 107 | 95
  Change at Week 24 | 0.05 (0.013) | 0.08 (0.013) | 0.05 (0.013) | 0.08 (0.014)
  Change at Week 48: number analyzed (Participants) | 89 | 82 | 99 | 83
  Change at Week 48 | 0.13 (0.018) | 0.15 (0.018) | 0.13 (0.017) | 0.13 (0.018)
  Change at Week 72: number analyzed (Participants) | 85 | 79 | 85 | 84
  Change at Week 72 | 0.22 (0.023) | 0.22 (0.024) | 0.22 (0.023) | 0.22 (0.024)
  Change at Week 96: number analyzed (Participants) | 72 | 74 | 79 | 65
  Change at Week 96 | 0.29 (0.029) | 0.29 (0.030) | 0.28 (0.029) | 0.35 (0.031)
Statistical Analysis 1: Comparison: Placebo vs ABBV-8E12 300 mg; Week 24; Test type: Superiority; p = 0.147, repeated measures model — The statistical model: ADCOMS change from baseline = baseline + treatment + site + visit + baseline*visit + treatment*visit; variance-covariance structure = Unstructured; LS Mean of Difference = 0.03, 95% CI 2-sided [-0.010 to 0.064], Standard Error of Mean 0.019
Statistical Analysis 2: Comparison: Placebo vs ABBV-8E12 300 mg; Week 24; Test type: Superiority; Effect size/pooled SD = -0.20, Standard Deviation 0.14 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 24; Test type: Superiority; p = 0.795, repeated measures model — [p-value comment as in outcome 47, analysis 1]; LS Mean of Difference = -0.00, 95% CI 2-sided [-0.041 to 0.031], Standard Error of Mean 0.018
Statistical Analysis 4: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 24; Test type: Superiority; Effect size/pooled SD = 0.12, Standard Deviation 0.147 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 5: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 24; Test type: Superiority; p = 0.095, repeated measures model — [p-value comment as in outcome 47, analysis 1]; LS Mean of Difference = 0.03, 95% CI 2-sided [-0.006 to 0.069], Standard Error of Mean 0.019
Statistical Analysis 6: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 24; Test type: Superiority; Effect size/pooled SD = -0.24, Standard Deviation 0.13 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 7: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; p = 0.390, repeated measures model — [p-value comment as in outcome 47, analysis 1]; LS Mean of Difference = 0.02, 95% CI 2-sided [-0.028 to 0.072], Standard Error of Mean 0.025
Statistical Analysis 8: Comparison: Placebo vs ABBV-8E12 300 mg; Week 48; Test type: Superiority; Effect size/pooled SD = -0.12, Standard Deviation 0.18 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 9: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; p = 0.898, repeated measures model — [p-value comment as in outcome 47, analysis 1]; LS Mean of Difference = -0.00, 95% CI 2-sided [-0.052 to 0.045], Standard Error of Mean 0.025
Statistical Analysis 10: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = 0.02, Standard Deviation 0.19 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 11: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Superiority; p = 0.800, repeated measures model — [p-value comment as in outcome 47, analysis 1]; LS Mean of Difference = 0.01, 95% CI 2-sided [-0.044 to 0.057], Standard Error of Mean 0.026
Statistical Analysis 12: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 48; Test type: Superiority; Effect size/pooled SD = -0.04, Standard Deviation 0.18
Statistical Analysis 13: Comparison: Placebo vs ABBV-8E12 300 mg; Week 72; Test type: Superiority; p = 0.977, repeated measures model — [p-value comment as in outcome 47, analysis 1]; LS Mean of Difference = -0.00, 95% CI 2-sided [-0.066 to 0.064], Standard Error of Mean 0.033
Statistical Analysis 14: Comparison: Placebo vs ABBV-8E12 300 mg; Week 72; Test type: Superiority; Effect size/pooled SD = 0.00, Standard Deviation 0.23 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 15: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 72; Test type: Superiority; p = 0.990, repeated measures model — [p-value comment as in outcome 47, analysis 1]; LS Mean of Difference = 0.00, 95% CI 2-sided [-0.063 to 0.064], Standard Error of Mean 0.032
Statistical Analysis 16: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 72; Test type: Superiority; Effect size/pooled SD = -0.00, Standard Deviation 0.24 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 17: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 72; Test type: Superiority; p = 0.944, repeated measures model — [p-value comment as in outcome 47, analysis 1]; LS Mean of Difference = 0.00, 95% CI 2-sided [-0.063 to 0.067], Standard Error of Mean 0.033
Statistical Analysis 18: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 72; Test type: Superiority; Effect size/pooled SD = -0.01, Standard Deviation 0.23 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 19: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; p = 0.942, repeated measures model — [p-value comment as in outcome 47, analysis 1]; LS Mean of Difference = 0.00, 95% CI 2-sided [-0.079 to 0.085], Standard Error of Mean 0.042
Statistical Analysis 20: Comparison: Placebo vs ABBV-8E12 300 mg; Week 96; Test type: Superiority; Effect size/pooled SD = -0.01, Standard Deviation 0.28 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 21: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; p = 0.876, repeated measures model — [p-value comment as in outcome 47, analysis 1]; LS Mean of Difference = -0.01, 95% CI 2-sided [-0.087 to 0.074], Standard Error of Mean 0.041
Statistical Analysis 22: Comparison: Placebo vs ABBV-8E12 1000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = 0.02, Standard Deviation 0.27 — [estimate comment as in outcome 30, analysis 2]
Statistical Analysis 23: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; p = 0.163, repeated measures model — [p-value comment as in outcome 47, analysis 1]; LS Mean of Difference = 0.06, 95% CI 2-sided [-0.024 to 0.143], Standard Error of Mean 0.043
Statistical Analysis 24: Comparison: Placebo vs ABBV-8E12 2000 mg; Week 96; Test type: Superiority; Effect size/pooled SD = -0.21, Standard Deviation 0.28 — [estimate comment as in outcome 30, analysis 2]

ADVERSE EVENTS:
Time Frame: From the time of study drug administration until 20 weeks following discontinuation of study drug administration. Overall median time on study was 680.0 days.
Arm/Group | Placebo | ABBV-8E12 300 mg | ABBV-8E12 1000 mg | ABBV-8E12 2000 mg
All-Cause Mortality (participants affected / at risk) | 1/116 | 2/108 | 2/116 | 1/113
Serious Adverse Events (participants affected / at risk) | 26/116 | 19/108 | 22/116 | 17/113
Other Adverse Events (participants affected / at risk) | 83/116 | 68/108 | 86/116 | 91/113
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=116) | ABBV-8E12 300 mg (N=108) | ABBV-8E12 1000 mg (N=116) | ABBV-8E12 2000 mg (N=113)
ARTERIOSCLEROSIS CORONARY ARTERY (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
ATRIAL FLUTTER (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BRADYCARDIA (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
MYOCARDITIS (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RIGHT VENTRICULAR FAILURE (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SINUS NODE DYSFUNCTION (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DYSPHAGIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GASTRIC ULCER HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PANCREATITIS ACUTE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
STOMACH MASS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ASTHENIA (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
CHEST PAIN (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
NON-CARDIAC CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PYREXIA (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DIVERTICULITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
ENDOCARDITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
EPIGLOTTITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ERYSIPELAS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GASTROENTERITIS VIRAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
PYELONEPHRITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SINUSITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
CHEST INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CLAVICLE FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 3 (4) | 0 (0) | 0 (0) | 1 (1)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HIP FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
MULTIPLE INJURIES (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PNEUMOTHORAX TRAUMATIC (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RIB FRACTURE (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SKIN LACERATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SOFT TISSUE INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
TRAUMATIC INTRACRANIAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
WEIGHT DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ATLANTOAXIAL SUBLUXATION (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CERVICAL SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BREAST CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GASTROINTESTINAL STROMAL TUMOUR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PROSTATIC ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CEREBRAL MASS EFFECT (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
DEMENTIA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DEMENTIA ALZHEIMER'S TYPE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ENCEPHALOPATHY (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HEADACHE (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
MOTOR NEURONE DISEASE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NORMAL PRESSURE HYDROCEPHALUS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PRESYNCOPE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SCIATICA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SEIZURE (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
SYNCOPE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
THALAMUS HAEMORRHAGE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
AGGRESSION (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
AGITATION (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
DELIRIUM (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MENTAL STATUS CHANGES (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PSYCHOTIC DISORDER DUE TO A GENERAL MEDICAL CONDITION (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SUICIDAL IDEATION (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NEPHROLITHIASIS (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
POLYURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RENAL FAILURE (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
RESPIRATORY TRACT CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
URTICARIA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPERTENSIVE CRISIS (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYPOTENSION (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=116) | ABBV-8E12 300 mg (N=108) | ABBV-8E12 1000 mg (N=116) | ABBV-8E12 2000 mg (N=113)
DIARRHOEA (Gastrointestinal disorders) | 9 (10) | 12 (15) | 10 (11) | 12 (12)
NAUSEA (Gastrointestinal disorders) | 2 (2) | 5 (9) | 4 (5) | 10 (12)
VOMITING (Gastrointestinal disorders) | 3 (4) | 5 (5) | 2 (2) | 11 (14)
FATIGUE (General disorders) | 11 (12) | 6 (6) | 7 (7) | 8 (31)
SEASONAL ALLERGY (Immune system disorders) | 6 (6) | 3 (3) | 2 (3) | 2 (2)
BRONCHITIS (Infections and infestations) | 6 (6) | 0 (0) | 1 (1) | 3 (3)
INFLUENZA (Infections and infestations) | 0 (0) | 2 (2) | 3 (3) | 6 (6)
NASOPHARYNGITIS (Infections and infestations) | 11 (12) | 11 (12) | 12 (16) | 12 (14)
SINUSITIS (Infections and infestations) | 8 (10) | 0 (0) | 3 (3) | 3 (4)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 9 (13) | 7 (11) | 12 (14) | 18 (19)
URINARY TRACT INFECTION (Infections and infestations) | 12 (17) | 11 (12) | 13 (16) | 11 (11)
CONTUSION (Injury, poisoning and procedural complications) | 8 (10) | 6 (7) | 8 (8) | 5 (6)
FALL (Injury, poisoning and procedural complications) | 22 (39) | 21 (33) | 17 (23) | 25 (37)
SKIN ABRASION (Injury, poisoning and procedural complications) | 2 (5) | 7 (8) | 2 (2) | 1 (2)
SKIN LACERATION (Injury, poisoning and procedural complications) | 6 (6) | 4 (4) | 6 (6) | 7 (7)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 9 (11) | 7 (7) | 12 (14) | 10 (12)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 7 (8) | 9 (12) | 11 (11) | 11 (11)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 6 (9) | 2 (2)
CEREBRAL MICROHAEMORRHAGE (Nervous system disorders) | 4 (4) | 2 (2) | 6 (6) | 3 (3)
DIZZINESS (Nervous system disorders) | 10 (13) | 14 (20) | 9 (11) | 14 (14)
HEADACHE (Nervous system disorders) | 11 (12) | 9 (11) | 11 (15) | 20 (29)
ANXIETY (Psychiatric disorders) | 11 (11) | 3 (4) | 9 (11) | 16 (17)
DEPRESSION (Psychiatric disorders) | 11 (11) | 10 (10) | 8 (10) | 12 (13)
INSOMNIA (Psychiatric disorders) | 3 (3) | 7 (7) | 2 (2) | 3 (3)
COUGH (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 3 (3) | 7 (7) | 9 (11)
HYPERTENSION (Vascular disorders) | 2 (2) | 2 (2) | 6 (6) | 5 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2020-10-02): https://cdn.clinicaltrials.gov/large-docs/56/NCT02880956/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-19): https://cdn.clinicaltrials.gov/large-docs/56/NCT02880956/SAP_001.pdf